Statistical Analysis Plan I1F-MC-RHCF (v2)

A 52-Week Multicenter, Randomized, Open-Label, Parallel-Group Study Evaluating the Efficacy and Safety of Ixekizumab versus Adalimumab in Patients with Psoriatic Arthritis Who Are Biologic Disease-Modifying Anti-Rheumatic Drug Naïve

NCT03151551

Approval Date: 03-Dec-2018

# 1. Statistical Analysis Plan:

I1F-MC-RHCF: A 52-Week Multicenter, Randomized,
Open-Label, Parallel-Group Study Evaluating the Efficacy
and Safety of Ixekizumab versus Adalimumab in Patients
with Psoriatic Arthritis Who Are Biologic DiseaseModifying Anti-Rheumatic Drug Naive

#### **Confidential Information**

The information contained in this document is confidential and the information contained within it may not be reproduced or otherwise disseminated without the approval of Eli Lilly and Company or its subsidiares.

Note to Regulatory Authorities: This document may contain protected personal data and/or commercially confidential information exempt from public disclosure. Eli Lilly and Company requests consultation regarding release/redaction prior to any public release. In the United States, this document is subject to Freedom of Information Act (FOIA) Exemption 4 and may not be reproduced or otherwise disseminated without the written approval of Eli Lilly and Company or its subsidiaries.

#### Ixekizumab (LY2439821) Psoriatic Arthritis

Study I1F-MC-RHCF is a Phase 3b/4, multicenter, randomized, open-label, parallel-group study with blinded outcomes assessments evaluating the efficacy and safety of ixekizumab versus adalimumab in patients with psoriatic arthritis who are biologic disease-modifying anti-rheumatic drug naive during a 52-week treatment period.

Eli Lilly and Company Indianapolis, Indiana USA 46285 Protocol I1F-MC-RHCF Phase 3b/4

Statistical Analysis Plan Version 1 electronically signed and approved by Lilly on Aug 21, 2017.

Statistical Analysis Plan Version 2 electronically signed and approved by Lilly on date provided below.

Approval Date: 03-Dec-2018 GMT

# 2. Table of Contents

| Section | | Page |
|---|---|---|
| Randon<br>Efficac<br>with Ps | cal Analysis Plan: I1F-MC-RHCF: A 52-Week Multicenter, mized, Open-Label, Parallel-Group Study Evaluating the sy and Safety of Ixekizumab versus Adalimumab in Patients soriatic Arthritis Who Are Biologic Disease-Modifying Anti-natic Drug Naive | 1 |
| 2. Table o | of Contents | 2 |
| 3. Revisio | on History | 7 |
| 4. Study 0 | Objectives | 9 |
| 5. Study I | Design | 12 |
| | nmary of Study Design | |
| 5.2. Det | ermination of Sample Size | 13 |
| 5.3. Met | thod of Assignment to Treatment | 14 |
| 6. A Prior | ri Statistical Methods | 15 |
| 6.1. Gen | neral Considerations | 15 |
| 6.1.1. | General Considerations for the Open-Label Treatment Period (Period 2) | 16 |
| 6.1.2. | General Considerations for the Post-Treatment Follow-Up<br>Period (Period 3) | 17 |
| 6.1.3. | Analysis Populations | 17 |
| 6.2. Ana | llysis Methods | 18 |
| 6.2.1. | Categorical | 18 |
| 6.2.2. | Continuous Endpoints | 18 |
| 6.3. Adj | ustments for Covariates | 19 |
| 6.4. Han | dling of Dropouts or Missing Data | 19 |
| 6.4.1. | Non-Responder Imputation (NRI) for Clinical Response | |
| 6.4.2. | Modified Baseline Observation Carried Forward (mBOCF) | 19 |
| 6.4.3. | Missing Data Imputation for Adverse Event and Concomitant Medication Dates | 20 |
| 6.5. Mul | ticenter Studies | 20 |
| 6.6. Mul | tiple Comparisons/Multiplicity | 20 |
| 6.7. Met | chodology for Noninferiority Test. | 21 |
| 6.8. Pati | ent Disposition | 21 |
| 6.9. Pati | ent Characteristics | |
| 6.9.1. | Demographics and Baseline Characteristics. | 23 |
| 6.9.2. | Previous Therapy for Psoriatic Arthritis | 25 |
| 6.9.3. | Historical Illness and Pre-existing Conditions | 26 |

| 6.10. Treatment Compliance | 26 |
|---|---|
| 6.11. Concomitant Therapy | 27 |
| 6.12. Efficacy Analyses | 28 |
| 6.12.1. Analysis Methodology for Primary and Major Secondary | |
| Outcomes | 48 |
| 6.12.1.1. Primary Outcome and Methodology | 48 |
| 6.12.1.2. Methodology for Major Secondary Outcomes | 48 |
| 6.12.1.3. Other Secondary Outcomes | 48 |
| 6.13. Health Outcomes/Quality-of-Life Analyses | 49 |
| 6.14. Bioanalytical and Pharmacokinetic/Pharmacodynamic Methods | 61 |
| 6.15. Safety Analyses | 61 |
| 6.15.1. Extent of Exposure | 61 |
| 6.15.2. Adverse Events | 62 |
| 6.15.2.1. Analyses of Adverse Events | 62 |
| 6.15.2.2. Common Adverse Events | 63 |
| 6.15.3. Deaths, Other Serious Adverse Events, and Other Notable | |
| Adverse Events | 64 |
| 6.15.3.1. Special Safety Topics Including Adverse Events of Special Interest | 64 |
| 6.15.4. Clinical Laboratory Evaluation | 76 |
| 6.15.4.1. Leukocytes (White Blood Cells) and Platelets | 77 |
| 6.15.4.2. Neutrophil Follow-Up | 78 |
| 6.15.5. Vital Signs and Other Physical Findings | 78 |
| 6.15.6. Columbia-Suicide Severity Rating Scale | 80 |
| 6.15.7. Immunogenicity | 81 |
| 6.15.8. Electrocardiograms | 81 |
| 6.16. Subgroup Analyses | 81 |
| 6.16.1. Safety Subgroup Analyses | 81 |
| 6.16.2. Efficacy Subgroup Analyses | 82 |
| 6.17. Protocol Violations | 83 |
| 6.18. Interim Analyses and Data Monitoring | |
| 6.19. Clinical Trial Registry Analyses | |
| 7. References | |
| 8. Appendices | |
| o. Appendices | 102 |

### **Table of Contents**

| Table | Page |
|---|---|
| Table RHCF.4.1. Objectives and Endpoints | 9 |
| Table RHCF.6.1. Treatment Groups for Each Treatment Period and Analysis Population. | 16 |
| Table RHCF.6.2. Efficacy, Health Outcomes, and Safety Measures Summarized and/or Analyzed for Each Analysis Population | 18 |
| Table RHCF.6.3. Description and Derivation of Primary and Secondary Efficacy Outcomes | 29 |
| Table RHCF.6.4. Description of Primary and Secondary Efficacy Analyses | 40 |
| Table RHCF.6.5. Description and Derivation of Health Outcomes and Quality-of-Life Measures | 50 |
| Table RHCF.6.6. Description of Health Outcomes and Quality-of-Life Analyses | 58 |
| Table RHCF.6.7. Definitions and Analyses of Special Safety Topics | 66 |
| Table RHCF.6.8. Categorical Criteria for Abnormal Treatment-Emergent Blood Pressure and Pulse Measurement, and Categorical Criteria for Weight and Changes for Adults | |
| Table RHCF.6.9. Identification and Action of Important Protocol Violations | 84 |

| Ρ | ac | ıe | 5 |
|---|----|----|---|

| | | _ | _ | | |
|-----|-----|------------|------------|-----|-----|
| Tab | | | <b>^</b> - | 4 - | 1_ |
| ıar | מוו | $\Delta T$ | . ^ | nto | nte |

| Figure | | Page |
|---|---|---|
| Figure RHCF.5.1. | Illustration of study design for Clinical Protocol I1F-MC-RHCF. | 13 |

### **Table of Contents**

| Appendix | | Page |
|---|---|---|
| Appendix 1. | Definition of Numbers Needed to Treat (NNT) | 103 |
| Appendix 2. | Algorithm for Determining ACR Responses | 106 |
| Appendix 3. | Algorithm for Calculating Joint Counts. | 108 |
| Appendix 4. | Algorithm for Calculating the HAQ-DI | 109 |
| Appendix 5. | Algorithm for Calculating CPDAI and mCPDAI | 111 |
| Appendix 6. | Deviation of SF-36v2® Health Survey, Acute Version Scores | 113 |
| Appendix 7. | Anti-infective Treatments and Anatomical Therapeutic Chemical (ATC) Code List | 119 |
| Appendix 8. | Lilly-Defined MedDRA V21.0 Preferred Terms for Opportunistic Infections (OIs) | 124 |
| Appendix 9. | MedDRA Preferred Terms for each Category Associated with Criterion 2 for Anaphylactic Allergic Reactions/Hypersensitivity Events | 134 |
| Appendix 10. | Allergic Reactions/Hypersensitivity MedDRA Preferred Term List | 136 |
| Appendix 11. | Lilly-Defined MedDRA V21.0 Preferred Terms for Inflammatory Bowel Disease (IBD) | 139 |

# 3. Revision History

Statistical Analysis Plan (SAP) Version 1 was approved prior to first patient visit (FPV).

Statistical Analysis Plan (SAP) Version 2 was approved prior to interim 1 database lock (24 week).

Revisions since Version 1:

| Section | Action |
|---|---|
| Section 6.1 General Considerations | Updated p-values to 3 decimal places. |
| | Corrected typo. |
| Section 6.1.1 General | Revised baseline definition to last available value "on or prior to" the first |
| Considerations for Open-Label | injection of the study drug. |
| Treatment Period (Period 2) | |
| Section 6.7 Methodology for | Updated references. |
| Noninferiority Test | |
| Section 6.9.1 Demographics and | Removed Composite Psoriatic Disease Activity Index (CPDAI). |
| Baseline Characteristics | |
| Section 6.9.3 Historical Illness and | Clarified definitions of historical illness and pre-existing conditions. |
| Pre-existing Conditions | |
| Section 6.11 Concomitant Therapy | Removed unnecessary analyses for concomitant therapy. |
| Section 6.12 Efficacy Analyses | Updated imputation mehods for MDA, LEI and LDI-B. |
| Table 6.3 | |
| Section 6.12 Efficacy Analyses | Added Kaplan-Meier plots for time to first simultaneous ACR50 and PASI |
| Table 6.4 | 100 response. |
| | Updated time points of Kaplan Meier plots. |
| Section 6.12.1.3 Other Secondary | Removed by-patient listings for secondary efficacy measure. |
| Outcomes | |
| Section 6.13 Health | Removed by-patient listings for health outcome measure. |
| Outcomes/Quality-of-Life Analyses | |
| Section 6.13 Health | Update analysis population for analyses regrading to Itch NRS = 0. |
| Outcomes/Quality-of-Life Analyses | |
| Table 6.6 | |
| Section 6.15.1 Extent of Exposure | Removed by-patient listing for extent of exposure. |
| Section 6.15.3.1 Special Safety | Text updates for definition/derivation of AESIs to be consistent with PSAP |
| Topics Including Adverse Events of | V8 |
| Special Interest Table 6.7 | Removed duplicated or unnecessary analyses |
| Table 6.7 | Changed Covance to performing lab reference range |
| | Wording updates per most recent PSAP for Infections, Allergic |
| Section 6.15 A Clinical Laboratory | Reactions/Hypersensitivities, Injection Site Reactions, CV, IBD, ILD. |
| Section 6.15.4 Clinical Laboratory | Updated population for laboratory analyses. |
| Evaluation | Removed by-patient listings. |
| Section 6.15.5 Vital Signs and Other | Updated population for vital signs analyses. |
| Physical Findings | Removed by-patient listing. |

| Section | Action |
|---|---|
| Section 6.15.6 Columbia-Suicide | Updated C-SSRS analyses. |
| Severity Rating Scale | |
| Section 6.16.1 Efficacy Subgroup | Added additional exploratory subgroup analyses. |
| Analyses | |
| Section 6.17 Protocol Violations | Added potential additional analyses. |
| Section 6.17 Protocol Violations | Updated important protocol violations per most recent Trial Issue |
| Table 6.9 | Management Plan. |
| Section 6.19 Planned Exploratory | Removed exploratory subgroup analyses. |
| Analyses | |
| Appendix 1 | Updated NNT CI calculation method. |
| Appendix 2 | Removed Appendix 2. |
| Appendix 4 | Clarified the algorithm for calculating Joint Counts. |
| Appendix 7 | Updated norms to 2009. |
| Appendices 9-12 | Updated per PSAP V8. |

# 4. Study Objectives

Table RHCF.4.1 shows the objectives and endpoints of the study.

Table RHCF.4.1. Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | • |
| To assess whether ixekizumab | |
| is superior to adalimumab at | |
| Week 24 in the treatment of | D C C C C C C C C C C C C C C C C C C C |
| patients with active PsA as | Proportion of patients simultaneously achieving ACR50 and PASI 100 ACR50 and PASI 100 |
| measured by American College | at Week 24 |
| of Rheumatology 50 (ACR50) | |
| and Psoriasis Area and Severity | |
| Index 100 (PASI 100) | |
| Major Secondary Objectives: | |
| To assess whether ixekizumab | |
| is noninferior to adalimumab at | <ul> <li>Proportion of patients achieving ACR50 in each treatment group at</li> </ul> |
| Week 24 in the treatment of | Week 24 |
| patients with active PsA as | |
| measured by ACR50 | |
| To assess whether ixekizumab | |
| is superior to adalimumab at | <ul> <li>Proportion of patients achieving PASI 100 in each treatment group at</li> </ul> |
| Week 24 in the treatment of | Week 24 |
| patients with active PsA as | |
| measured by PASI 100 | |
| Other Secondary Objectives: | PsA Endpoints |
| To assess the effect of treatment | Time course of response to treatment over 52 weeks as measured by: |
| with ixekizumab compared with | <ul> <li>Proportion of patients achieving ACR20, ACR50, and ACR70 responses</li> </ul> |
| adalimumab as measured by | Change from baseline in individual components of the American |
| efficacy and quality of life | College of Rheumatology (ACR) Core Set - tender joint count, swollen |
| outcomes | joint count, patient's pain assessment, Patient's Global Assessment of |
| | Disease Activity, Physician's Global Assessment of Disease Activity, |
| | C-reactive protein (CRP), and Health Assessment Questionnaire— |
| | Disability Index (HAQ-DI) score |
| | Proportion of patients simultaneously achieving ACR50 and Proportion of patients simultaneously achieving ACR50 and Proportion of patients simultaneously achieving ACR50 and Proportion of patients simultaneously achieving ACR50 and |
| | PASI 100 response |
| | Change from baseline in the Disease Activity Score (28 diarthrodial (2) + (3) + (3) + (3) + (4) + ( |
| | joint count) based on C-reactive protein (DAS28-CRP) |
| | Proportion of patients achieving Minimal Disease Activity (MDA) Proportion of patients achieving Proportion Activities Proportion of Criterian Output Description of Proportion of Proportion Activities Proportion of Pro |
| | Proportion of patients achieving Psoriatic Arthritis Response Criteria (P-ABC) |
| | (PsARC) Change from baseline in Medified Commonite Provide Disease Activity |
| | Change from baseline in Modified Composite Psoriatic Disease Activity Index (CRDA) seems. |
| | Index (CPDAI) score |
| | Proportion of patients achieving low disease activity or remission according to the Modified Composite Psoriatic Disease Activity Index |
| | according to the Modified Composite Psoriatic Disease Activity Index |
| | definition |

| Objectives | Endpoints |
|---|---|
| | <ul> <li>Proportion of patients with HAQ-DI improvement ≥0.35</li> <li>Change from baseline in the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index score in patients with enthesitis at baseline (ie, baseline SPARCC Enthesitis Index (LEI) score in patients with enthesitis at baseline (ie, baseline LEI score &gt;0)</li> <li>Proportion of patients with resolution in enthesitis in the subgroup of patients with enthesitis at baseline as measured by the SPARCC Enthesitis Index (ie, baseline SPARCC Enthesitis Index score &gt;0)</li> <li>Proportion of patients with resolution in enthesitis in the subgroup of patients with enthesitis at baseline as measured by the LEI (ie, baseline LEI score &gt;0)</li> <li>Change from baseline in the Leeds Dactylitis Index-Basic (LDI-B) score in patients with dactylitis at baseline (ie, baseline LDI-B score &gt;0)</li> <li>Proportion of patients with resolution in dactylitis in the subgroup of patients with dactylitis at baseline as measured by the LDI-B (ie, baseline LDI-B score &gt;0)</li> </ul> |
| | <ul> <li>Psoriasis/Nail Endpoints</li> <li>Time course of response to treatment over 52 weeks as measured by: <ul> <li>Change from baseline in body surface area (BSA)</li> </ul> </li> <li>Proportion of patients who achieve the following PASI scores: <ul> <li>PASI 75, PASI 90, or PASI 100 (defined as 75%, 90%, and 100% improvement from baseline in PASI criteria, respectively)</li> </ul> </li> <li>Proportion of patients achieving an absolute PASI score ≤1 or ≤2 or ≤3</li> <li>Change from baseline in the Nail Psoriasis Severity Index (NAPSI) <ul> <li>Fingernails score in the subgroup of patients with fingernail involvement at baseline (ie, baseline NAPSI Fingernails score &gt;0)</li> </ul> </li> </ul> |
| | <ul> <li>QoL Endpoints</li> <li>Time course of response to treatment over 52 weeks as measured by: <ul> <li>Change from baseline in the Itch Numeric Rating Scale (NRS) score</li> <li>Proportion of patients with Itch NRS score equal to 0</li> <li>Change from baseline in Fatigue Severity NRS score</li> <li>Change from baseline in Medical Outcomes Study 36-Item Short Form Health Survey (SF-36)</li> <li>Physical Component Summary score</li> <li>Mental Component Summary score</li> <li>Change from baseline in measures of health utility (European Quality of Life-5 Dimensions 5 Level health outcomes instrument [EQ-5D-5L])</li> <li>Change from baseline in Dermatology Life Quality Index (DLQI) total score</li> <li>Change from baseline in Treatment Satisfaction Questionnaire</li> </ul> </li> </ul> |
| | Safety ■ Change from baseline in Columbia—Suicide Severity Rating Scale (C-SSRS) |

Abbreviations: ACR50 = American College of Rheumatology 50; BSA = body surface area; CPDAI = Composite Psoriatic Disease Activity Index; CRP = C-reactive protein; C-SSRS = Columbia–Suicide Severity Rating Scale; DAS28-CRP = Disease Activity Score (28 diarthrodial joint count) based on C-reactive protein; DLQI = Dermatology Life Quality Index; EQ-5D-5L = European Quality of Life–5 Dimensions 5 Level health outcomes instrument; HAQ-DI = Health Assessment Questionnaire–Disability Index; LDI-B = Leeds Dactylitis Index-Basic; LEI = Leeds Enthesitis Index; MDA = Minimal Disease Activity; NAPSI = Nail Psoriasis Severity Index; NRS = Numeric Rating Scale; PASI 100 = Psoriasis Area and Severity Index 100; PsA = psoriatic arthritis; PsARC = Psoriatic Arthritis Response Criteria; SF-36 = 36-Item Short Form Health Survey; SPARCC = Spondyloarthritis Research Consortium of Canada.

# 5. Study Design

### 5.1. Summary of Study Design

Study I1F-MC-RHCF (RHCF) is a Phase 3b/4, multicenter, randomized, open-label, parallel-group study with blinded outcomes assessments evaluating the efficacy and safety of ixekizumab versus adalimumab in patients with active psoriatic arthritis (PsA) who are naive of biologic disease-modifying anti-rheumatic drug (bDMARD) during a 52-week treatment period.

The study will consist of 3 periods:

- Period 1: Screening Period (Visit 1) up to 28 days before randomization (Visit 2)
- Period 2: Open-Label Treatment Period (Visit 2 through Visit 11) from Week 0 to Week 52
- Period 3: Post-Treatment Follow-Up Period occurring from the last treatment visit during Period 2 or Early Termination Visit (ETV) up to a minimum of 12 weeks after that visit

All patients randomized to ixekizumab will receive a starting dose of 160 mg at randomization (Visit 2 [Week 0]). Patients with moderate-to-severe plaque psoriasis will receive ixekizumab 80 mg every 2 weeks (Q2W) from Week 2 to Week 12 and every 4 weeks (Q4W) thereafter. Patients not meeting criteria for moderate-to-severe plaque psoriasis at randomization will receive ixekizumab 80 mg Q4W starting at Week 4.

Patients randomized to adalimumab with moderate-to-severe plaque psoriasis will receive a starting dose of 80 mg at randomization (Visit 2 [Week 0]) followed by 40 mg Q2W starting at Week 1. Patients not meeting criteria for moderate-to-severe plaque psoriasis will receive a starting dose of 40 mg at randomization (Visit 2) followed by 40 mg Q2W starting at Week 2 (see Section 7.1 of study protocol for details regarding treatments administered).

Figure RHCF.5.1 illustrates the study design.



Abbreviations: D = days; LTV = last treatment visit during Period 2 or Early Termination Visit; n = number of subjects; V = visit; W = week.

a See Section 7.1 of RHCF Study Protocol for dosing details.

Figure RHCF.5.1. Illustration of study design for Clinical Protocol I1F-MC-RHCF.

#### 5.2. Determination of Sample Size

Approximately 550 patients who meet all criteria for enrollment at Visits 1 and 2 will be randomized in a 1:1 ratio at Week 0 (Visit 2) in Period 2 to ixekizumab or adalimumab (275 patients per treatment group).

Sample size was calculated assuming the proportion of patients simultaneously achieving 50% improvement in American College of Rheumatology criteria (ACR50) and 100% improvement from baseline in Psoriasis Area and Severity Index criteria (PASI 100) as 13.6% and 31.3% in the adalimumab and ixekizumab treatment groups, respectively, as observed in the conventional synthetic disease-modifying anti-rheumatic drugs (csDMARD)-experienced population from Study I1F-MC-RHAP (RHAP). According to the nQuery software, a total sample size of 550 (ie, 275 per treatment group) using a 2-sided Fisher's exact test at 0.05 level of significance would yield approximately 99% power for testing ixekizumab versus adalimumab.

This sample size would yield 78% power for testing the noninferiority of ixekizumab to adalimumab at a 1-sided 0.025 level of significance based on a noninferiority margin of -12% and using ACR50 response rates of 43.8% and 44.1% as observed for the ixekizumab and adalimumab treatment groups, respectively, in the csDMARD-experienced population from Study RHAP. For testing superiority of ixekizumab to adalimumab based on PASI 100 response rates of 46.9% and 23.7% as observed for ixekizumab and adalimumab in the csDMARD-experienced population from Study RHAP, this sample size would yield approximately 99% power using a 2-sided Fisher's exact test at 0.05 level of significance.

#### **5.3.** Method of Assignment to Treatment

Patients who meet all Visit 1 and Visit 2 eligibility criteria for enrollment will be randomized at Visit 2 (Week 0) in a 1:1 ratio to open-label treatment with ixekizumab or adalimumab at Week 0 (Visit 2). Assignment to treatment groups will be determined by a computer-generated random sequence using an interactive web-response system (IWRS). The IWRS will be used to assign investigational product to each patient. Site personnel will confirm that they have located the correct investigational product by entering a confirmation number found on the investigational product into the IWRS. The randomization will be stratified by concomitant csDMARD use at baseline (Yes, No) and moderate-to-severe plaque psoriasis involvement (Yes, No).

#### 6. A Priori Statistical Methods

#### 6.1. General Considerations

This plan describes a priori statistical analyses that will be performed. Statistical analysis of this study will be the responsibility of Eli Lilly and Company (hereafter Lilly). The statistical analyses will be performed using SAS® Version 9.2 or higher. Lilly will be responsible for producing the tables, figures, and listings, unless otherwise specified. All tables, figures, and listings will be checked independently for consistency and integrity by Lilly. This analysis plan also includes exploratory analyses that are intended to be produced separately from the clinical study report (CSR) outputs, as noted below.

Additional efficacy, health outcomes, and safety analyses for Health Technology Assessment (HTA) purposes will be described in a separate document, and results will be reported separately from the CSR.

Continuous data will be summarized in terms of the number of observations, mean, standard deviation (SD) and/or standard error of the mean (SEM), if applicable, median, minimum, and maximum. The minimum and maximum will be reported to the same number of decimal places as the raw data recorded in the database. The mean and median will be reported to 1 more decimal place than the raw data recorded in the database. The SD and SEM will be reported to 2 more decimal places than the raw data. In general, the maximum number of decimal places reported shall be 4 for any summary statistic.

Categorical data will be summarized in terms of the number of patients in the analysis population, the number of patients with non-missing data at the relevant time point, frequency counts, and the percentages based on the appropriate method. Percentages will be presented to 1 decimal place. Percentages will not be presented for zero counts.

Change from baseline will be calculated as the post-baseline value minus the baseline value. Percent change from baseline is defined as (100 x [post-baseline – baseline]/baseline). Percent improvement from baseline is calculated as the positive percent change from baseline if a higher value at post-baseline means improvement from baseline. Similarly, percent improvement from baseline is calculated as the negative percent change from baseline if a lower value at post-baseline means improvement from baseline. If the baseline value is missing for a particular variable, then the change from baseline and the percent improvement from baseline will not be calculated.

Data collected at early termination visits will be mapped to the next planned visit number for that patient. For by-visit summaries, only visits in which a measure was scheduled to be collected will be summarized. Unplanned/unscheduled measurements will be excluded from the mixed-effects model of repeated measures (MMRM) analysis. However, the data will still be used in other analyses; such analyses include, but are not limited to, shift analyses and modified baseline observation carried forward (mBOCF) endpoint analyses.

All confidence intervals (CIs) and statistical tests will be 2-sided with an  $\alpha$  level of 0.05 unless specified otherwise. P-values that are greater than or equal to 0.001, and less than or equal to 0.999, will be presented to 3 decimal places. All other p-values that are less than 0.001 will be presented as <0.001, while p-values greater than 0.999 will be presented as >0.999. Confidence intervals will be presented to 1 more decimal place than the raw data.

Age, sex, and race will be reported on all by-patient listings unless otherwise specified. Sex will be abbreviated as follows: female (F) and male (M). Race will be abbreviated as follows: American Indian or Alaska Native (AI), Asian (AS), Black or African American (BL), Native Hawaiian or other Pacific Islander (NH), White (WH), and Multiple (MU).

Table RHCF.6.1 gives the treatment groups to be displayed for each treatment period and analysis population. Analysis populations are defined in Section 6.1.3. Note: "IXE" and "ADA" will be included in treatment group names for ixekizumab and adalimumab, respectively, in the statistical reports where applicable.

Table RHCF.6.1. Treatment Groups for Each Treatment Period and Analysis Population

| Treatment<br>Period | Analysis<br>Population | Treatment Groups | Abbreviation | Comparison |
|---|---|---|---|---|
| Open-Label<br>Treatment Period<br>(Period 2) | Intent-to-Treat Population; Safety Population | Ixekizumab 80 mg Q4W (or Q2W/Q4W) | IXE | IXE vs ADA |
| | | Adalimumab 40 mg Q2W | ADA | |
| Post-Treatment<br>Follow-up Period<br>(Period 3) <sup>a</sup> | Follow-up<br>Population | Ixekizumab 80 mg Q4W<br>(or Q2W/Q4W) | IXE | Not applicable |
| | | Adalimumab 40 mg Q2W | ADA | |

Abbreviations = ADA = adalimumab; IXE = ixekizumab; O2W = every 2 weeks; O4W = every 4 weeks.

# 6.1.1. General Considerations for the Open-Label Treatment Period (Period 2)

Baseline will be defined as the last available value on or prior to the first injection of the study drug for both efficacy, health outcomes, and safety analyses. In most cases, this will be the measurement recorded at Week 0 (Visit 2).

Categorical and continuous data will be summarized as described in Section 6.1.

<sup>&</sup>lt;sup>a</sup> Treatment group refers to the dosage regimen that the patient received immediately prior to entering the Post-Treatment Follow-up Period.

Comparisons of ixekizumab versus adalimumab will be performed for all outcome variables in Period 2, as deemed appropriate, using methods described in Section 6.2.

Safety will be assessed by summarizing and analyzing adverse events (AEs), laboratory analytes including neutrophil counts, vital signs, and concomitant medications. The duration of exposure will also be summarized.

# 6.1.2. General Considerations for the Post-Treatment Follow-Up Period (Period 3)

Unless otherwise specified, the baseline for the safety analyses in Period 3 is defined as the last nonmissing assessment on or prior to entering Period 3, that is on or prior to Week 52 (Visit 11) or ETV.

The categorical safety measures will be summarized with incidence rates. The mean change of the continuous safety measures will be summarized by visits.

#### 6.1.3. Analysis Populations

The follow analysis populations will be used:

**Intent to Treat Population (ITT):** The ITT Population consists of all randomized patients. Even if the patient does not take the assigned treatment, does not receive the correct treatment, does not receive any medication, or otherwise does not follow the protocol, the patients will be analyzed according to the treatment to which they were assigned at Week 0. Unless otherwise specified, all efficacy and health outcomes analyses for the Open-Label Treatment Period (Period 2) will be conducted on the ITT population.

**Safety Population:** The Safety Population is defined as all randomized patients who received at least 1 dose of study treatment. Patients will be analyzed according to the treatment to which they were assigned at Week 0. Unless otherwise specified, all safety analyses for the Open-Label Treatment Period will be conducted on the Safety Population.

**Post-Treatment Follow-Up Population**: The Post-Treatment Follow-Up Population consists of all randomized patients who received at least 1 dose of study treatment during Period 2 and have entered the Post-Treatment Follow-Up Period. Safety analyses for Period 3 (Post-Treatment Follow-Up Period) will be conducted on this population. Patients will be analyzed according to the last treatment they received before entering Period 3 (see treatment groups defined in Table RHCF.6.1).

Table RHCF.6.2 gives the description of each of the population sets in the study as well as their intended analysis purposes.

Table RHCF.6.2. Efficacy, Health Outcomes, and Safety Measures Summarized and/or Analyzed for Each Analysis Population

| Population Name | Measurement Summarization of Population |
|---|---|
| All Patients Entered | Tables for patient allocation and analysis populations, patient |
| | disposition |
| Intent-to-Treat Population | Tables, listings and/or figures for the following: patient disposition, |
| | important protocol deviations, patient characteristics, historical |
| | diagnoses, pre-existing conditions, previous therapies, concomitant |
| | medications, primary and secondary efficacy measures, health |
| | outcomes, exploratory measures for the Open-Label Treatment Period |
| | (Period 2) |
| Safety Population | Tables, listings and/or figures for safety assessments, treatment |
| | compliance, duration of exposure for the Open-Label Treatment Period |
| | (Period 2) |
| Follow-Up Population | Tables, listings and/or figures for the following: patient disposition, |
| | concomitant medications, and safety assessments for the Post-Treatment |
| | Follow-Up Period (Period 3) |

#### 6.2. Analysis Methods

#### 6.2.1. Categorical

Unless specified otherwise, the primary analysis method for the binary categorical efficacy and health outcome variables will be a logistic regression model with treatment, concomitant csDMARD use at baseline, and moderate-to-severe plaque psoriasis involvement as factors. The odds ratios and the corresponding 95% CIs will be reported. Fisher's exact test will be used as the secondary analysis method.

For ordinal categorical variables, a logistic regression model using cumulative logits will be used.

Treatment differences (Absolute Risk Reductions [ARR]), Relative Risks (RR), Numbers Needed to Treat (NNT) estimates, and their corresponding 95% CIs (using normal approximation) will also be reported. See Appendix 1 for more details.

The statistical methodology for assessing noninferiority of ixekizumab to adalimumab for ACR50 is described in Section 6.7.

# 6.2.2. Continuous Endpoints

Unless specified otherwise, the primary analysis method for all continuous efficacy and health outcome variables will be a MMRM analysis. The model will include treatment group, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, visit-as-fixed factors, baseline value as covariate and baseline-by-visit and treatment-by-visit interaction terms. The MMRM analyses will be conducted using a restricted maximum likelihood (REML)-based repeated measures approach. The covariance structure to model the within-patient errors will be unstructured. If the unstructured covariance matrix results in a lack

of convergence, the heterogeneous Toeplitz covariance structure, followed by the heterogeneous autoregressive covariance structure, followed by the compound symmetry structure will be used. The first structure to yield convergence will be used for inference. The Newton-Raphson with ridging optimization technique will be used to aid with convergence. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom and adjust standard errors. Type III tests for the least squares (LS)Means will be used for the statistical comparison; the 95% CI will also be reported.

An analysis of covariance (ANCOVA) model and mBOCF imputation method as detailed in Section 6.4.2 will be used as the secondary analysis method for treatment comparisons on continuous efficacy and health outcome variables. The ANCOVA model will include treatment, concomitant csDMARD use at baseline, moderate-to-severe plaque psoriasis involvement, and baseline value in the model. Type III sums of squares for the LSMeans will be used for the statistical comparison; the 95% CI will be reported.

#### 6.3. Adjustments for Covariates

The randomization at the beginning of Open-Label Treatment Period (Period 2) is stratified by concomitant csDMARD use at baseline (Yes, No) and moderate-to-severe plaque psoriasis involvement (Yes, No). Unless otherwise specified, all efficacy and health outcome analyses during Period 2 will include the concomitant csDMARD use at baseline and moderate-to-severe plaque psoriasis involvement in the model. In general, when an MMRM is to be used for analyses, baseline value and baseline-by-visit interactions will be included as covariates; when an ANCOVA is to be used for analyses, baseline value will be included as a covariate.

The OBSMARGINS/OM option will be used in the LSMEANS statement in SAS to account for imbalance in the stratification variables.

## 6.4. Handling of Dropouts or Missing Data

# 6.4.1. Non-Responder Imputation (NRI) for Clinical Response

Analysis of categorical efficacy and health outcome variables will be based on treatment success/failure. This approach yields results numerically identical to non-responder imputation (NRI), but it is interpreted differently. Patients will be considered treatment failures (or non-responders) if they do not meet the clinical response criteria or have missing clinical response data at a particular time point of analysis.

# 6.4.2. Modified Baseline Observation Carried Forward (mBOCF)

Missing data for continuous efficacy and health outcomes variables will be imputed using a mBOCF method. For patients discontinuing investigational product due to an AE, including death, the baseline observation will be carried forward to the corresponding primary endpoint for evaluation. For patients discontinuing investigational product for any other reason, the last non-missing post-baseline observation before discontinuation will be carried forward to the corresponding time point of evaluation. Randomized patients without at least 1 post-baseline

observation will not be included for evaluation with the exception of patients discontinuing study treatment due to an AE (including death).

# 6.4.3. Missing Data Imputation for Adverse Event and Concomitant Medication Dates

If a medication date (prior therapy or concomitant medication) or event (historical event, preexisting condition, or AE) date is completely or partially missing, the following imputation rules should be utilized in the analysis unless otherwise stated:

- For the start date:
  - o If year, month, and day are missing, then use the earlier of the patient's first visit date or the consent date.
  - o If either month or month and day are missing, then use January 1.
  - o If only day is missing, impute the first day of the month.
  - o The imputed date should not be before the minimum of the patient's first visit or consent date.
- For the start time:
  - o Impute as 23:59.
- For the end date:
  - o If year, month, and day are missing, then use the patient's last visit date.
  - o If either month or month and day are missing, then use December 31.
  - o If only day is missing, then use the last day of the month.
  - o The imputed date should not be beyond the patient's last visit date.
- For the end time:
  - o Impute as 23:59.

If there is any doubt for the start and end date/times for events, the event will be flagged as treatment-emergent or follow-up emergent according to the corresponding study period. If a follow-up emergent event was already counted as treatment-emergent during the prior treatment period, it will not be counted as a follow-up emergent event. For medications, the medication will be flagged as concomitant.

#### 6.5. Multicenter Studies

This study will be conducted by multiple investigators at multiple sites internationally. The primary endpoint at Week 24 will be summarized by sites using descriptive statistics only.

# 6.6. Multiple Comparisons/Multiplicity

A multiple testing procedure for the primary and major secondary endpoints will be implemented to control the family-wise type I error rate at a 2-sided  $\alpha$  level of 0.05. The primary and major secondary endpoints will be sequentially tested in the following order to compare ixekizumab versus adalimumab, using the primary analysis method.

- 1. Test 1 for Primary Endpoint Proportion of patients simultaneously achieving ACR50 and PASI 100 at Week 24: A superiority test of the primary endpoint will be performed at an overall 2-sided  $\alpha = 0.05$  using the methods described in Section 6.2.1.
- 2. Test 2 for Major Secondary Endpoint #1 Proportion of patients achieving ACR50 at Week 24: If the test for the primary endpoint is significant, then a noninferiority test for the major secondary endpoint #1 will be performed using the methods described in Section 6.7.
- 3. Test 3 for Major Secondary Endpoint #2 Proportion of patients achieving PASI 100 at Week 24: If the test for major secondary endpoint #1 is significant, then a superiority test for major secondary endpoint #2 will be performed using the methods described in Section 6.2.1.

If a test in this sequence is not significant, all subsequent tests will be considered nonsignificant.

There will be no adjustment for multiple comparisons for any other analyses.

### 6.7. Methodology for Noninferiority Test

For assessing noninferiority of ixekizumab to adalimumab, missing data will be imputed using the NRI method. Noninferiority analysis will be performed on the ITT population using a prespecified fixed margin approach. There is no universally accepted value for what is considered to be a clinically unimportant difference between 2 treatments for a particular efficacy measure. We will consider the points from EMEA Committee for Medicinal Products for Human Use (CHMP) (CHMP 2005) and FDA guidance (2016) which state that an appropriate noninferiority margin should be based on both clinical and statistical grounds.

The null hypothesis will be rejected if the lower bound of the 2-sided 95% CI for the difference in proportions of responders on ixekizumab minus adalimumab is greater than the prespecified margin, meaning ixekizumab will be deemed noninferior to adalimumab. If the lower bound of the CI exceeds 0 (the corresponding p-value from the logistic regression model will also be produced), and ixekizumab will be deemed superior to adalimumab based on the p-value. The 95% CIs for the difference in proportions will be calculated using the simple asymptotic method, without continuity correction (that is, normal approximation to the binomial distribution).

Based on EMEA CHMP (CHMP [WWW]), FDA guidance (FDA [WWW]), and Weinblatt et al. (2013), a noninferiority margin of -12.0% for ACR50 between ixekizumab and adalimumab (ie, response rate of ixekizumab – response rate of adalimumab) is considered appropriate. This noninferiority margin represents an approximately 50% preservation of the adalimumab treatment effect (based on the difference between adalimumab and placebo) observed in a historical Phase 3 study for adalimumab 40 mg twice weekly compared with placebo (Mease et al. 2005) and Study RHAP (Mease et al. 2016).

# 6.8. Patient Disposition

Patient flow will be summarized from entered to randomized to completion, and analysis populations will be listed and summarized by treatment group.

The following patient disposition summaries will be provided for Open-Label Treatment Period (Period 2):

- The number and percentage of patients in the ITT population completing the Open-Label Treatment Period or prematurely discontinuing from the Open-Label Treatment Period, by treatment group and primary reason for discontinuation.
  Fisher's exact test will be used to test for treatment differences between treatment groups in the percentage of patients discontinuing from the Open-Label Treatment Period, and in the percentage of patients discontinuing for each reason.
- The number and percentage of patients in the ITT population completing the Open-Label Treatment Period or prematurely discontinuing from the Open-Label Treatment Period, by treatment group, visit, and primary reason for discontinuation.
- The time to discontinuation from the Open-Label Treatment Period due to any reason (in weeks).

Time to discontinuation due to any reason (in weeks) and due to an AE (in weeks) will be summarized graphically for the ITT population by treatment group using Kaplan-Meier techniques. The time to discontinuation (in weeks) from the Open-Label Treatment Period will be calculated as:

(Date of discontinuation from Open-Label Treatment Period – Date of randomization + 1)/7

Patients completing the Open-Label Treatment Period will be censored at the date of completion (ie, the date of Visit 11 [Week 52]). Patients without a date of Open-Label Treatment Period completion or discontinuation will be censored at the last nonmissing date out of the following dates: date of last dose and date of last study visit up to and including Visit 11 (Week 52) (scheduled or unscheduled). Descriptive statistics including 25th percentile, median, 75th percentile, and corresponding 95% CIs, as well as probability of discontinuation by Week 52 will be summarized by treatment group. The log-rank test will be used to test for differences in the time to discontinuation between the treatment groups.

The following patient disposition summary will be provided for the Post-Treatment Follow-Up Period (Period 3):

• The number and percentage of patients in the Post-Treatment Follow-Up Population completing each follow-up visit or prematurely discontinuing from the Post-Treatment Follow-Up Period, by treatment group, visit, and primary reason for discontinuation.

Patient allocation by region, country, and center/site will be summarized with number of patients who entered the study, number of ITT patients for each treatment group, number of patients discontinued from study treatment, and number of patients discontinued from study.

#### 6.9. Patient Characteristics

#### 6.9.1. Demographics and Baseline Characteristics

Demographic variables and baseline characteristics (including baseline clinical measures) will be summarized for the ITT population. For weight, body mass index (BMI), tobacco use and alcohol consumption, baseline is defined in the same manner as the safety baseline (as defined in Section 6.15).

The continuous variables will be summarized using descriptive statistics, and the categorical variables will be summarized using frequency counts and percentages. The comparisons among treatment groups will be conducted using an ANOVA model with treatment as a factor for continuous data and using a Fisher's exact test for categorical data. (For categorical variables that have more than 2 categories, Monte Carlo estimates of exact p-values will be used.)

The demographic variables to be presented include the following:

- Age (in years)
- Age group: <65 years or  $\ge 65$  years
- Sex
- Age group within sex
- Ethnicity: Hispanic or Latino, Non-Hispanic and Non-Latino
- Race
- Country
- Geographic Regions:
  - o Europe, Rest of the World
- Height (cm)
- Weight (kg)
- Weight category: <100 kg or ≥100 kg
- Weight category:  $<80 \text{ kg}, \ge80 \text{ kg}$  and <100 kg, or  $\ge100 \text{ kg}$
- Body mass index (BMI, kg/m<sup>2</sup>)
- Body mass index category (underweight (<18.5 kg/m²); normal (≥18.5 and <25 kg/m²); overweight (≥25 and <30 kg/m²); obese (≥30 and <40 kg/m²); or extremely obese (≥40 kg/m²)</li>
- Tobacco use: never, current, or former
- Alcohol use: never, current, or former
- Other baseline characteristics to be presented include the following:
  - o Time since PsA onset (years) calculated as

 $(date\ of\ informed\ consent-date\ of\ PsA\ onset+1)/365.25$ 

Patients who have a completely missing date of onset will have a missing value for the time since PsA onset, otherwise, "January" and "01" will be imputed for the missing month and day, respectively, in cases where these 2 date components are missing.

o Time since PsA diagnosis (years) – calculated as

Patients who have a completely missing date of diagnosis will have a missing value for the time since diagnosis, otherwise "January" and "01" will be imputed for the missing month and day, respectively, in cases where these 2 date components are missing.

- o Time since PsA onset (years): <5 or ≥5
- Time since PsA diagnosis (years):  $\leq 2$  or  $\geq 2$
- Time since psoriasis (Ps) onset (years) calculated as

(date of informed consent – date of Ps onset + 1) 
$$/ 365.25$$

Patients who have a completely missing date of onset will have a missing value for the time since Ps onset, otherwise, "January" and "01" will be imputed for the missing month and day, respectively, in cases where these 2 date components are missing.

• Time since Ps diagnosis (years) – calculated as

Patients who have a completely missing date of diagnosis will have a missing value for the time since diagnosis, otherwise "January" and "01" will be imputed for the missing month and day, respectively, in cases where these 2 date components are missing.

- Tender Joint Counts (TJC) based on 68 joints
- Swollen Joint Counts (SJC) based on 66 joints
- Physician's global assessment of disease activity (mm)
- Patient's Global Assessment (PatGA) of Disease Activity (mm)
- Patient's assessment of joint pain (mm)
- Health Assessment Questionnaire–Disability Index (HAQ-DI) total score
- C-reactive protein (CRP) (mg/L)
- CRP categories;  $>6 \text{ mg/L or } \le 6 \text{ mg/L}$
- Rheumatoid Factor Positive (RF+); yes or no
- Disease Activity Score-C-Reactive Protein (DAS28-CRP)
- DAS28-CRP; <2.6,  $\ge 2.6$  and <3.2,  $\ge 3.2$  and <5.1,  $\ge 5.1$
- Enthesitis (LEI >0); yes or no
- Enthesitis (SPARCC >0); yes or no
- Leeds Enthesitis Index (LEI) for patients with baseline enthesitis (LEI >0)
- Spondyloarthritis Research Consortium of Canada (SPARCC) for patients with baseline enthesitis (SPARCC >0)
- Dactylitis (LDI-B score >0); yes or no
- Leeds Dactylitis Index Basic (LDI-B) for patients with baseline dactylitis (LDI-B score >0)

- Modified CPDAI without the spinal disease assessment (Ankylosing Spondylitis Quality of Life Questionnaire [AsQoL] and BASDAI)
- Psoriasis Area and Severity Index (PASI) total score
- PASI total score:  $\langle 12, \geq 12 \rangle$
- Static Physician Global Assessment of Psoriasis (sPGA) score
- sPGA score:  $\langle 3, \rangle 3$
- Moderate to Severe Psoriasis (defined as PASI  $\geq$ 12, sPGA  $\geq$ 3, and BSA  $\geq$ 10); yes or no
- Percentage of Body Surface Area (BSA)
- BSA: <10%, ≥10%
- Itch Numeric Rating Scale (Itch NRS) score
- Itch NRS score; 0, >0 and  $\le 3, >3$
- Nail Psoriasis (NAPSI > 0): yes or no
- Nail Psoriasis Severity Index (NAPSI) score for patients with baseline fingernail involvement (NAPSI >0)
- Fatigue Severity Numeric Rating Scale (Fatigue NRS) score
- SF-36 Physical Component Summary score
- SF-36 Mental Component Summary score
- Dermatology Life Quality Index (DLQI) total score
- Columbia Suicide Severity Rating Scale (C-SSRS)
- Self-Harm Supplement Form
- Self-Harm Follow-Up Form
- Concomitant Glucocorticoids use at baseline; yes or no
- Concomitant Glucocorticoids mean daily dose at baseline
- Concomitant Methotrexate use at baseline; yes or no
- Concomitant Methotrexate mean weekly dose at baseline
- Concomitant Conventional disease-modifying antirheumatic drugs (csDMARD) use at baseline; yes or no
- Number of prior csDMARD therapies: 1, 2, 3, or >3
- European Quality of Life 5 dimensions 5 level (EQ-5D 5L)
- Latent TB; yes or no.

By-patient listings of demographic and baseline characteristics, respectively, for the ITT population will be provided.

## 6.9.2. Previous Therapy for Psoriatic Arthritis

The number and percentage of patients who received previous therapy for PsA (as recorded on the *Previous Therapy: Psoriatic Arthritis* electronic case report form [eCRF] page) will be summarized by treatment group, overall, and preferred name. The number and percentage of patients with each reason for discontinuing previous therapy for PsA will also be presented by treatment group.

Previous therapy for PsA will be summarized for the ITT population.

Treatment group comparisons for the ITT population will be conducted using Fisher's exact test.

Listing of previous therapy for PsA will be provided for the ITT population.

#### 6.9.3. Historical Illness and Pre-existing Conditions

Historical illnesses and pre-existing conditions will be classified using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) dictionary. Historical illness/condition is defined as the condition/event recorded on the *Pre-Existing Conditions and Medical History* eCRF page or on the *Prespecified Medical History* eCRF page with an end date prior to the date of informed consent. Pre-existing conditions for the Open-Label Treatment Period (Period 2) are defined as those conditions recorded on the *Pre-Existing Conditions and Medical History* eCRF page or on the *Prespecified Medical History* eCRF pages with a start date prior to the date of informed consent, and no end date (ie, the event is ongoing) or an end date after the date of informed consent. Adverse events occurring prior to the date of first study injection will also be reported for the open-label treatment period (Period 2). If a pre-existing condition worsens in severity on or after the date of informed consent, it will be considered an AE from the date of worsening onwards. Patients will only be counted once, regardless of how many conditions are included under the same System Organ Class (SOC) and Preferred Term (PT).

The number and percentage of patients with historical illnesses, pre-existing conditions and adverse events occurring prior to the first dose will be provided by treatment group, overall, and by SOC and PT for the Open-Label Treatment Period for the ITT population. For condition/event that is gender specific (as defined by MedDRA), the denominator and computation of the percentage will include only patients from the given gender.

Treatment group comparisons for ITT population will be conducted using Fisher's exact test.

Listing of historical illnesses and pre-existing conditions will be provided for ITT population.

# 6.10. Treatment Compliance

Study treatment dispensed will be listed (including the CT Lot number) for all entered patients. Study treatment administration and compliance will be listed for all entered patients.

Patients will record information in a Study Drug Administration Log (captured in the *Exposure* eCRF page), including the date, time, and anatomical location of administration of investigational product, syringe number, who administered the investigational product, and the reason if the investigational product was not fully administered.

Treatment compliance (%) for each patient will be calculated as:

$$100 \times \frac{Total\ number\ of\ injections\ administered}{Total\ number\ of\ injections\ prescribed}$$

• Number of injections prescribed (that is, expected) is 17 injections for patients on ixekizumab with moderate-to-severe plaque psoriasis. Patients will receive 2 ixekizumab 80 mg injections at Week 0, 1 ixekizumab 80 mg injection every 2 weeks from Week 2 to Week 12, and 1 ixekizumab 80 mg injection every 4 weeks from Week 16 to Week 48.

- Number of injections prescribed (that is, expected) is 14 injections for patients on ixekizumab without moderate-to-severe plaque psoriasis. Patients will receive 2 ixekizumab 80 mg injections at Week 0 and 1 ixekizumab 80 mg injection every 4 weeks from Week 4 to Week 48.
- Number of injections prescribed (that is, expected) is 28 injections for patients on adalimumab with moderate-to-severe plaque psoriasis. Patients will receive 2 adalimumab 40 mg injections at Week 0 and 1 adalimumab 40 mg injection every 2 weeks from Week 1 to Week 51.
- Number of injections prescribed (that is, expected) is 26 injections for patients on adalimumab without moderate-to-severe plaque psoriasis. Patients will receive 1 adalimumab 40 mg injection every 2 weeks from Week 0 to Week 50.
- For patients who discontinue during Period 2, the number of injections prescribed can be derived from the IWRS study drug dispense dataset.
- The total number of injections administered will be derived using the response to the question, "Was dose administered?" on the *Exposure* eCRF page.

Overall compliance for the Open-Label Treatment Period will be considered if the patient misses no more than 20% of the expected doses, does not miss 2 consecutive doses, and does not overdose (that is, take more injections at the same time point than specified in the protocol) within the study period.

Treatment compliance with investigational product will be summarized for the Open-Label Treatment Period (ITT population).

Treatment group comparisons will be conducted for the ITT population using a Fisher's exact test.

# 6.11. Concomitant Therapy

Medications will be classified into anatomical therapeutic chemical (ATC) drug classes using the latest version of the World Health Organization (WHO) drug dictionary.

Medication start and stop dates will be compared to the date of first dose of treatment in the treatment period to allow medications to be classified as either Prior or Concomitant for the Open-Label Treatment Period and Post-Treatment Follow-Up period.

Prior medications are those medications that start and stop prior to the date of first dose of treatment in corresponding treatment period. Concomitant therapy for Period 2 is defined as a therapy that starts before, on, or after the first day of study treatment in Period 2 and before the last visit date in Period 2 and continues into Period 2, that is, either no end date (the therapy is ongoing) or an end date on or after the first day of study treatment in Period 2. Note that a concomitant therapy will belong to Period 2 if the therapy starts and ends on the exact same day as the first day of study treatment in Period 2. Concomitant therapy for the Post-Treatment Follow-Up Period (Period 3) is defined as a therapy that starts before, on, or after the last visit date in Period 2 and continues into Period 3, that is, either no end date (the therapy is ongoing) or

an end date after the last visit date in Period 2. A concomitant therapy will belong to Period 2 if the therapy starts and ends on the exact same day as the last visit date in Period 2.

Concomitant therapies and prior therapies will both be summarized for the following periods and populations:

- Open-Label Treatment Period (ITT Population)
- Post-Treatment Follow-Up Period (Post-Treatment Follow-Up Population).

The comparisons will be conducted using Fisher's exact test.

The following summaries will be provided:

Concomitant therapy by WHO ATC Level 4 and WHO PT

A by-patient listing of all concomitant and prior medications will be provided for the ITT Population.

## 6.12. Efficacy Analyses

Table RHCF.6.3 includes the description and derivation of the primary and secondary efficacy outcomes.

Table RHCF.6.4 provides the detailed analyses including analysis type, method and imputation, population, time point, and comparisons for primary and secondary efficacy analyses.

 Table RHCF.6.3.
 Description and Derivation of Primary and Secondary Efficacy Outcomes

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| American College of | A composite of clinical, laboratory, | ACR20/50/70 | See Appendix 2 for details. | See Appendix 2 for details. |
| Rheumatology | and functional measures in PsA to | Time to first ACR20/50/70 | | |
| (ACR) Responder | assess relief of signs and symptoms; | response | | |
| Index | responses are presented as the minimal | | | |
| | numeric disease assessment criteria. | | | |
| Psoriasis Area and | For patients with plaque psoriasis, | PASI total score | The composite PASI score is | If any individual score is |
| Severity Index | combines assessments of the extent of | Total PASI score $\leq 1$ , $\leq 2$ , or | calculated by multiplying the | missing, the PASI score will |
| (PASI) | body-surface involvement in 4 | _≤3 | sum of the individual-severity | not be calculated, hence |
| | anatomical regions (head and neck, | | scores for each area by the | missing. |
| | trunk, arms, and legs) and the severity | | weighted area-of-involvement | |
| | of scaling (S), redness (R), and plaque | | score for that respective area, | |
| | induration/infiltration thickness (T) in | | and then summing the 4 | |
| | each region, yielding an overall score | | resulting quantities as follows: | |
| | of 0 for no psoriasis to 72 for the most | | $PASI = 0.1(R_h + T_h + S_h)A_h +$ | |
| | severe disease (Fredriksson and | | $0.2(R_u + T_u + S_u)A_u + 0.3(R_t + T_t)$ | |
| | Pettersson 1978). Severity is rated for | | $+ S_t)A_t + 0.4(R_1 + T_1 + S_1)A_1$ | |
| | each index (R, S, T) on a 0-4 scale (0 | | Where, | |
| | for no involvement; up to 4 for very | | $R_h$ , $R_u$ , $R_t$ , $R_l$ = redness score of | |
| | severe involvement): | | plaques on the head, upper limb, | |
| | 0 = none | | trunk, and lower limb, scored 0-4 | |
| | 1 = slight | | respectively; | |
| | 2 = moderate | | $T_h$ , $T_u$ , $T_t$ , $T_l$ = thickness score of | |
| | 3 = severe | | plaques on the head, upper limb, | |
| | 4 = very severe | | trunk, and lower limb, scored 0-4 | |
| | The body is divided into 4 anatomical | | respectively; | |
| | regions comprising the head (h), upper | | $S_h$ , $S_u$ , $S_t$ , $S_l$ = scaliness score of | |
| | limb (u), trunk (t), and lower limb (l). | | plaques on the head, upper limb, | |
| | In each of these areas, the fraction of | | trunk, and lower limb, scored 0-4 | |
| | total BSA affected is graded on a 0-6 | | respectively; | |
| | scale (0 for no involvement; up to 6 for | | $A_h$ , $A_u$ , $A_t$ , $A_l$ = numerical value | |
| | 90% to 100% involvement): | | translation of % area of psoriatic | |
| | 0 = 0% (clear) | | involvement score for the head, | |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | 1 = >0% to <10%<br>2 = 10% to <30%<br>3 = 30% to <50%<br>4 = 50% to <70%<br>5 = 70% to <90%<br>6 = 90% to 100% | | upper limb, trunk, and lower limb, respectively. PASI scores are treated as a continuous score, with 0.1 increments within these values. | |
| | The various body regions are weighted to reflect their respective proportion of BSA. | Change from baseline in PASI total score | Calculated as: observed PASI score – baseline PASI score | Missing is baseline or observed value is missing |
| | | • PASI 75/90/100 | Defined as at least 75%, 90%, or 100% improvement in PASI total score from baseline | Single item, missing if PASI total score is missing |
| ACR50 and PASI<br>100 | Patients who achieve ACR50 and PASI 100 simultaneously. | • Simultaneous ACR50 and PASI 100 | | Missing if either ACR score or PASI score is missing. |
| Percentage of Body<br>Surface Area (BSA) | The investigator will evaluate the percentage involvement of psoriasis on each patient's BSA on a continuous scale from 0% (no involvement) to | • BSA | Collected as a single item on the eCRF. Range from 0% to 100% | Single item, missing if missing. |
| | 100% (full involvement), in which 1% corresponds to the size of the patient's hand (including the palm, fingers, and thumb) (National Psoriasis Foundation [NPF] 2009). | Change from baseline in BSA | Calculated as: observed BSA – baseline BSA | Missing is baseline or observed value is missing |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| Nail Psoriasis Severity Index (NAPSI) NAPSI will be used if the patient has fingernail psoriasis at baseline. The NAPSI is a numeric, reproducible, objective tool for evaluation of fingernail psoriasis. This scale is used to evaluate the severity of fingernail bed psoriasis and fingernail matrix psoriasis by area of involvement in the fingernail unit. In this study, only fingernail involvement will be assessed. The fingernail is divided with imaginary horizontal and longitudinal lines into quadrants. Each | NAPSI score | The NAPSI score of a fingernail is the sum of scores in fingernail bed and fingernail matrix from each quadrant (maximum of 8). Each fingernail is evaluated, and the sum of all the fingernails is the total NAPSI score (range, 0 to 80), usually indicated as NAPSI score. | For each fingernail, if either the bed or matrix score is missing or not done, then the score for that finger is missing. If <50% of the finger scores from 10 fingers are missing, the imputation will be performed by using the average score of the remaining fingernails. If ≥50% of the finger scores are missing, the NAPSI score will be left as missing | |
| | fingernail is given a score for fingernail bed psoriasis (0-4) and fingernail matrix psoriasis (0-4), depending on the presence (score of 1) or absence (score of 0) of any of the features of fingernail bed and fingernail matrix psoriasis in each | Change from<br>baseline in NAPSI<br>score | Calculated as: observed<br>NAPSI – baseline NAPSI | Missing if baseline or observed value is missing |
| | quadrant: 0 = None 1 = present in one quadrant of nail 2 = present in two quadrants of nail 3 = present in three quadrants of nail 4 = present in four quadrants of nail | • NAPSI = 0 | NAPSI score equals to 0, indicating resolution of nail psoriasis. | Single item, missing if observed NAPSI score missing. |
| Tender Joint Count<br>(TJC) (68 joint<br>count) | The number of tender and painful joints will be determined by examination of 68 joints (34 joints on each side of the patient's body). The 68 joints to be assessed and classified | • TJC score | Adjusted sum of the painful/tender joints for all 68 joints: (sum of the evaluable individual joint | If more than half of the joint scores are nonevaluable, the total score will be missing. |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | as tender or not tender. | | scores)/(number of evaluable joints)×68 | |
| | | | See Appendix 3 for complete details. | |
| | | Change from baseline in TJC score | Calculated as: observed TJC score – baseline TJC score | Missing if baseline or observed value is missing |
| Swollen Joint Count<br>(SJC) (66 joint<br>count) | The number of swollen joints will be determined by examination of 66 joints (33 joints on each side of the patient's body). The 66 joints to be assessed and classified as swollen or not swollen. | SJC score | Adjusted sum of the swollen joints for all 66 joints: (sum of the evaluable individual joint scores)/(number of evaluable joints)×66 See Appendix 3 for complete details. | If more than half of the joint scores are nonevaluable, the total score will be missing. |
| | | Change from baseline in SJC score | Calculated as: observed SJC score – baseline SJC score | Missing if baseline or observed value is missing |
| Patient's<br>Assessment of Pain<br>Visual Analog Scale<br>(VAS) | Assesses the patient's current level of joint pain by marking a vertical tick on a 100-mm horizontal VAS. | Patient's pain VAS score | Range: 0 to 100 mm 0 represents no joint pain 100 represents the worst joint pain | Single item, missing if missing |
| | | Change from baseline in patient's pain VAS score | Calculated as: observed patient's pain VAS- baseline patient's pain VAS | Missing if baseline or observed value is missing |
| Patient's Global<br>Assessment of<br>Disease Activity<br>Visual Analog Scale<br>(VAS) | Assesses the patient's overall assessment of his or her PsA activity by marking a 100-mm horizontal VAS. | Patient's global assessment VAS score | Range: 0 to 100 mm 0 represents no disease activity 100 represents extremely active disease activity | Single item, missing if missing |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | | Change from baseline in patient's global assessment VAS score | Calculated as: observed patient's global assessment VAS— baseline patient's global assessment VAS | Missing if baseline or observed value is missing |
| Physician's Global<br>Assessment of<br>Disease Activity<br>Visual Analog Scale<br>(VAS) | Overall assessment of the severity of the patient's current PsA activity using a 100-mm horizontal VAS. The investigator making the assessment must be a rheumatologist or medically | Physician's global<br>assessment VAS<br>score | Range: 0 to 100 mm 0 represents no disease activity 100 represents extremely active disease activity | Single measure, missing if missing. |
| | qualified physician. | Change from baseline in physician's global assessment VAS score | Calculated as: observed<br>physician's global assessment<br>VAS– baseline physician's<br>global assessment VAS | Missing if baseline or observed value is missing |
| Patient's Assessment of Physical Function Health Assessment Questionnaire— Disability Index (HAQ-DI) | Patient-reported standardized questionnaire that is commonly used in PsA to measure disease-associated disability (assessment of physical function). It consists of 24 questions referring to 8 domains: dressing/grooming, arising, eating, | HAQ-DI score | Sum of the highest sub-<br>category scores within 8<br>categories and adjusted for<br>aids/devices and/or help from<br>another person.<br>See Appendix 4 for complete<br>details. | The patient must have a score for at least 6 of the 8 domains. If there are <6 domains completed, a HAQ-DI will be missing. |
| | walking, hygiene, reach, grip, and other daily activities | Change from baseline in HAQ-DI score HAQ-DI | Calculated as: observed HAQ-DI score—baseline HAQ-DI score Change from baseline < -0.35 | Missing if baseline or observed value is missing Missing if baseline or |
| | | improvement ≥0.35 | in HAQ-DI score | observed value is missing |
| C-Reactive Protein (CRP) | The ACR Core Set measure of acute phase reactant. It will be measured with a high sensitivity assay at the central laboratory to help assess the effect of ixekizumab on the patient's PsA. | • CRP (mg/L) | Raw laboratory result, no derivation will be applied with the exception of converting the units to mg/L when the results are reported in units other than mg/L | Single lab measure, missing if missing |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | | Change from baseline in CRP (mg/L) | Calculated as: observed CRP – baseline CRP | Missing if baseline or observed value is missing |
| Psoriatic Arthritic<br>Response Criteria<br>(PsARC) | PsARC is a composite criteria reported in terms of the percentage of patients achieving response according to the following criteria: PGA, PatGA, TJC, and SJC. Overall response is defined by improvement from the baseline assessment in 2 of the 4 criteria, 1 of which must be a joint count; there must not be worsening in any of the 4 criteria: At least 30% reduction in TJC At least 30% reduction in SJC At least a 1-point reduction in physician's assessment At least a 1-point reduction in patient's assessment The PsARC response was modified in this study by using the PGA and the PatGA on a 100-mm VAS instead of a 5-point Likert scale in the original criteria. The results from the 2 VAS measures were assessed as a difference from baseline (in mm), and criteria 3 and 4, above, were changed to "at least a 20 mm reduction" (Clegg 1996). | PsARC | Overall response is defined by improvement from the baseline assessment in 2 of the 4 criteria, 1 of which must be a joint count; there must not be worsening in any of the 4 criteria: At least 30% reduction in TJC At least 30% reduction in SJC At least a 20-mm reduction in physician's assessment At least a 20-mm reduction in patient's assessment | If the patient achieves PsARC with the non-missing measures, then impute as achieving PsARC; otherwise, the result is missing. |
| Coates criteria for<br>Minimal Disease<br>Activity (MDA) (6<br>entheseal points) | Uses a composite of 7 key outcome measures (includes PASI) used in PsA to encompass all of the domains of the disease to measure the overall state of | Coates criteria for MDA (6 entheseal points) | Patients are classified as achieving Coates criteria for MDA (6 entheseal points) if they fulfill 5 of 7 outcome | If the patient achieves MDA with the non-missing measures, then impute as achieving MDA; otherwise, |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | a patients' disease (Coates et al. 2010a; Coates and Helliwell 2010b). The LEI is used to assess tender entheseal points. | | measures: TJC ≤1 SJC ≤1 PASI total score ≤1 or BSA ≤3 patient pain VAS score of ≤15 patient global assessment VAS score of ≤20 HAQ-DI score ≤0.5 | the result is missing. |
| | | | tender entheseal points (6<br>entheseal points) ≤1 | |
| Coates criteria for<br>Minimal Disease<br>Activity (MDA) (18<br>entheseal points) | Uses a composite of 7 key outcome measures (includes PASI) used in PsA to encompass all of the domains of the disease to measure the overall state of a patients' disease (Coates et al. 2010a; Coates and Helliwell 2010b). The LEI and SPARCC are used to assess tender entheseal points. | Proportion of patients<br>achieving Coates criteria for<br>MDA (18 entheseal points) | Patients are classified as achieving Coates criteria for MDA (18 entheseal points) if they fulfill 5 of 7 outcome measures: TJC ≤1 SJC ≤1 PASI total score ≤1 or BSA ≤3 patient pain VAS score of ≤15 patient global VAS score of ≤20 HAQ-DI score ≤0.5 tender entheseal points ≤1 (based on 18 entheseal points) | If the patient achieves MDA with the non-missing measures, then impute as achieving MDA; otherwise, the result is missing. |
| Leeds Enthesitis<br>Index (LEI) | For patients with enthesitis, an assessment that consists of 18 entheseal points is performed by site personnel. The LEI has been developed specifically for use in PsA | LEI score | Each of the 6 sites is assigned a score of 0 (absent) or 1 (present) and the results are added to produce a total score (range: 0-6). | If one or more of the 6 sites are missing, then set LEI score to missing. |
| | and measures enthesitis at 6 sites (lateral epicondyle [left and right], | Change from baseline in LEI | Calculated as: observed LEI score – baseline LEI score | Missing if baseline or observed value is missing |
| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | medial femoral condyle [left and right], and Achilles tendon insertion [left and right]) (Healy and Helliwell 2008). | • LEI score = 0 | LEI score equals to 0, indicating complete resolution in enthesitis. | Missing if observed value are missing |
| Spondyloarthritis Research Consortium of Canada (SPARCC) | If the patient has enthesitis, the SPARCC will be administered by a blinded assessor. The SPARCC enthesitis index evaluates tenderness in a total of 16 enthesitis sites: the greater trochanter (right/left [R/L]), | SPARCC enthesitis score | Tenderness at each site is quantified on a dichotomous basis: 0 = nontender and 1 = tender. The results from each site are then added to produce a total score (range 0 to 16). | If 1 or more sites are missing, then set to missing. |
| | quadriceps tendon insertion into the patella (R/L), patellar ligament insertion into the patella and tibial tuberosity (R/L), Achilles tendon insertion (R/L), plantar fascia insertion (R/L), medial and lateral epicondyles (R/L), and the supraspinatus insertion (R/L) (Mease 2011). | Change from baseline in SPARCC enthesitis score | Calculated as: observed SPARCC enthesitis score – baseline SPARCC enthesitis score SPARCC enthesitis score | Missing if baseline or observed value is missing |
| | | • SPARCC enthesitis score = 0 | equals to 0, indicating complete resolution in enthesitis. | Missing if observed value is missing |
| Leeds Dactylitis<br>Index-Basic (LDI-B) | If the patient has dactylitis, the LDI-B will be administered by a blinded assessor. The LDI-B has been developed to measure the severity of dactylitis. Once the presence of dactylitis is established in each digit, the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot is measured (Helliwell et al. 2005). | • LDI-B score | Each dactylitic digit is defined by a minimum increase of 10% in circumference over the contralateral digit. If the same digits on each hand or foot are thought to be involved, the clinician will refer to a table of normative values (provided to study sites) for a value that will be used to provide the comparison. If the ratio is >1.1, then subtract 1 from the calculated ratio and multiply it by 100 and the tenderness | If 1 or more sites are missing, then set to missing. |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | | | score of 0 (not tender) or 1 | <u> </u> |
| | | | (tender). Otherwise, if the | |
| | | | ratio of the circumference of | |
| | | | the digit is $\leq 1.1$ , then the LDI- | |
| | | | B score is set to 0. Tenderness | |
| | | | is assessed in the area between | |
| | | | the joints. The results of each | |
| | | | digit are then added to produce | |
| | | | a total score (Healy and | |
| | | | Helliwell 2007). | |
| | | Change from | Calculated as: observed LDI- | Missing if baseline or |
| | | baseline in LDI-B | B score – baseline LDI-B | observed value are missing |
| | | | score | |
| | | • LDI-B score = 0 | LDI-B score equals to 0, | Missing if observed value is |
| | | | indicating complete resolution | missing |
| | | | in dactylitis. | |
| Disease Activity | The DAS28-CRP is a measure of | DAS28-CRP score | The following equation will be | If one or more variables are |
| Score based on C- | disease activity in 28 joints that | | used to calculate the DAS28 | missing, then set to missing. |
| Reactive Protein | consists of a composite numerical | | (Vander Cruyssen et al. 2005): | |
| (DAS28-CRP) | score utilizing the following variables: | | DAS28 - CRP | |
| | TJC, SJC, hs-CRP (measured in | | $=0.56(\sqrt{TJC\ 28})$ | |
| | mg/L), and PatGA recorded by | | $+ 0.28(\sqrt{SJC\ 28})$ | |
| | patients on a 0- to 100-mm VAS. | | $+ 0.36(\ln(CRP + 1))$ | |
| | For DAS28-CRP, the 28 joints to be | | + 0.014(VAS) + 0.96 | |
| | examined and assessed as tender or not | | Where | |
| | tender for TJC (TJC 28) and as | | TJC 28 is calculated as: | |
| | swollen or not swollen for SJC (SJC | | (sum of the evaluable | |
| | 28) are a subset of those assessed for | | individual joint | |
| | the TJC and SJC and include 14 joints | | scores)/(number of evaluable | |
| | on each side of the patient's body: the | | joints)×28; | |
| | 2 shoulders, the 2 elbows, the 2 wrists, | | SJC 28 is calculated as: | |
| | the 10 metacarpophalangeal joints, the | | (sum of the evaluable | |
| | 2 interphalangeal joints of the thumb, | | individual joint | |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | the 8 proximal interphalangeal joints, and the 2 knees (Smolen et al. 1995). | | scores)/(number of evaluable joints)×28 | |
| | | | See Appendix 3 for complete details. | |
| | | <ul> <li>DAS28-CRP &lt;2.6</li> <li>DAS28-CRP ≥2.6</li> <li>and &lt;3.2</li> <li>DAS28-CRP ≥3.2</li> <li>and &lt;5.1</li> <li>DAS28-CRP ≥5.1</li> </ul> | DAS28-CRP score falls in intervals $<2.6$ $\ge 2.6$ and $< 3.2$ $\ge 3.2$ and $< 5.1$ $\ge 5.1$ | Missing if DAS28-CRP score is missing |
| | | Change from baseline in DAS28- CRP | Calculated as: observed DAS28-CRP score – baseline DAS28-CRP score | Missing if baseline or observed value are missing |
| Modified Composite<br>Psoriatic Disease<br>Activity Index<br>(mCPDAI) | A validated instrument to assess composite psoriatic disease activity and response to therapy (Mumtaz et al. 2011). This instrument assesses individual domains: • peripheral arthritis as assessed by the number of tender and swollen joints and the HAQDI • skin as assessed by the PASI and the Dermatology Life Quality Index (DLQI) | mCPDAI total score | Each domain with the exception of spinal disease is scored from 0-3. Individual domain scores are summed to give an overall composite score (range 0-12) with a higher score indicating higher disease activity (see Appendix 5). | If 1 or more components are missing, then set to missing. |

| Measure | Description | Variable • Change from baseline in mCPDAI total score | Derivation/Comment Calculated as: observed mCPDAI score – baseline mCPDAI score | Imputation Approach if with Missing Components Missing if baseline or observed value are missing |
|---|---|---|---|---|
| | | • mCPDAI <u>&lt;</u> 5 | mCPDAI score ≤5, indicating low disease activity or remission in modified CPDAI (Salaffi et al. 2014) | Missing if observed mCPDAI is missing |

Abbreviations: BSA = body surface area; eCRF = electronic case report form; PsA = psoriatic arthritis.

 Table RHCF.6.4.
 Description of Primary and Secondary Efficacy Analyses

| Measure | Variable | Analysis Method<br>(Section 6.2) | Population (Section 6.1.3) | Comparison/Time<br>Point | Analysis Type |
|---|---|---|---|---|---|
| Composite endpoint<br>of American College<br>of Rheumatology<br>(ACR) 50 and | <ul> <li>Proportion of<br/>patients with<br/>ACR50 and<br/>PASI 100</li> </ul> | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at Week<br>24 and all other post-<br>baseline visits | Primary analysis (IXE vs ADA at Week 24) Secondary analysis |
| Psoriasis Area and<br>Severity Index<br>(PASI) 100 | simultaneously<br>(Primary<br>Endpoint at<br>Week 24) | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at Week<br>24 and all other post-<br>baseline visits | Secondary analysis |
| | <ul> <li>Time to first<br/>simultaneous<br/>ACR50 and<br/>PASI 100</li> </ul> | Log-rank Test<br>Kaplan-Meier product<br>limit method | ITT population | IXE vs ADA up to<br>Week 24 and Week 52 | Exploratory analysis |
| | response | Kaplan-Meier plots<br>(survival curve) | ITT population | IXE vs ADA up to<br>Week 24 and Week 52 | Exploratory analysis |
| American College of<br>Rheumatology<br>(ACR) Responder<br>Index 20, 50, and 70 | <ul> <li>Proportion of patients with ACR20</li> <li>Proportion of</li> </ul> | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at Week<br>24 and all other post-<br>baseline visits | Major secondary<br>analysis (ACR50: IXE<br>vs ADA at Week 24)<br>Secondary analysis |
| • | patients with ACR50 (Major Secondary Endpoint at Week 24) • Proportion of patients with ACR70 | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at Week<br>24 and all other post-<br>baseline visits | Secondary analysis |
| | • Time to first ACR20 response | Log-rank Test<br>Kaplan-Meier product<br>limit method | ITT population | IXE vs ADA up to<br>Week 24 and Week 52 | Exploratory analysis |

| | | Analysis Method | Population | Comparison/Time | |
|---|---|---|---|---|---|
| Measure | • Time to first ACR50 response • Time to first | (Section 6.2) Kaplan-Meier plots (survival curve) | (Section 6.1.3) ITT population | IXE vs ADA up to Week 24 and Week 52 | Analysis Type Exploratory analysis |
| Tender Joint Count (TJC) (68 joint | ACR70 response • Change from baseline in | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| count) | TJC Score | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Swollen Joint Count (SJC) (66 joint | • Change from baseline in | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| count) | SJC Score | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Patient's Assessment of Pain | Change from baseline in | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Visual Analog Scale<br>(VAS) | patient's pain<br>VAS score | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Patient's Global<br>Assessment of | Change from baseline in | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Disease Activity Visual Analog Scale (VAS) | patient's<br>global<br>assessment<br>VAS score | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Physician's Global<br>Assessment of | Change from baseline in | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Disease Activity Visual Analog Scale | physician's<br>global | ANCOVA model using mBOCF (see Section | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |

| Measure | Variable | Analysis Method<br>(Section 6.2) | Population (Section 6.1.3) | Comparison/Time<br>Point | Analysis Type |
|---|---|---|---|---|---|
| (VAS) | assessment<br>VAS score | 6.4.2) | | | |
| Patient's Assessment of Physical Function Health Assessment Questionnaire— | Change from baseline in HAQ-DI score | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Disability Index<br>(HAQ-DI) | | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | <ul> <li>Proportion of patients with HAQ-DI</li> </ul> | Logistic regression using the NRI method (see Section 6.4.1) | ITT population - patients with HAQ-DI ≥0.35 at baseline | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | improvement<br>≥0.35 | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population - patients with HAQ-DI \( \geq 0.\) 35at baseline | IXE vs ADA at each post-baseline visit | Secondary analysis |
| C-Reactive Protein (CRP) | Change from baseline in | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | CRP (mg/L) | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Disease Activity<br>Score based on C-<br>Reactive Protein<br>(DAS28-CRP) | Change from baseline in | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | DAS28-CRP | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | Proportion of patients with DAS28-CRP categories: | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Exploratory analysis |

| Measure | Variable | Analysis Method<br>(Section 6.2) | Population (Section 6.1.3) | Comparison/Time<br>Point | Analysis Type |
|---|---|---|---|---|---|
| | <2.6<br>≥2.6 and <3.2<br>≥3.2 and <5.1<br>≥5.1 | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Exploratory analysis |
| Psoriatic Arthritic<br>Response Criteria<br>(PsARC) | Proportion of patients achieving PsARC | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Psoriasis Area and<br>Severity Index<br>(PASI) | <ul> <li>Proportion of patients with PASI 75</li> <li>Proportion of patients with PASI 90</li> </ul> | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Major secondary<br>analysis (PASI 100:<br>IXE vs ADA at Week<br>24)<br>Secondary Analysis<br>(other visits) |
| | Proportion of patients with PASI 100 (major secondary endpoint at Week 24) | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |

| Measure | Variable | Analysis Method<br>(Section 6.2) | Population (Section 6.1.3) | Comparison/Time<br>Point | Analysis Type |
|---|---|---|---|---|---|
| | Change from baseline in PASI score | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | <ul> <li>Proportion of patients with absolute PASI</li> </ul> | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | score $\leq 1$ or $\leq 2$ or $\leq 3$ | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | Time to first PASI 75 response | Log-rank Test<br>Kaplan-Meier product<br>limit method | ITT population | IXE vs ADA up to<br>Week 24 and Week 52 | Exploratory analysis |
| | <ul> <li>Time to first PASI 90 response</li> <li>Time to first PASI 100 response</li> </ul> | Kaplan-Meier plots<br>(survival curve) | ITT population | IXE vs ADA up to<br>Week 24 and Week 52 | Exploratory analysis |
| Coates criteria for<br>Minimal Disease<br>Activity (MDA) (6 | Proportion of patients<br>achieving MDA (6<br>entheseal points) | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| entheseal points) | | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Coates criteria for<br>Minimal Disease<br>Activity (MDA) (18 | Proportion of patients<br>achieving Coates<br>criteria for MDA (18 | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| entheseal points) | entheseal points) | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |

| Measure | Variable | Analysis Method<br>(Section 6.2) | Population (Section 6.1.3) | Comparison/Time<br>Point | Analysis Type |
|---|---|---|---|---|---|
| Leeds Enthesitis Index (LEI) | Change from baseline in LEI score | MMRM | ITT population - patients with baseline enthesitis (LEI >0) | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population - patients with baseline enthesitis (LEI >0) | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | Proportion of patients with complete resolution in enthesitis | Logistic regression using the NRI method (see Section 6.4.1) | ITT population - patients<br>with baseline enthesitis<br>(LEI >0) | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | (LEI score = 0) | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population for patients with baseline enthesitis (LEI >0) | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Leeds Dactylitis<br>Index-Basic (LDI-B) | • Change from baseline in LDI-B score | MMRM | ITT population - patients<br>with baseline dactylitis<br>(LDI-B>0) | IXE vs ADA at or after<br>Week 12 | Secondary analysis |
| | | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population - patients<br>with baseline dactylitis<br>(LDI-B >0) | IXE vs ADA at or after<br>Week 12 | Secondary analysis |
| | Proportion of patients with complete resolution in dactylitis | Logistic regression using the NRI method (see Section 6.4.1) | ITT population - patients<br>with baseline dactylitis<br>(LDI-B >0) | IXE vs ADA at or after<br>Week 12 | Secondary analysis |
| | (LDI-B score = 0) | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population for patients with baseline dactylitis (LDI-B >0) | IXE vs ADA at or after<br>Week 12 | Secondary analysis |
| Spondyloarthritis<br>Research<br>Consortium of | • Change from baseline in SPARCC | MMRM | ITT population - patients with baseline enthesitis (SPARCC >0) | IXE vs ADA at each post-baseline visit | Secondary analysis |

| | | <b>Analysis Method</b> | Population | Comparison/Time | |
|---|---|---|---|---|---|
| Measure | Variable | (Section 6.2) | (Section 6.1.3) | Point | Analysis Type |
| | | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population - patients with baseline enthesitis (SPARCC >0) | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | Proportion of patients with complete resolution in enthesitis | Logistic regression using the NRI method (see Section 6.4.1) | ITT population - patients with baseline enthesitis (SPARCC >0) | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | (SPARCC enthesitis score = 0) | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population for patients with baseline enthesitis (SPARCC >0) | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Modified Composite<br>Psoriatic Disease<br>Activity Index | Change from baseline in modified | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| (mCPDAI) | CPDAI total scores | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | Proportion of patients with low disease activity or remission | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | (mCPDAI ≤5) | Fisher's exact test using the NRI method (see Section 6.4.1) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Body Surface Area (BSA) | • change from baseline in BSA | MMRM | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| | | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | IXE vs ADA at each post-baseline visit | Secondary analysis |
| Nail Psoriasis<br>Severity Index<br>(NAPSI) | Change from baseline in NAPSI score | MMRM | ITT population - patients with baseline fingernail involvement (NAPSI >0) | IXE vs ADA at or after<br>Week 12 | Secondary analysis |

| | | Analysis Method | Population | Comparison/Time | |
|---|---|---|---|---|---|
| Measure | Variable | (Section 6.2) | (Section 6.1.3) | Point | Analysis Type |
| | | ANCOVA model using | ITT population - patients | IXE vs ADA at or after | Secondary analysis |
| | | mBOCF (see Section | with baseline fingernail | Week 12 | |
| | | 6.4.2) | involvement (NAPSI >0) | | |
| | Proportion of patients | Logistic regression using | ITT population - patients | IXE vs ADA at each | Exploratory analysis |
| | with complete | the NRI method (see | with baseline fingernail | post-baseline visit at or | |
| | resolution in nail | Section 6.4.1) | involvement (NAPSI >0) | after Week 12 | |
| | psoriasis (NAPSI = 0) | Fisher's exact test using | ITT population - patients | IXE vs ADA at each | Exploratory analysis |
| | | the NRI method (see | with baseline fingernail | post-baseline visit at or | |
| | | Section 6.4.1) | involvement (NAPSI >0) | after Week 12 | |

Abbreviations: ADA = adalimumab; ANCOVA = analysis of covariance; ITT = intent to treat; IXE = ixekizumab; mBOCF = modified baseline observation carried forward; MMRM = mixed-effects model of repeated measures; NRI = non-responder imputation.

# 6.12.1. Analysis Methodology for Primary and Major Secondary Outcomes

### 6.12.1.1. Primary Outcome and Methodology

The primary efficacy endpoint is the proportion of patients simultaneously achieving both ACR50 and PASI 100 responses at Week 24.

ACR50 response is an efficacy measure for which a patient must satisfy the following:

- 1. ≥50% improvement from baseline in TJC and
- 2.  $\geq$ 50% improvement from baseline in SJC and
- 3.  $\geq$ 50% improvement from baseline in at least 3 of the following 5 ACR Core Set criteria:
  - a. Patient's Assessment of Pain Visual Analog Scale (VAS)
  - b. PatGA VAS
  - c. PGA VAS
  - d. patient's assessment of physical function as measured by the HAQ-DI
  - e. acute-phase reactant as measured by high sensitivity (assay) CRP (hs-CRP)

Full details of the algorithm to calculate ACR Response can be found in Appendix 2.

PASI 100 is an efficacy measure for which a patient must meet an improvement of 100% in the PASI compared to baseline.

The primary analysis for comparison of ixekizumab with adalimumab at Week 24 using the primary efficacy endpoint will be a logistic regression analysis as described in Section 6.2.1 based on the ITT population in the Open-Label Treatment Period (Period 2). Missing data will be imputed using the NRI method described in Section 6.4.1.

### 6.12.1.2. Methodology for Major Secondary Outcomes

The major secondary endpoints are as follows:

- 1. Proportion of patients achieving ACR50 in each treatment group at Week 24
- 2. Proportion of patients achieving PASI 100 in each treatment group at Week 24

The analyses of the secondary endpoints will be based on the ITT population in the Open-Label Treatment Period (Period 2) comparing ixekizumab versus adalimumab at Week 24 using methods described in Section 6.7 for the major secondary endpoint #1 and using methods from Section 6.2.1 for the major secondary endpoint #2. Missing data will be imputed using the NRI method described in Section 6.4.1.

A multiple testing procedure, as described in Section 6.6, will be used for testing the primary and major secondary endpoints.

#### 6.12.1.3. Other Secondary Outcomes

There will be no adjustment for multiple comparisons for other secondary analyses. The secondary analyses are detailed in Table RHCF.6.3 and Table RHCF.6.4.

By-patient listings for primary efficacy measurements ACR and PASI will be provided.

## 6.13. Health Outcomes/Quality-of-Life Analyses

The health outcomes and quality of life (QOL) measures are Itch NRS, Fatigue Severity NRS, SF-36, EQ-5D-5L, DLQI, and Treatment Satisfaction Questionnaire. Table RHCF.6.5 includes the description and derivation of the health outcomes and QOL measures.

The analyses of health outcome variables for Period 2 will be based on the ITT population.

Table RHCF.6.6 provides the detailed analyses including analysis type, method and imputation, population, time point, and treatment group comparisons for health outcomes and QOL analyses.

 Table RHCF.6.5.
 Description and Derivation of Health Outcomes and Quality-of-Life Measures

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| Itch Numeric Rating<br>Scale (NRS) | A single-item, patient-reported outcome (PRO) measure designed to | Itch NRS score | Range from 0 to 10 | Single item, missing if missing |
| | capture information on the overall severity of a patient's itching due to their psoriatic skin condition by having | Change from baseline in Itch NRS score | Calculated as: observe Itch NRS score – baseline Itch NRS score | Missing is baseline or observed value is missing |
| | the patient selecting the integer that best describes the worst level of itching in the past 24 hours on an 11-point NRS anchored at 0 representing "no itching" and 10 representing "worst itch imaginable." | • Itch NRS=0 | Defined as a post-baseline Itch<br>NRS score of 0 | Missing if Itch NRS score is missing |
| Fatigue Severity Numeric Rating | A patient-administered single-item 11-<br>point horizontal scale anchored at 0 | Fatigue Severity NRS | Range from 0 to 10. | Single item, missing if missing |
| Scale (NRS) | and 10, on which 0 represents "no fatigue" and 10 represents "as bad as you can imagine." Patients rate their fatigue (feeling tired or worn out) by selecting the single number that describes their worst level of fatigue during the past 24 hours. | Change from baseline in Fatigue severity NRS | Calculated as: observe Fatigue<br>NRS score – baseline Fatigue<br>NRS score | Missing is baseline or observed value is missing |
| Medical Outcomes<br>Study 36-item Short<br>Form Health Survey<br>(SF-36) | A 36-item patient-administered measure designed to be a short, multipurpose assessment of health in the areas of physical functioning, role-physical, role-emotional, bodily pain, vitality, social functioning, mental health, and general health. The 2 overarching domains of mental well-being and physical well-being are captured by the Mental Component Summary (MCS) and Physical Component Summary (PCS) scores. | Observed and change from baseline in: 8 associated domain scores: • Physical Functioning • Role Physical • Bodily Pain • General Health • Vitality • Social Functioning • Role Emotional • Mental Health | Per copyright owner, the Quality Metric Health Outcomes <sup>TM</sup> Scoring Software 4.5 will be used to derive SF-36 domain and component scores. After data quality-controls, the SF-36 software will re-calibrate the item-level responses for calculation of the domain and component scores. These raw scores will be transformed into the domain scores (t-scores) | Missing data handling<br>offered by SF-36 software<br>will not be used |

| | | | | Imputation Approach if |
|---|---|---|---|---|
| Measure | Description | Variable | Derivation/Comment | with Missing Components |
| | Items are answered on Likert scales of | 2 component Scores: | using the 1-week recall period. | |
| | varying lengths. The SF-36 version 2 | <ul> <li>MCS Score</li> </ul> | The procedure to derive the SF- | |
| | (acute version) health survey will be | <ul> <li>PCS Score</li> </ul> | 36 scores is described in | |
| | used, which has a 1-week recall period | | Appendix 6. The summary | |
| | (Brazier et al. 1992; Ware and | | scores range from 0 to 100. It | |
| | Sherbourne 1992). | | entails exporting the patient data | |
| | | | in a CSV or tab-delimited file | |
| | | | for import, generation of the SF- | |
| | | | 36 scores and reports, and export | |
| | | | of the calculated scores in a CSV | |
| | | | or tab-delimited file for | |
| | | | integration into SDTM/ADaM | |
| | | | datasets. The summary scores | |
| | | | range from 0 to 100. | |

| Москина | Description | Variable | Desiration/Comment | Imputation Approach if |
|---|---|---|---|---|
| Measure European Quality of Life - 5 Dimensions - 5 Level (EQ-5D-5L) | The EQ-5D-5L is a standardized measure of health status used to provide a simple, generic measure of health for clinical and economic appraisal. The EQ-5D-5L consists of 2 components: a descriptive system of the respondent's health and a rating of his or her current health state using a 0- to 100-mm VAS. The descriptive system comprises the following 5 dimensions: item 1: mobility item 2: self-care item 3: usual activities item 4: pain/discomfort item 5: anxiety/depression The respondent is asked to indicate his or her health state by ticking (or placing a cross) in the box associated with the most appropriate statement in each of the 5 dimensions. The EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, may be converted into a single summary index by applying a formula that essentially attaches values (also called weights) to each of the levels in each dimension (EuroQol Group [WWW]). The VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labeled 100 = "best imaginable health state" and 0 = "worst imaginable health state." This information can be used as a | Variable • EQ-5D mobility, • EQ-5D self-care, • EQ-5D usual activities, • EQ-5D pain/discomfort, • EQ-5D anxiety/depression, | Derivation/Comment 5 health profile dimensions, each dimension has 5 levels: 1 = no problems 2 = slight problems 3 = moderate problems 4 = severe problems It should be noted that the numerals 1 to 5 have no arithmetic properties and should not be used as a primary score. | with Missing Components Each dimension is a single item, missing if missing. (Note: Score of 9 is missing.) |

| | | | | Imputation Approach if |
|---|---|---|---|---|
| Measure | Description | Variable | Derivation/Comment | with Missing Components |
| | | EQ-5D VAS | Range from $0 =$ "worst | Single item, missing if |
| | | | imaginable health state" to 100 = | missing |
| | | | "best imaginable health state". | |
| | | | Note: higher value indicates | |
| | | | better health state. | |
| | | EQ-5D-5L UK Population- | Uses the concatenation of the | If any of the items is missing |
| | | based index score | value of each EQ- 5D-5L | or equal to 9, the index score |
| | | | dimension score in the order: | is missing |
| | | | item1; item2; item3; item4; | |
| | | | item5. Derive EQ-5D-5L UK | |
| | | | Population-based index score | |
| | | | according to the link by using | |
| | | | the UK algorithm (Szende et | |
| | | | al. 2007) to produce a patient- | |
| | | | level index score between -0.59 | |
| | | | and 1.0 (continuous variable): | |
| | | | http://www.euroqol.org/fileadmi | |
| | | | n/user_upload/Documenten/Exc | |
| | | | el/Crosswalk_5L/EQ-5D- | |
| | | | 5L_Crosswalk_Value_Sets.xls | |

| | | | | Imputation Approach if |
|---|---|---|---|---|
| Measure | Description | Variable | Derivation/Comment | with Missing Components |
| Dermatology Life | The DLQI is a validated, dermatology- | DLQI symptoms and | Sum of responses of questions | If 1 question in a domain is |
| Quality Index | specific, patient-reported measure that | feelings domain | #1 and #2: | missing, that domain is |
| (DLQI) | evaluates patient's health-related | | #1. How itchy, sore, painful or | missing. |
| | quality of life. This questionnaire has | | stinging has your skin been? | |
| | 10 items that are grouped in 6 | | #2. How embarrassed or self- | |
| | domains, including symptoms and | | conscious have you been | |
| | feelings, daily activities, leisure, work | | because of your skin? | |
| | and school, personal relationships, and | | | |
| | treatment. The recall period of this | | | |
| | scale is over the "last week." | | | |
| | Response categories and | | | |
| | corresponding scores are: | | | |
| | Very much = 3 | | | |
| | A lot = 2 | | | |
| | A little $= 1$ | | | |
| | Not at all $= 0$ | | | |
| | Not relevant = 0 | | | |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | - | DLQI daily activities | Sum of responses of questions | If 1 question in a domain is |
| | | domain | #3 and #4: | missing, that domain is |
| | | | #3. How much has your skin interfered with you going | missing. |
| | | | shopping or looking after your | |
| | | | home or garden? | |
| | | | #4. How much has your skin | |
| | | | influenced the clothes you wear? | |
| | | DLQI leisure domain | Sum of responses of questions | If 1 question in a domain is |
| | | | #5 and #6: | missing, that domain is |
| | | | #5. How much has your skin | missing. |
| | | | affected any social or leisure | |
| | | | activities? | |
| | | | #6. How much has your skin | |
| | | | made it difficult for you to do | |
| | | 5.0. | any sport? | |
| | | DLQI work and school | Sum of responses of questions | If the answer to question |
| | | domain | #7A and #7B: | #7A is missing, this domain |
| | | | #7A. Has your skin prevented | is missing. If #7A is No, |
| | | | you from working or studying?<br>#7B. If No: how much has your | and #7B is missing, this domain is missing. |
| | | | skin been a problem at work or | domain is missing. |
| | | | studying? | |
| | | DLQI personal and | Sum of responses of questions | If 1 question in a domain is |
| | | relationships domain | #8 and #9: | missing, that domain is |
| | | | #8. How much has your skin | missing. |
| | | | created problems with your | |
| | | | partner or any of your close | |
| | | | friends or relatives? | |
| | | | #9. How much has your skin | |
| | | DI OI | caused any sexual difficulties? | 704 |
| | | DLQI treatment | Response of question #10: | If 1 question in a domain is |
| | | | #10. How much of a problem | missing, that domain is |

| Measure | Description | Variable | Derivation/Comment | Imputation Approach if with Missing Components |
|---|---|---|---|---|
| | <b>,</b> | , 33-33-33 | has the treatment for your skin<br>been, for example by making<br>your home messy, or by<br>taking up time? | missing. |
| | | DLQI total score | A DLQI total score is calculated by summing all 10 question responses and has a range of 0 to 30 (less to more impairment) (Finlay and Khan 1994; Basra et al. 2008). | If 2 or more questions are missing, the total score is missing. Note: #7B could be a valid missing while #7A is not "No." That is, #7 should be considered as 1 question. |
| | | Change from baseline in | Calculated as observed DLQI – | Missing if baseline or |
| | | DLQI total score | baseline DLQI | observed value are missing |
| | | DLQI (0,1) | A DLQI (0,1) response is defined as a post-baseline DLQI total score of 0 or 1. A DLQI total score of 0 to 1 is considered as having no effect on a patient's HRQoL (Khilji et al. 2002; Hongbo et al. 2005). | Missing if DLQI total score is missing |
| Treatment<br>Satisfaction<br>Questionnaire (TSQ) | The TSQ is a clinician-administered questionnaire that provides an assessment of the patient's opinion of the effectiveness, safety, and overall satisfaction of the study medication. Patients will be asked to respond to questionnaire items using a 4-point | Question #1 = "mostly satisfied" | Patient's answer to Question #1:<br>Please tell me whether you are<br>mostly satisfied, somewhat<br>satisfied, somewhat dissatisfied,<br>or mostly dissatisfied with the<br>effectiveness of this medication<br>is mostly satisfied. | Single item, missing if missing |

| | | | | Imputation Approach if |
|---|---|---|---|---|
| Measure | Description | Variable | Derivation/Comment | with Missing Components |
| | | Question #2 = "mostly | Patient's answer to Question #2: | Single item, missing if |
| | | satisfied" | Please tell me whether you are | missing |
| | | | mostly satisfied, somewhat | |
| | | | satisfied, somewhat dissatisfied, | |
| | | | or mostly dissatisfied with the | |
| | | | effectiveness over time of this | |
| | | | medication is mostly satisfied. | |
| | | Question #3 = "mostly | Patient's answer to Question #3: | Single item, missing if |
| | | satisfied" | Please tell me whether you are | missing |
| | | | mostly satisfied, somewhat | |
| | | | satisfied, somewhat dissatisfied, | |
| | | | or mostly dissatisfied with the | |
| | | | long term safety of this | |
| | | | medication is mostly satisfied. | |
| | | Question #4 = "mostly | Patient's answer to Question #4: | Single item, missing if |
| | | satisfied" | How would you rate your overall | missing |
| | | | satisfaction with this medication | |
| | | | is mostly satisfied. | |

Table RHCF.6.6. Description of Health Outcomes and Quality-of-Life Analyses

| Measure | Variable | Analysis Method<br>(Section 6.2) | Population (Section 6.1.3) | Comparison/Time Point | Analysis Type |
|---|---|---|---|---|---|
| Itch NRS | Change in baseline for Itch NRS | MMRM ANCOVA model using mBOCF (see | ITT population ITT population | At each post-baseline visit At each post-baseline visit | Secondary analysis Secondary analysis |
| | Itch NRS = 0 | Section 6.4.2) Logistic regression using the NRI method (see Section 6.4.1) | ITT population for patients with baseline Itch NRS >0 | At each post-baseline visit | Secondary analysis |
| | | Fisher's exact test<br>using the NRI<br>method (see Section<br>6.4.1) | ITT population for patients with baseline Itch NRS >0 | At each post-baseline visit | Secondary analysis |
| NRS bas | Change from baseline in fatigue severity NRS score | MMRM | ITT population | At Week 4, 12, 16, 24, 32, and 52 | Secondary analysis |
| | | ANCOVA model<br>using mBOCF (see<br>Section 6.4.2) | ITT population | At Week 4, 12, 16, 24, 32, and 52 | Secondary analysis |
| Medical<br>Outcomes Study<br>36-item Short- | Change from baseline in: • Mental component summary score | MMRM | ITT population | At Week 4, 12, 16, 24, 32, and 52 | Secondary analysis |
| Form Health<br>Survey | Physical component<br>summary score | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | At Week 4, 12, 16, 24, 32, and 52 | Secondary analysis |
| | Change from baseline in 8 domain scores | MMRM | ITT population | At Week 4, 12, 16, 24, 32, and 52 | Exploratory analysis |
| | | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | At Week 4, 12, 16, 24, 32, and 52 | Exploratory analysis |

| Measure | Variable | Analysis Method<br>(Section 6.2) | Population (Section 6.1.3) | Comparison/Time Point | Analysis Type |
|---|---|---|---|---|---|
| DLQI | Change from baseline in DLQI total score | MMRM | ITT population | At each post-baseline visit | Secondary analysis |
| | | ANCOVA model using mBOCF (see Section 6.4.2) | ITT population | At each post-baseline visit | Secondary analysis |
| | • DLQI (0,1) | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | At each post-baseline visit | Exploratory<br>analysis |
| | | Fisher's exact test<br>using the NRI<br>method (see Section<br>6.4.1) | ITT population | At each post-baseline visit | Exploratory<br>analysis |
| EQ-5D-5L | Change from baseline in EQ-5D VAS | MMRM ANCOVA model using mBOCF (see Section 6.4.2) | ITT Population ITT Population | At Week 4, 12, 16, 24, 32, and 52 At Week 4, 12, 16, 24, 32, and 52 | Secondary analysis Secondary analysis |
| | Change from baseline<br>in EQ-5D-5L UK<br>Population-based index<br>score | MMRM ANCOVA model using mBOCF (see Section 6.4.2) | ITT Population ITT Population | At Week 4, 12, 16, 24, 32, and 52 At Week 4, 12, 16, 24, 32, and 52 | Secondary analysis Secondary analysis |
| TSQ | Proportion of patients answering "mostly satisfied" to • Question #1 | Logistic regression using the NRI method (see Section 6.4.1) | ITT population | At Week 12, 24, and 52 | Secondary analysis |
| | <ul><li> Question #2</li><li> Question #3</li><li> Question #4</li></ul> | Fisher's exact test<br>using the NRI<br>method (see Section<br>6.4.1) | ITT population | At Week 12, 24, and 52 | Secondary analysis |

Abbreviations: ANCOVA = analysis of covariance; EQ-5D-5L = European Quality of Life-5 Dimensions 5 Level Health Outcomes Instrument; DLQI = Dermatology Life Quality Index; ITT = intent-to-treat; mBOCF = modified baseline observation carried forward; MMRM = mixed-effects model of repeated measures; NRI = non-responder imputation; NRS = Numeric Rating Scale; TSQ = Treatment Satisfaction Questionnaire; UK = United Kingdom; VAS = Visual Analog Scale.

## **6.14.** Bioanalytical and Pharmacokinetic/Pharmacodynamic Methods N/A

## 6.15. Safety Analyses

The primary safety analyses will focus on comparisons of ixekizumab versus adalimumab in the Open-Label Treatment Period (Period 2). Fisher's exact test will be used for all AEs and other categorical safety data. Continuous vital sign and laboratory values will be analyzed by an ANCOVA with treatment and baseline value in the model. Type 3 sums of squares will be used. The significance of within-treatment group changes from baseline will be evaluated by testing whether the treatment group LSMean changes from baseline are different from zero using a t-statistic. In addition to the LSMeans and tests, the standard deviation, minimum, median, and maximum will be displayed. Unless otherwise specified, change from baseline will include only those subjects with both baseline and post-baseline measures.

For safety analyses, p-values should be interpreted with caution as the analyses are intended to be descriptive and should not be thought of as hypothesis testing, unless there is a prespecified hypothesis. P-values and CIs, if reported, provide some evidence of the strength of the finding and are only useful as a flagging mechanism.

Summaries of safety data collected during the Post-Treatment Follow-Up Period will be presented separately. The categorical safety measures will be summarized with incidence rates. The continuous safety measures will be summarized using mean changes.

## 6.15.1. Extent of Exposure

Duration of exposure to study drug will be summarized by treatment group using descriptive statistics; the summary will also include the total exposure in patient years, mean, and median total dose. Exposure of safety population in the Open-Label Treatment Period (Period 2) will be summarized.

The duration of exposure will be calculated as follows:

- Duration of exposure (days) =
   Date of last visit (scheduled or unscheduled) during the treatment period –
   Date of first injection for the treatment period + 1
- Total exposure in patient years will be calculated as follows:

Total exposure in patient years  $= \frac{Sum \ of \ duration \ (days) \ of \ exposures \ for \ all \ patients \ in \ treatment \ group}{365.25}$ 

- Total dose (in mg) is calculated by the summation of dose for each active injection taken during the treatment period.
- Note that the total number of injections received will be calculated using the response to the question "Was the injection given?" on the *Study administration* electronic eCRF page.

Descriptive statistics will be provided for patient days of exposure and the frequency of patients falling into the following different exposure ranges (that is, only the exposure ranges that fall within the treatment period will be presented) will be summarized:

- $>0, \ge 7 \text{ days}, \ge 14 \text{ days}, \ge 30 \text{ days}, \ge 60 \text{ days}, \ge 90 \text{ days}, \ge 120 \text{ days}, \ge 183 \text{ days}, \ge 365 \text{ days}.$
- >0 to <7 days, ≥7 to <14 days, ≥14 to <30 days, ≥30 to <60 days, ≥60 to <90 days, ≥90 to <120 days, ≥120 to <183 days, ≥183 to <365 days, and ≥365 days.

#### 6.15.2. Adverse Events

### 6.15.2.1. Analyses of Adverse Events

Adverse events are classified based on MedDRA. A treatment-emergent adverse event (TEAE) is defined as an event that first occurred or worsened in severity after the first dose of the study medication and on or prior to the date of the last visit within the treatment period. Both the date/time of the event and the date/time of the dose (that is, injection) are considered when determining TEAEs. The MedDRA Lowest Level Term (LLT) will be used in the treatment-emergent computation. The maximum severity for each LLT during the baseline period will be used as baseline severity (in some cases baseline period is a single time point). Events with a missing severity during the treatment period will be considered treatment emergent. The treatment period will be included as post-baseline for the analysis. If an event is pre-existing during the baseline period but it has missing severity, and the event persists during the treatment period, then it will be considered as treatment-emergent, regardless of the post-baseline level of severity. Adverse events with a particular LLT will be classified as treatment-emergent if they first start on or after the first dose date in the treatment period (ie, a patient has no pre-existing conditions with that LLT) or if the severity is greater than the pre-treatment severity for that LLT.

A follow-up emergent adverse event (FEAE) is defined as an event that first occurred or worsened in severity after the date of Week 52 (Visit 11) or the ETV. The MedDRA LLT will be used when classifying FEAEs as follow-up emergent. For AEs that are ongoing at the date of Week 52 (Visit 11) or ETV, the maximum severity recorded for each LLT on the date of Week 52 (Visit 11) or ETV will be used as the follow-up baseline severity for that LLT.

If a partial or completely missing AE start date/time or end date/time is present, the following imputation rules will be utilized in the analysis:

- For the start date:
  - o If year, month, and day are missing, then use the earlier of the patient's first visit date or the consent date.
  - o If either month or month and day are missing, then use January 1.
  - o If only day is missing, impute the first day of the month.
  - o The imputed date should not be before the minimum of the patient's first visit or consent date.
- For the start time:
  - o Impute as 23:59

- For the end date:
  - o If year, month, and day are missing, then use the patient's last visit date in the follow-up period.
  - o If either month or month and day are missing, then use December 31.
  - o If only day is missing, then use the last day of the month.
  - The imputed date will not be beyond the patient's last visit date in the follow-up period.
- For the end time:
  - o Impute as 23:59.
- If there is any doubt, the event will be flagged as treatment-emergent or follow-up emergent according to the corresponding study period. If a follow-up emergent event was already counted as treatment-emergent during the prior treatment period, it will not be counted as a follow-up emergent event.

An overview table will be provided and will include the frequency and percentage of patients who experienced a TEAE, TEAE by maximum severity, a treatment-emergent adverse events of special interest (AESI), serious adverse event (SAE), death, or discontinued from the study due to an AE (including death) will be summarized by treatment group for the Open-Label Treatment Period.

In general, for all AE-related summaries, the number and percentage of patients experiencing the events will be presented by dosing regimen. When the SOC is presented, events will be ordered by decreasing frequency in the ixekizumab treatment group within SOC. When the SOC is not presented, the events will be ordered by decreasing frequency in the ixekizumab treatment group. For incidence counts, each patient will be counted only once within each PT and within each SOC. Percentages will be based on the number of patients in a particular treatment group. For events that are gender specific, the denominator and computation of the percentage will include only patients from the given gender.

The following summary tables will be provided for the Open-Label Treatment Period (Safety Population):

- An overview summary of AEs
- TEAEs, by SOC and PT
- TEAEs, by PT
- TEAEs by maximum severity, by SOC and PT

The following summary tables will be provided for the Post-Treatment Follow-Up Period (Follow-Up Population):

• FEAEs, by maximum severity, by SOC and PT

By-patient listing of all TEAEs will be provided.

#### 6.15.2.2. Common Adverse Events

The number and percentages of patients with common TEAEs will be summarized by treatment group for each treatment period using similar methods described in Section 6.15.2.1. Common

TEAEs will be defined as those TEAEs that occurred in ≥1% before rounding of total treated patients including all ixekizumab dose regimens. Events will be ordered by decreasing frequency within SOC or PT in the combined ixekizumab dose group.

The following summary tables will be provided for the Open-Label Treatment Period (Safety Population):

• TEAEs, by PT

## 6.15.3. Deaths, Other Serious Adverse Events, and Other Notable Adverse Events

By-patient listings of deaths, SAEs, and AEs leading to discontinuation will be provided, respectively.

All deaths will be included, regardless of the investigator's or the sponsor's judgment about causality, including the following:

- any deaths occurring during participation in the study in the database for which data are being presented
- any deaths occurring after a patient leaves (is discontinued from or completed) the study in the database for which data are being presented if the death is:
  - o the result of a process initiated during the study, regardless of when it actually occurred, or
  - o occurs during Period 3 after discontinuation of study drug

An SAE is any AE that results in one of the following outcomes: death; life-threatening, initial, or prolonged hospitalization; disability or permanent damage; congenital anomaly or birth defect; or any other serious/important medical events.

The following summary tables (including treatment group comparison for Period 2) will be provided for the Safety Population during the Open-Label Treatment Period (Period 2):

- SAEs by SOC and PT
- AEs that lead to treatment discontinuation (including death) by SOC and PT

The following summary tables (by treatment group during Period 2) will be provided for the Post-Treatment Follow-Up Population during the Post-Treatment Follow-Up Period (Period 3):

- Follow-up emergent SAEs (FESAEs) by SOC and PT
- FEAEs that lead to treatment discontinuation (including death) by SOC and PT

## 6.15.3.1. Special Safety Topics Including Adverse Events of Special Interest

Safety information on special topics including AESI will be presented by treatment group and by study period. Table RHCF.6.7 provides the definitions/derivations and analyses methods (including analyses, summaries, and by-patient listings) of special safety topics including AESIs.

Potential AESIs will be identified by a standardized MedDRA query (SMQ) or a Lilly-defined MedDRA PT listing. Preferred terms within an SMQ will be classified as broad or narrow. In

the Lilly-defined MedDRA PT listings, Lilly has provided the broad and narrow classification. The Lilly-defined broad terms are for a more sensitive search of potential events of interest and the Lilly-defined narrow terms are for a more specific search. Therefore, the summaries will include the classifications of broad term (same as pooling narrow and broad terms together) and narrow term. In the event that the listing of terms or analysis changes for a special safety topic, it will be documented in the program safety analysis plan (PSAP), which will supersede this document; it will not warrant an amendment to the individual study SAP.

 Table RHCF.6.7.
 Definitions and Analyses of Special Safety Topics

| Special Safety<br>Topic | Definition/Derivation | Analysis/Summary/Listing |
|---|---|---|
| Hepatic | Hepatic AE analysis will include events that are potentially drug-related hepatic disorders by using the MedDRA PTs contained in any of the following SMQ or sub-SMQ as defined in MedDRA: • Broad and narrow terms in the Liver-related investigations, signs and symptoms (20000008) • Broad and narrow terms in the Cholestasis and jaundice of hepatic origin (20000009) • Broad and narrow terms in the Hepatitis, non-infectious (20000010) • Broad and narrow terms in the Hepatic failure, fibrosis and cirrhosis and other liver damage (20000013) • Narrow terms in the Liver-related coagulation and bleeding disturbances (20000015) | Open-Label Treatment Period (Safety Population): TEAE by PT within SMQ or sub-SMQ |
| | Elevations in hepatic laboratory tests (ALT, AST, ALP, total bilirubin) using Performing Laboratory Reference Ranges are defined as: • Include scheduled visits, unscheduled visits, and repeat measurements. • ALT or AST: maximum post-baseline measurement ≥3 times (3×), 5 times (5×), 10 times (10×), and 20 times (20×) the Performing Lab ULN for all patients with a post-baseline value. • The analysis of 3× ULN will contain 4 subsets: patients whose non-missing maximum baseline value is ≤1× ULN, patients whose maximum baseline is >1× ULN but <3× ULN, patients whose maximum baseline value is ≤0× ULN will contain 5 subsets: patients whose non-missing maximum baseline value is ≤ to 1× ULN, patients whose maximum baseline is >1× ULN but <3× ULN, patients whose maximum baseline is ≥5× ULN, patients whose maximum baseline value is ≥5× ULN, and patients whose baseline value is ≥5× ULN, patients whose baseline value is ≤1× ULN, patients whose maximum baseline value is ≤1× ULN, patients whose maximum baseline is ≥1× ULN but <3× ULN, patients whose maximum baseline is ≥5× ULN but <10× ULN, patients whose maximum baseline value is ≥10× ULN, and patients whose baseline values are missing. • The analysis of 20× ULN will contain 7 subsets: patients whose non-missing maximum baseline value is ≤1× ULN, patients whose maximum baseline is >1× ULN but <3× ULN, patients whose maximum baseline is >1× ULN but <3× ULN, patients whose maximum baseline value is ≤1× ULN, patients whose maximum baseline is ≥1× ULN but <3× ULN, patients whose maximum baseline is ≥1× ULN but <3× ULN, patients whose maximum baseline is ≥1× ULN but <20× ULN, patients whose maximum baseline is ≥5× ULN but <10× ULN, patients whose maximum baseline is ≥10× ULN but <20× ULN, patients whose maximum baseline is ≥1× ULN but <20× ULN, patients whose maximum baseline value is ≤1× ULN will contain 4 subsets: patients whose non-missing maximum baseline value is ≤1× ULN, >1× ULN to <3× ULN, ≥3× ULN, or missing. | Open-Label Treatment Period (Safety Population): Elevations in hepatic laboratory tests: maximum baseline category to abnormal maximum post-baseline category |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| Topic | <ul> <li>Definition/Derivation</li> <li>The analysis of 5× ULN will contain 5 subsets: patients whose non-missing maximum baseline value is ≤1× ULN, &gt;1× ULN to &lt;3× ULN, ≥3× ULN to &lt;5× ULN, ≥5× ULN, or missing.</li> <li>The analysis of 10× ULN will contain 6 subsets: patients whose non-missing maximum baseline value is ≤1× ULN, &gt;1×ULN to &lt;3× ULN, ≥3× ULN to &lt;5× ULN, ≥5× ULN to &lt;10× ULN, ≥10× ULN, or missing.</li> <li>The analysis of 20× ULN will contain 7 subsets: patients whose non-missing maximum baseline value is ≤1×ULN, &gt;1×ULN to &lt;3× ULN, ≥3× ULN to &lt;5× ULN, ≥5× ULN to &lt;10× ULN, ≥10× ULN to &lt;20× ULN, ≥20× ULN, or missing.</li> <li>Total bilirubin: The number and percentages of patients with a total bilirubin measurement ≥1.5 times (1.5×), and ≥2 times (2×) the Performing Lab ULN during the treatment period will be summarized for all patients with a post-baseline value.</li> <li>The analysis of 1.5× ULN will contain 4 subsets: patients whose non-missing maximum baseline value is ≤1× ULN, patients whose maximum baseline is &gt;1× ULN but &lt;1.5× ULN, patients whose maximum baseline values are missing.</li> <li>The analysis of 2× ULN will contain 5 subsets: patients whose non-missing maximum baseline value is ≤1× ULN, patients whose maximum baseline is &gt;1× ULN but &lt;1.5× ULN, patients whose maximum baseline value is ≥1× ULN, patients whose maximum baseline value is ≥1× ULN, patients whose maximum baseline value is ≥1× ULN, patients whose maximum baseline value is ≥2× ULN, and patients whose baseline values are missing.</li> <li>ALP: The number and percentages of patients with an ALP measurement &gt;1.5× the Performing Lab</li> </ul> | Analysis/Summary/Listing |
| | <ul> <li>ULN during the treatment period will be summarized for all patients with a post-baseline value, and divided into 4 subsets: patients whose non-missing maximum baseline value is ≤1× ULN, patients whose maximum baseline is &gt;1× ULN but ≤1.5× ULN, patients whose maximum baseline value is &gt;1.5× ULN, and patients whose baseline values are missing.</li> <li>The number and percentages of patients meeting the following elevated hepatic criteria: maximum ALT ≥3× ULN and maximum Total Bilirubin ≥2× ULN during the treatment period will be summarized.</li> </ul> | |
| | Shift for ALT, AST, and total bilirubin from maximum baseline to maximum post-baseline will be | Open-Label Treatment |
| | produced with the requirements using Performing Lab Reference Ranges: | Period (Safety Population): |
| | Include scheduled visits, unscheduled visits, and repeat measurements. | Shifts from maximum baseline |
| | Use the maximum non-missing value in the baseline period. | to maximum post-baseline |
| | Use the maximum non-missing post-baseline value within each study period. | category |
| | • Categories are: | |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| Topic | <ul> <li>ALT: ≤1× ULN, &gt;1 to &lt;3× ULN, ≥3 to &lt;5× ULN, ≥5 to &lt;10× ULN, ≥10 to &lt;20× ULN, and ≥20× ULN</li> <li>AST: ≤1× ULN, &gt;1 to &lt;3× ULN, ≥3 to &lt;5× ULN, ≥5 to &lt;10× ULN, ≥10× to &lt;20× ULN, and ≥20× ULN</li> <li>Total bilirubin: ≤1× ULN, &gt;1 to &lt;1.5× ULN, ≥1.5 to &lt;2× ULN, and ≥2× ULN</li> <li>ALP: ≤1× ULN, &gt;1 to ≤1.5× ULN, and &gt;1.5× ULN</li> <li>With additional categories: <ul> <li>Decreased: post-baseline category &lt; baseline category</li> <li>Increased: post-baseline category &gt; baseline category</li> <li>Same: post-baseline category = baseline category</li> </ul> </li> </ul> | |
| | Elevated hepatic criteria: maximum ALT ≥3× ULN and maximum total bilirubin ≥2× ULN. Listing of patients who meet any of the following criteria: • Elevated hepatic criteria: defined as maximum ALT ≥3× ULN, maximum total bilirubin ≥2× ULN • An ALT or AST ≥3× ULN • An ALP ≥1.5× ULN • A total bilirubin ≥2× ULN The listing will include patient demographics, concomitant medications, ALT/AST/ALP/total bilirubin/GGT by visit, treatment start and stop dates, and reason for treatment discontinuation | Open-Label Treatment Period (Safety Population): Elevated hepatic criteria |
| | eDISH plot: Use maximum ALT measurement and maximum total bilirubin measurement with patients having at least 1 post-baseline ALT and total bilirubin, which contributes 1 point to the plot. The measurements do not need to be taken at the same blood draw. | Open-Label Treatment Period (Safety Population): eDISH plot (to be prepared in spotfire) |
| Cytopenias | Cytopenias are defined using the PTs from the following 2 sub-SMQs of the Haematopoietic cytopenias SMQ (20000027) as specified in MedDRA: Broad and narrow terms in the Haematopoietic leukopenia (20000030) Broad and narrow terms in the Haematopoietic thrombocytopenia (20000031) | Open-Label Treatment Period (Safety Population): TEAE by PT within sub-SMQ |
| Infections | Infections are events including all infections (defined using all the MedDRA PTs from the Infections and infestations SOC), serious infections, potential opportunistic infections, and infections resulting in anti-infective medication administration (i.e., antibacterial, antiviral, antifungal, antiparasitic treatment.). The relationship between TEAE infections and other clinical, laboratory, and hematology parameters will be examined using Spotfire tool. | Open-Label Treatment Period (Safety Population): TEAE by PT TEAE by maximum severity by PT* SAE by PT* |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| | | AEs leading to discontinuation of study drug* |
| | | *Included in overall TEAE by maximum severity, SAE and DCAE. |
| | Anti-infective medications are defined in Appendix 8 including antibiotics, antifungals, antivirals, or antiprotozoals. | |
| | The OIs are defined in Appendix 9. This list contain PTs as contained within Categories (narrow or broad) from the Infections and Infestations SOC and from the Investigations SOC that can assist in identifying potential OIs. The narrow terms are considered OIs unless medical review determines that the reported term is not consistent with the patient's clinical history/presentation/course. Medical review of broad terms is needed for final determination of patients meeting the program definition of OIs. | Open-Label Treatment Period (Safety Population): TEAE of OIs by PT within category |
| | The number and percentage of patients with TEAEs that represent potential OIs and as potential OIs will be summarized by treatment group using MedDRA PT nested within categories. Events will be ordered by decreasing frequency in the ixekizumab group nested within categories. | Listing:<br>TEAE of OIs |
| | The duration of each common TEAE PT of Infections and narrow terms for OIs is defined as: Duration of treatment-emergent AE Infections (in weeks) = (End date of AE – Start date of AE + 1) / 7 Patients who do not have the PT will not be included in the analysis. If the TEAE has not been reported as ended by the date of completion from the study, or date of early discontinuation, it will be censored as of that date. If a patient has multiple episodes of the same TEAE, the episode with the greatest severity will be used for the duration of event calculation. If a patient has multiple episodes of the same TEAE with the same severity, the episode with the longest duration will be used for the duration of event calculation. | Open-Label Treatment Period (Safety Population): Duration of Common TEAE Duration of OIs (narrow terms) (to be prepared in spotfire) Duration of Candida infections (to be prepared in spotfire) |

| Special Safety | Definition/Derivation | Analysis/Summary/Listing |
|---|---|---|
| Topic | | Analysis/Summary/Listing |
| Allergic | Allergic reactions/hypersensitivity events will be categorized as either anaphylaxis or non-anaphylaxis | Open-Label Treatment |
| Reactions/ | events (these will refer to events that are not localized to the site of injection) and summarized separately. | Period (Safety Population): |
| Hypersensitivit | Allergic Reactions/Hypersensitivity Events, Anaphylaxis: Anaphylaxis has been broadly defined as "a | TEAE by PT within Category TEAE by maximum severity by |
| ies | serious allergic reaction that is rapid in onset and may cause death" (Sampson et al. 2006). Identification of cases of potential anaphylaxis from the clinical trial data involves two screening criteria: | PT |
| | 1) designed to specifically identify cases (following Criterion 1) based on narrow terms from the | SAE by PT within Category |
| | MedDRA SMQ for anaphylactic reaction (20000021). Criterion 1 for anaphylaxis is defined by the | AE leading to discontinuation |
| | presence of a TEAE based on the following MedDRA PTs from the anaphylactic reaction SMQ: | of study drug within Category |
| | Anaphylactic reaction | of study drug within Category |
| | Anaphylactic shock | |
| | <ul> <li>Anaphylactoid reaction</li> <li>Anaphylactoid shock</li> </ul> | |
| | Kounis Syndrome | |
| | Type 1 hypersensitivity | |
| | 2) to identify possible cases, following Criterion 2 as defined by Sampson et al. (2006). Criterion 2 for | |
| | anaphylaxis requires having TEAEs from two or more of four categories of AEs as described by | |
| | Sampson et al. (2006). Occurrence of these events should be nearly coincident; based on recording | |
| | of events or CRFs. All qualifying events must be within 1 day of study drug injection. | |
| | The 4 categories to be considered in Criterion 2 are: | |
| | Category A: Involvement of the skin-mucosal tissue | |
| | Category B: Respiratory compromise | |
| | Category C: Reduced blood pressure or associated symptoms | |
| | Category D: Persistent gastrointestinal symptoms | |
| | The specific MedDRA PTs covered by each of these Criterion 2 categories are shown in Appendix 10. | |
| | Summaries of Criterion 2 anaphylactic TEAEs will be provided by the specific combination of categories | |
| | as follows: | |
| | AB: events based on meeting Category A and Category B (but no other category) | |
| | AC: events based on meeting Category A and Category C (but no other category) | |
| | AD: events based on meeting Category A and Category D (but no other category) | |
| | BC: events based on meeting Category B and Category C (but no other category) | |
| | BD: events based on meeting Category B and Category D (but no other category) | |
| | <ul> <li>CD: events based on meeting Category C and Category D (but no other category)</li> <li>ABC: events based on meeting Category A, Category B, and Category C (but no other category)</li> <li>ABD: events based on meeting Category A, Category B, and Category D (but no other category)</li> </ul> | |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| | ACD: events based on meeting Category A, Category C, and Category D (but no other category) BCD: events based on meeting Category B, Category C, and Category D (but no other category) ABCD: events based on meeting each of the 4 Criterion 2 categories Summaries of treatment-emergent anaphylactic AEs will be provided for patients meeting each of the 2 criteria and for patients who meet either criteria overall. Separate summaries will be provided for TEAEs by maximum severity, SAEs, and AEs resulting in study drug discontinuation. Severity of treatment-emergent Criterion 2 anaphylactic AEs will be based on the maximum severity of the specific events met by the patient. Maximum severity of an (overall) treatment-emergent anaphylactic AE will be based on the maximum severity within Criterion 1 and/or Criterion 2. Allergic Reactions/Hypersensitivity Events, Non-Anaphylaxis: TEAEs of allergic reaction/hypersensitivity categorized as non-anaphylaxis events are defined by the narrow terms within Hypersensitivity SMQ (20000214) excluding the PTs noted in Appendix 11 and excluding the anaphylactic events as defined above. | |
| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| Injection Site | Injection site reaction is defined using the PTs from the MedDRA HLT of Injection site reactions as | <b>Open-Label Treatment</b> |
| Reactions | defined by MedDRA excluding the following 10 PTs: | Period (Safety Population): |
| | 1) Embolia cutis medicamentosa | TEAE by PT within HLT |
| | 2) Injection site joint discomfort | TEAE by maximum severity by |
| | 3) Injection site joint effusion | PT within HLT |
| | 4) Injection site joint redness | AE leading to discontinuation |
| | 5) Injection site joint infection | of study drug within HLT |
| | 6) Injection site joint inflammation | |
| | 7) Injection site joint movement impairment | |
| | 8) Injection site joint pain | |
| | 9) Injection site joint swelling | |
| | 10) Injection site joint warmth. | |
| | Patients with TEAE of injection site reactions will be categorized into 3 groups: patients with 1 TEAE of injection site reaction event, patients with 2 or 3 events, and patients with ≥4 events. Redness (Scored 0-4) • [0] Subject's normal skin color, no increased redness • [1] Noticeable, but very mild redness • [2] Clearly red | Period (Safety Population): TEAE identified by the investigator by PT within HLT TEAE identified by the investigator by maximum severity by PT within HLT |
| | • [3] Bright red | TEAE identified by the |
| | • [4] Dark with some scar formation | investigator by max redness |
| | Swelling (Scored 0-4 after running a finger over injected area) | category within HLT |
| | • [0] No bump | TEAE identified by the |
| | • [1] Barely noticeable | investigator by max swelling |
| | • [2] Clear bump but very thin | category within HLT |
| | • [3] Clear bump 1 mm thick | TEAE identified by the |
| | • [4] Clear bump 2 mm thick or more | investigator by max pain |
| | Pain (including burning) (Scored 0-3) | category within HLT |
| | • [1] Mild | |
| | • [2] Moderate | |
| | • [3] Severe | |

| <b>Special Safety</b> | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| Cerebro- | Cerebro-cardiovascular events will be externally adjudicated by the CEC at the Cleveland Clinic, as | Open-Label Treatment |
| cardiovascular | outlined in the Manual of Operations. The CEC will adjudicate investigator-reported events selected for | Period (Safety Population): |
| Events | adjudication and render an assessment as to whether the event represents a confirmed event (meeting the | TEAE by PT within |
| | event definition with all necessary documentation), a non-event (does not meet the event definition and | Subcategory |
| | likely represents an alternative or nonevent diagnosis), or lacks sufficient documentation for confirmation | |
| | of an event. All events which qualify for CEC adjudication will be used for the analysis of cerebro- | |
| | cardiovascular events. The categories and subcategories of adjudicated events used for the analysis will | |
| | include the following: | |
| | Cardiovascular | |
| | o Death (Cardiovascular) | |
| | o MI | |
| | Hospitalization for Unstable Angina | |
| | Hospitalization for Heart Failure | |
| | o Serious Arrhythmia | |
| | Hospitalization for Hypertension | |
| | Resuscitated Sudden Death | |
| | Cardiogenic Shock due to Myocardial Infarction | |
| | o Coronary Revascularization | |
| | Neurologic | |
| | o Cerebrovascular Event: Transient Ischemic Attack or Stroke (Hemorrhagic, Ischemic, and | |
| | Undetermined) | |
| | Peripheral Vascular Events | |
| | o Peripheral Arterial Event | |
| | o Peripheral Revascularization | |
| | Events will be analyzed using MedDRA PT nested within the CEC assessment (confirmed event, no | |
| | event, or insufficient documentation for event determination) and the subcategory. Subcategories of | |
| | stroke (Hemorrhagic Stroke, Ischemic Stroke, and Unknown Stroke Type) will be displayed in the | |
| | analyses nested within stroke. Subcategories of Serious Arrhythmia (Atrial Arrhythmia, Ventricular | |
| | Arrhythmia, Heart Block, Other, Unknown) will be displayed nested within Serious Arrhythmia. | |
| MACE | MACE (requiring adjudication as defined above) is defined as: | Open-Label Treatment |
| | Vascular death (including cardiovascular and cerebro-vascular causes excluding hemorrhagic deaths | Period (Safety Population): |
| | outside of the central nervous system) | TEAE by maximum severity |
| | Non-fatal myocardial infarction | PT within Category |

| Special Safety | | |
|---|---|---|
| Topic | Definition/Derivation | Analysis/Summary/Listing |
| Торіс | <ul> <li>Non-fatal stroke (subcategories: ischemic, hemorrhagic, unknown stroke type)</li> <li>Where,</li> <li>Vascular death should be captured as an Event on Adjudication - Death eCRF page with Adjudication Death Type = "Cardiovascular."</li> <li>Non-fatal myocardial infarction should be captured as an Event on Adjudication - Cardiac Ischemic Event eCRF page with Type of Ischemic Event = "Myocardial Infarction" and the Event is NOT on Adjudication - Death eCRF page.</li> <li>Non-fatal strokes (ischemic, hemorrhagic) should be captured as an Event on Adjudication - Cerebrovascular Event eCRF page with Stroke Cerebrovascular Event Subtype in one of the following</li> </ul> | Analysis/Summary/Listing |
| | categories: hemorrhagic stroke, ischemic stroke, undetermined stroke type, and the Event is NOT on <i>Adjudication - Death</i> eCRF page. Subcategories of non-fatal stroke (Hemorrhagic Stroke, Ischemic Stroke, and Undetermined Stroke Type) will be displayed nested within non-fatal stroke category. | |
| Malignancies | Malignancy is defined using PTs from the Malignant or unspecified tumors SMQ as defined in MedDRA (SMQ: 20000091, which includes the sub-SMQs: (1) 20000194 [Malignant tumours], including sub-SMQs of 20000227 [Haematological malignant tumours] and 20000228 [Non-haematological malignant tumours]; (2) 20000195 [Tumours of unspecified malignancy], including sub-SMQs of 20000229 [Haematological tumours of unspecified malignancy] and 20000230 [Non-haematological tumours of unspecified malignancy]. Events will be summarized by the following categories: NMSC Basal Cell Carcinoma, PTs include: Basosquamous carcinoma Basosquamous carcinoma of skin Squamous Cell Carcinoma, PTs include: Squamous cell carcinoma of skin Bowen's disease Lip squamous cell carcinoma Skin squamous cell carcinoma metastatic Keratoacanthoma Malignancies excluding NMSC: all PTs in the Malignant or unspecified tumors SMQ excluding the 8 defined NMSC PTs. | Open-Label Treatment Period (Safety Population): TEAE by PT within Category |
| Depression | Depression and suicide/self-injury is defined using the PTs from the Depression and suicide/self-injury SMQ as specified in MedDRA (SMQ: 20000035, which includes the sub-SMQs: 20000037 | Open-Label Treatment Period (Safety Population): |

| Special Safety<br>Topic | Definition/Derivation | Analysis/Summary/Listing |
|---|---|---|
| | [Suicide/self-injury] and 20000167 [Depression (excluding suicide and self-injury)]). | TEAE by PT within SMQ |
| IBD | IBD will be identified using the following subcategory and MedDRA PTs. The narrow terms are considered IBD. Medical reviews of patients identified with broad terms are needed for final determination of patients with IBD. IBD Specific Terms (Narrow terms) Inflammatory Bowel Disease: Inflammatory bowel disease Crohn's Disease: Crohn's disease Ulcerative Colitis: Acute hemorrhagic ulcerative colitis; Colitis ulcerative; Proctitis ulcerative IBD Non-Specific Terms: The PTs in this category are listed in Appendix 11. | Open-Label Treatment Period (Safety Population): TEAE by PT within subcategory |
| ILD | ILD is defined using the following terms: Narrow terms in the Interstitial lung disease SMQ (20000042) Additional 6 PTs from Eosinophilic pneumonia SMQ (20000157): Angiolymphoid hyperplasia with eosinophilia (Narrow) Eosinophilic bronchitis (Narrow) Hypereosinophilic syndrome (Narrow) Loeffler's syndrome (Narrow) Pulmonary eosinophilia (Narrow) Pulmonary vasculitis (Narrow) | Open-Label Treatment Period (Safety Population): TEAE by PT by maximum severity by PT within interstitial lung disease |

Abbreviations: AE = adverse event; AESI = adverse event of special interest; ALP = alkaline phosphatase; ALT = alanine aminotransferase; AST = aspartate aminotransferase; CEC = Central Events Committee; eCRF = electronic case report form; eDISH = Evaluation of Drug-Induced Serious Hepatotoxicity; GGT = gamma-glutamyltransferase; HLT = High Level Term; IBD = inflammatory bowel disease; ILD = Interstitial Lung Disease; ITT = intent-to-treat; MACE = Major Adverse Cerebro-Cardiovascular Events; MedDRA = Medical Dictionary for Regulatory Activities; MI = myocardial infarction; NMSC = Nonmelanoma Skin Cancer; OI = opportunistic infection; PsA = psoriatic arthritis; PT = preferred term; SAE = serious adverse event; SMQ = standardized MedDRA query; SOC = System Organ Class; TB = tuberculosis; TEAE = treatment-emergent adverse event; ULN = upper limit of normal.

#### 6.15.4. Clinical Laboratory Evaluation

Laboratory evaluations will be summarized and analyzed for the following periods:

- Open-Label Treatment Period (Safety Population)
- Post-Treatment Follow-Up Period (Post-Treatment Follow-Up Population)

Laboratory analyses will include planned analytes only. Planned analytes are those specified in the protocol. However, unplanned/unscheduled measurements of planned analytes will be included/ excluded as specified in the relevant sections. Examples of unplanned/unscheduled measurements include those that the clinical investigator orders as a repeat test or "retest" of a laboratory test if he or she has received an abnormal value, and those the investigator orders for a "follow-up visit" due to clinical concerns.

Laboratory test observed values at each visit (starting at baseline) and change from baseline to each visit will be displayed in box plots (with outliers displayed) for patients who have both a baseline and at least 1 post-baseline result for Period 2 and Period 3, respectively. Baseline will be the last nonmissing observation in the baseline period. Original-scale data will be used for the display. Unscheduled visits and repeat measurements will be excluded. In each of the plots displaying values at each visit, lines indicating the performing lab reference ranges will be added. Displays using both standard (SI) and conventional (CN) units will be provided (when different). The following summary statistics will be included in a table below the box plot: N, mean, standard deviation, minimum, Q1, median, Q3, and maximum. P-values and confidence limits will not be included in the summary statistics at the bottom of the box plot. Box plots will be used to evaluate trends over time and to assess a potential impact of outliers on central tendency summaries.

The number and percentages of patients with treatment-emergent abnormal, high, or low laboratory results at any time will be summarized by treatment for the treatment period. Scheduled visits, unscheduled visits, and repeat measurements will be included. Performing lab reference ranges will be used to define the low and high limits.

- Categorical laboratory tests:
  - A treatment-emergent **abnormal** result is defined as a change from normal at all baseline visits to abnormal at any time during the treatment period.
- Numerical laboratory tests:
  - o A treatment-emergent **high** result is defined as a change from a value less than or equal to the high limit at all baseline visits to a value greater than the high limit at any time during the treatment period.
  - o A treatment-emergent **low** result is defined as a change from a value greater than or equal to the low limit at all baseline visits to a value less than the low limit at any time during the treatment period.

Alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, alkaline phosphatase (ALP), neutrophils, leukocytes, platelets, and lymphocytes will not be included in this treatment-emergent abnormal, high, or low laboratory results analysis. A separate analysis

to address the risk of liver injury is described in Table RHCF.6.7 in which performing lab reference ranges will be used.

By-patient listing of abnormal laboratory test results (criteria defined in the shift tables excluding the normal category) for parameters of special interest (hepatic, leukocytes, and platelets) will be provided.

#### 6.15.4.1. Leukocytes (White Blood Cells) and Platelets

Further analyses will be conducted for total leukocytes, neutrophils, platelets, lymphocytes, monocytes, eosinophils, and basophils. Neutrophils will include both segmented neutrophils and absolute neutrophils (derived by adding segmented neutrophils and band neutrophil). The segmented neutrophils and absolute neutrophils will be summarized using the same categories.

Shift tables will be produced showing the number and percentage of patients with a minimum post-baseline result for neutrophils, lymphocytes (including Th17 lymphocytes), platelets, and leukocytes, and will be summarized overall and by treatment group and baseline result. Unless otherwise specified, neutrophils will be summarized for absolute neutrophils. Scheduled visits, unscheduled visits, and repeat measurements will be included. Baseline is defined as the minimum result during the defined baseline period.

The following LLNs will be defined for the analyses:

- Leukocytes: LLN= $4.0 \times 10^9$ /L
- Neutrophils: LLN= $2.0 \times 10^9$ /L
- Lymphocytes: LLN= $1.1 \times 10^9$ /L
- Platelets: LLN= $150 \times 10^9$ /L

Such shift tables will be produced using the following categories:

- Neutrophils:  $\ge 1 \times LLN$  (Normal), < LLN to  $\ge 1.5 \times 10^9/L$  (Grade 1),  $< 1.5 \times 10^9/L$  to  $\ge 1.0 \times 10^9/L$  (Grade 2),  $< 1.0 \times 10^9/L$  to  $\ge 0.5 \times 10^9/L$  (Grade 3), and  $< 0.5 \times 10^9/L$  (Grade 4).
- Leukocytes:  $\ge 1 \times LLN$  (Normal), < LLN to  $\ge 3.0 \times 10^9/L$  (Grade 1),  $< 3.0 \times 10^9/L$  to  $\ge 2.0 \times 10^9/L$  (Grade 2),  $< 2.0 \times 10^9/L$  to  $\ge 1.0 \times 10^9/L$  (Grade 3), and  $< 1.0 \times 10^9/L$  (Grade 4).
- Platelets:  $\ge 1 \times LLN$  (Normal), < LLN to  $\ge 75.0 \times 10^9/L$  (Grade 1),  $< 75.0 \times 10^9/L$  to  $\ge 50.0 \times 10^9/L$  (Grade 2),  $< 50.0 \times 10^9/L$  to  $\ge 25.0 \times 10^9/L$  (Grade 3), and  $< 25.0 \times 10^9/L$  (Grade 4).
- Lymphocytes:  $\ge 1 \times LLN$  (Normal), < LLN to  $\ge 0.8 \times 10^9/L$  (Grade 1),  $< 0.8 \times 10^9/L$  to  $\ge 0.5 \times 10^9/L$  (Grade 2),  $< 0.5 \times 10^9/L$  (Grade 3), and  $< 0.2 \times 10^9/L$  (Grade 4).

In addition, for the above parameters (neutrophils, leukocytes, platelets, and lymphocytes), the number and percentage of patients with minimum post-baseline results will be presented overall and by treatment within the following group using the categories as defined above:

- Decreased: post-baseline category < baseline category
- Increased: post-baseline category > baseline category
- Same: post-baseline category = baseline category

The number and percentages of patients with treatment-emergent low laboratory results at any time will be summarized for these 4 measures by treatment group for the Open-Label Treatment Period (Period 2) and Post-Treatment Follow-Up Period (Period 3). Shift tables will be produced showing the number and percentage of patients with a minimum post-baseline result for these 4 measures and will be summarized overall and by treatment group and baseline result.

The change from minimum baseline to minimum post-baseline result for each of these leukocytes and platelets will be summarized graphically using a box plot for Safety Population in Period 2.

#### 6.15.4.2. Neutrophil Follow-Up

Neutrophil counts will be followed throughout the study. Patients will continue to be followed in Period 3 until their neutrophil counts have recovered.

The neutrophil follow-up analysis will be conducted on the Neutrophil Follow-Up Population defined as patients who have an absolute neutrophil count <1500 cells/ $\mu$ L (SI units: <1.5 × 10<sup>9</sup>/L) at the last scheduled visit or early termination visit prior to entering the Post-Treatment Follow-Up Period (Period 3) and less than the patient's baseline absolute neutrophil count (that is, prior to first injection at Week 0). These patients are monitored during the Period 3 until neutrophil recovery.

Neutrophil clinical recovery is defined as an absolute neutrophil count  $\geq 1500$  cells/ $\mu$ L (SI units:  $\geq 1.5 \times 10^9$ /L) or greater than or equal to a patient's minimum absolute neutrophil count prior to first study drug injection at Week 0.

If a patient's neutrophil count has not recovered, within 12 weeks after entering the follow-up period (Visit 802), the patient will return for Visit 803 (12 weeks after Visit 802). Additional visits may be required for appropriate patient management depending upon the degree of neutropenia. If at Visit 802, a patient has met the criteria for neutrophil recovery, the patient's participation in the study will be considered complete, unless the investigator deems additional follow-up may be necessary.

The number and percentage of patients achieving neutrophil clinical recovery will be presented by dosing regimen and week interval for Neutrophil Follow-Up Population in the Post-Treatment Follow-Up Period (Period 3). The number and percentage of patients with an absolute neutrophil cell count that is at least 25%, 50%, 75%, or 100% of the patient's baseline absolute neutrophil count (that is, prior to first injection at Week 0), irrespective of absolute neutrophil minimum, will be included in the summary.

## 6.15.5. Vital Signs and Other Physical Findings

Vital signs and physical characteristics will be summarized and analyzed for the following periods:

- Open-Label Treatment Period (Safety Population)
- Post-Treatment Follow-up Period (Post-Treatment Follow-Up Population)

For vital signs and physical characteristics, the observed values at each visit (starting at baseline) and change from baseline to each scheduled visit, respectively, will be displayed in box plots for patients who have both baseline and at least 1 post-baseline result. Baseline will be the last nonmissing observation in the baseline period. Original-scale data will be used for the display. Unscheduled visits and repeat measurements will be excluded. Reference limits will not be displayed. The following summary statistics will be included in a table below the box plot: N, mean, standard deviation, minimum, Q1, median, Q3, and maximum. P-values and confidence limits will not be included in the summary statistics at the bottom of the box plot. Box plots will be used to evaluate trends over time and to assess a potential impact of outliers on central tendency summaries.

The frequency and percentages of patients with treatment-emergent high or low vital signs and physical characteristics results at any time will be summarized by treatment group for Period 2 and Period 3, respectively.

- A treatment-emergent **high** result is defined as a change from a value less than or equal to the high limit at all baseline visits to a value greater than the high limit at any time that meets the specified change criteria during the treatment period.
- A treatment-emergent **low** result is defined as a change from a value greater than or equal to the low limit at all baseline visits to a value less than the low limit at any time that meets the specified change criteria during the treatment period.

Table RHCF.6.8 will be used to define the low and high baseline values as well as the limits that are specified as treatment emergent. Note: Weight does not have an abnormal baseline; therefore, the treatment-emergent values are determined by change from baseline. For categorical variables, scheduled visits, unscheduled visits, and repeat measurements will be included.

Table RHCF.6.8. Categorical Criteria for Abnormal Treatment-Emergent Blood Pressure and Pulse Measurement, and Categorical Criteria for Weight and Changes for Adults

| Parameter | Low | High |
|---|---|---|
| Systolic BP (mm Hg) <sup>1</sup> (supine or sitting – forearm at heart level) | ≤90 and decrease from baseline ≥20 | ≥140 and increase from baseline ≥20 |
| Diastolic BP (mm Hg) <sup>1</sup> (supine or sitting – forearm at heart level) | ≤50 and decrease from baseline ≥10 | ≥90 and increase from baseline ≥10 |
| Pulse (bpm) <sup>1</sup> (supine or sitting) | <50 and decrease from baseline ≥15 | >100 and increase from baseline ≥15 |
| Weight (kg) | (Loss) decrease from baseline ≥7% | (Gain) increase from baseline ≥7% |

Abbreviations: BP = blood pressure; bpm = beats per minute.

#### 6.15.6. Columbia-Suicide Severity Rating Scale

The Columbia-Suicide Severity Rating Scale (C-SSRS) is an assessment tool that evaluates suicidal ideation and behavior. Information on the C-SSRS scale can be found through the following link: http://www.cssrs.columbia.edu.

Specifically, the following outcomes are C-SSRS categories and have binary responses (yes/no). The categories have been re-ordered from the actual scale to facilitate the definitions of the composite and comparative endpoints and to enable clarity in the presentation of the results.

Category 1 – Wish to be Dead

Category 2 – Non-specific Active Suicidal Thoughts

Category 3 – Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act

Category 4 – Active Suicidal Ideation with Some Intent to Act, without Specific Plan

Category 5 – Active Suicidal Ideation with Specific Plan and Intent

Category 6 – Preparatory Acts or Behavior

Category 7 – Aborted Attempt

Category 8 – Interrupted Attempt

Category 9 – Actual Attempt (non-fatal)

Category 10 – Completed Suicide.

Self-injurious behavior without suicidal intent is also a C-SSRS outcome (although not suicide related) and has a binary response (yes/no).

Composite endpoints based on the above categories are defined below.

- Suicidal ideation: A "yes" answer at any time during treatment to any 1 of the 5 suicidal ideation questions (Categories 1-5) on the C-SSRS.
- **Suicidal behavior:** A "yes" answer at any time during treatment to any 1 of the 5 suicidal behavior questions (Categories 6-10) on the C-SSRS.

<sup>1</sup> Baseline abnormal values are defined by the value presented.

• Suicidal ideation or behavior: A "yes" answer at any time during treatment to any 1 of the 10 suicidal ideation and behavior questions (Categories 1-10) on the C-SSRS.

The Self-Harm Supplement Form is a 1-question form that is completed, at any visit, including baseline visit, that asks for the number of suicidal behaviors, possible suicidal behaviors, or nonsuicidal self-injurious behaviors the patient has experienced since the last assessment. For each unique event identified, a questionnaire (Self-Harm Follow-Up Form) that collects supplemental information on the self-injurious behavior is to be completed.

Change from baseline to each post-baseline visit in C-SSRS total score will be analyzed using MMRM methods for the safety population during Period 2. If the number of patients in analysis is less than 10% of patients in total, only a by-patient listing will be provided.

The C-SSRS will be listed by patient and visit. Only patients that show suicidal ideation/behavior or self-injurious behavior without suicidal intent will be displayed (that is, if a patient's answers are all "no" for the C-SSRS, then that patient will not be displayed). However, if a patient reported any suicidal ideation/behavior or self-injurious behavior without suicidal intent at any time point, then all ideation and behavior for that patient will be displayed, even if not positive. Note, missing data should not been imputed.

The Self-Harm data will be listed by patient and visit if number of events on Self-Harm Supplement Form is not zero in the CRF "Self-Harm Questionnaire Supplement."

#### 6.15.7. Immunogenicity

Not applicable.

## 6.15.8. Electrocardiograms

Not applicable.

## 6.16. Subgroup Analyses

## 6.16.1. Safety Subgroup Analyses

Safety subgroup analysis for common TEAEs and AESIs of allergy/hypersensitivity, infections, and injection site reactions will be summarized by treatment and overall, during the Open-Label Treatment Period for the safety population.

Subgroups to be evaluated include the following:

- Patient Demographic Subgroups:
  - o Sex: female or male
  - o Age group: <65 years, or  $\ge 65$  years
- Geographic Region Subgroups:
  - o Geographic region: Europe, Rest of the World
- Concomitant Therapy:
  - o Concomitant csDMARD use at baseline: yes or no
  - o Concomitant methotrexate use at baseline: yes or no

- o Concomitant glucocorticoids use at baseline: yes or no
- Baseline Severity Groups:
  - o Moderate-to-severe plaque psoriasis involvement: yes or no

Treatment effects will be assessed within the subgroups using the Fisher's exact test. The most common TEAEs and AESI will be presented by MedDRA PT nested within SOC (SMQ or High Level Term where specified). A logistic regression model will be used to test the treatment-by-subgroup interaction. The response variable will be each AE. The explanatory variables will be treatment, subgroup, and treatment by-subgroup interaction. The interaction test will be evaluated at the 0.10 significance level. If any of the subgroups (for example, the age <65 group or the age ≥65 group) is less than 10% of the total population, only descriptive statistics will be provided for that subgroup (that is, no inferential testing).

## 6.16.2. Efficacy Subgroup Analyses

Subgroup analyses will be conducted for the following efficacy assessments:

 ACR50 and PASI 100 simultaneous response rate at Week 24 with ITT Population in the Open-Label Treatment Period

Subgroups to be evaluated include the following:

- Patient Demographic Subgroups:
  - Age group: <65 years or  $\ge 65$  years
  - o Ethnicity: Hispanic or Latino, Non-Hispanic and Non-Latino
- Geographic Region Subgroups:
  - o Geographic region: Europe, Rest of the World
- Concomitant Therapy:
  - o Concomitant csDMARD use at baseline: yes or no
  - o Concomitant methotrexate use at baseline: ves or no
  - o Concomitant glucocorticoids use at baseline: yes or no
  - o Number of prior csDMARD therapies: 1, 2, 3, or > 3
- Baseline Severity Groups:
  - o Moderate-to-severe plaque psoriasis involvement: yes or no

Additional exploratory subgroup analyses will be conducted for the following efficacy assessments:

- ACR20, 50, and 70 response rates at Week 24 with ITT population in the Open-Label Treatment Period
- PASI 75, 90, and 100 response rates at Week 24 with ITT population in the Open-Label Treatment Period

Subgroup to be evaluated includes:

- Concomitant Therapy:
  - o Concomitant csDMARD use at baseline: yes or no
  - o Concomitant methotrexate use at baseline: yes or no

- Baseline Severity Groups:
  - o Moderate-to-severe plaque psoriasis involvement: yes or no

A logistic regression model with treatment, subgroup, and the interaction of treatment-by-subgroup included as factors will be used. The treatment-by-subgroup interaction will be tested at the significance level of 0.10. Treatment group effects will be evaluated within each category of the subgroup using Fisher's exact test, regardless of whether the interaction is statistically significant. Missing data will be imputed using NRI, as described in Section 6.4.1. The treatment differences with 95% CIs by each subgroup category will be reported. If any of the subgroups (for example, the age <65 group or the age  $\ge65$  group) is less than 10% of the total population, only descriptive statistics will be provided for that subgroup (that is, no inferential testing).

#### 6.17. Protocol Violations

Protocol deviations will be identified throughout the study. Important protocol deviations are defined as those violations from the protocol likely to have a significant impact on the completeness, accuracy, and/or reliability of the study data or that may significantly affect a subject's rights, safety, or well-being.

Table RHCF.6.9 includes the categories and subcategories of important protocol violations, the source of identification for the violation, and the statistical programming guidance for the CSR.

A by-patient listing of important protocol deviations will be provided for all entered patients.

The number and percentage of patients having important protocol violation(s) will be summarized within category and subcategory of violations by treatment group for the following:

• Open-Label Treatment Period (ITT Population)

Additional analyses will be conducted on patients who don't have any or a subset of protocol violations for primary and/or major secondary endpoints.

 Table RHCF.6.9.
 Identification and Action of Important Protocol Violations

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| Category: Informed Consent | | |
| Sub-Category: Informed Consent not | Monitor and Stats | Either from monitor's list, or, |
| Obtained/Missing/Late | | If patient informed consent date is after Visit 1 date |
| | | or missing informed consent |
| Subcategory: Improper Informed Consent | Monitor | Monitor's list |
| Category: Eligibility | | |
| [1] Age <18 years | Monitor | Monitor's list |
| [1a] Male patients disagree to use a reliable method of | Monitor | Monitor's list: male patients who disagree to use a |
| birth control during the study. | | reliable method of birth control during the study. |
| [1b] Pregnancy confirmation at Visit 1 and prior to | Monitor | Monitor's list: positive pregnancy test result from |
| randomization at Visit 2. | | lab test at Visit 1, and check if patient was |
| | | randomized and takes drug. Check Visit 2 urine |
| | | pregnancy test. |
| [1b] Are women ≥40 and <60 years of age who have | Monitor and Stats | Monitor's list: Women ≥40 and <60 years of age |
| had a cessation of menses for at least 12 months, and | | who do not have negative bHCG results and who |
| FSH <40 mIU/mL | | have a FSH <40 mIU/mL at Visit 1. |
| [1b] Are women of non-childbearing potential, defined | Monitor | Monitor's list: women who have had surgical |
| as either women who have had surgical sterilization or | | sterilization. |
| who are ≥60 years of age | | |
| [2] No confirmed diagnosis of PsA of at least 6 | Monitor | Monitor's list |
| months prior to baseline or did not meet CASPAR | | |
| criteria | | |
| [3] <3 TJC or <3 SJC at Visit 1 or 2 | Monitor | Monitor's list. |
| | Monitor and Stats | Monitor's list. |
| [4] BSA <3% at Visit 1 or 2 | Womtor and Stats | Check if BSA < 3% either at Visit 1 or at Visit 2 |
| [50] Have not been treated with 1 or more csDMARDs | Monitor and Stats | Monitor's list and stats programming. |
| [30] Have not been treated with 1 of more CSDMARDS | Womtor and Stats | Check past or present use for MTX, sulfasalazine, |
| | | leflunomide, or hydroxychloroquine |
| | | remunormae, or nyaroxycmoroquine |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [6] Currently enrolled in any other clinical trial | Monitor | Monitor's list. |
| involving an investigational product or any other type | | |
| of medical research judged not to be scientifically or | | |
| medically compatible with this study | | |
| [7] Have received prior or currently receiving | Monitor | Monitor's list |
| treatment with any biologic or small molecule therapy | | |
| for PsA or Ps, including investigation therapies (such | | |
| as, but not limited to, a TNF inhibitor, IL-1 receptor | | |
| antagonists, IL-6 inhibitor; anti-IL-12/23p40, T cell or | | |
| B cell targeted therapies, or Janus kinase inhibitors). | | |
| Note: previous treatment of phosphodiesterase type 4 | | |
| inhibitors will be permitted. Treatment with | | |
| phosphodiesterase type 4 inhibitors must have been | | |
| discontinued at least 8 weeks before randomization | | |
| (Visit 2). | | |
| [8] Previous or current medication exposure at Visit 1 | Monitor | Monitor's list |
| to LY2439821 or IL-17 antagonists or previous | | |
| participation in the current study. | | |
| (Note: See protocol for patients who may be allowed | | |
| to re-screen.) | | |
| [9] Have history of drug-induced Ps. | Monitor | Monitor's list |
| [10] Use of csDMARDs (other than MTX, | Monitor | Monitor's list |
| leflunomide, sulfasalazine, or cyclosporinein) within 8 | | |
| weeks prior to Visit 2; or have discontinued MTX, | | |
| leflunomide, sulfasalazine, or cyclosporine within 12 | | |
| weeks prior to Visit 2. | | |
| [11] Have discontinued leflunomide within 4 weeks | Monitor and Stats | Monitor's list, or, |
| prior to Visit 2 or from 4 to 12 weeks prior without | | If the difference between Visit 2 date and medication |
| drug elimination procedure. | | end date <28 days for previous therapy, Leflunomide |
| [12] Use of oral corticosteroids at average daily doses | Monitor | Monitor's list |
| of >10 mg/day of prednisone or equivalent, use of | | |
| variable doses within 4 weeks prior to Visit 2. | | |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [13] Have received parenteral glucocorticoids within 6 weeks prior to Visit 2 or if use is anticipated during the first 24 weeks of open-label treatment period (Period 2) of the study | Monitor and Stats | Monitor's list, or, If a patient has a reported previous therapy of parenteral glucocorticoids with and either a start or end date <42 days prior to the Visit 2 date |
| [14] Concomitant use of NSAIDs or cyclooxygenase - 2 inhibitors unless on a stable dose for at least 2 weeks prior to Visit 2 | Monitor | Monitor's list |
| [15] Use of opiate analgesics at average daily doses of >30 mg/day of morphine or equivalent or variable doses within 6 weeks prior to Visit 2 | Monitor and Stats | Monitor's list, or, If a patient has either a reported previous therapy of opiate analgesics with average dose >30 mg/day or a concomitant medication with ATC codes of N02AA with a start or end date of <42 days prior to Visit 2 date. |
| [16] Have received systemic nonbiologic Ps therapy other than csDMARDs or corticosteroids as indicated above (including, but not limited to oral psoralens and ultraviolet A light therapy oral retinoids, thioguanine, hydroxyurea, sirolimus, azathioprine, fumaric acid derivatives, or 1, 25 dihydroxy vitamin D3 and analogs) or phototherapy (including either oral and topical ultraviolet A, ultraviolet B, or self-treatment with tanning beds or therapeutic sunbathing) within 4 weeks prior to randomization (Visit 2); or had topical Ps treatment within the previous 2 weeks prior to randomization (Visit 2). Note WHO Group 1 weak potency topical steroids are allowed. | Monitor and Stats | Monitor's list, or, If the patient has any record with a start date or an end date <28 days of the Visit 2 date for phototherapy for previous therapy. If the patient has any concomitant medications with a start date or an end date that is on or prior to Visit 2 date, and <28 days prior to the Visit 2 date for oral medications. If the patient has any concomitant medications with an end date that is on or prior to Visit 2 date, and ≤14 days prior to the Visit 2 date for topical medications. Note: ATC codes will be provided by medical in a separate file. |
| [17] Use of tanning booths for at least 4 weeks prior to Visit 2 and during the study for patients with plaque psoriasis. | Monitor | Monitor's list |
| [18] Have a known allergy or hypersensitivity to any biologic therapy that would pose an unacceptable risk to the patient if participating in this study. | Monitor | Monitor's list |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [19] Ever received efalizumab or natalizumab or other agents that target alpha-4-integrin | Monitor | Monitor's list |
| [20] Have been exposed to a live vaccine within 12 weeks prior to Visit 2 or intend to have a live vaccination during the course of the study, or within 12 weeks of completing treatment in this study, or participated in other vaccine clinical study within 12 weeks prior to Visit 2 | Monitor | Monitor's list |
| [21] Had a BCG (12 months prior to Visit 2), or intent to have this vaccine with BCG during the study or within 12 months of completion of the study | Monitor | Monitor's list |
| [22] Have diagnosis of other inflammatory arthritic syndrome | Monitor | Monitor's list |
| [23] Have active Crohn's disease or active ulcerative colitis | Monitor | Monitor's list |
| [24] Have current diagnosis of fibromyalgia or other chronic pain condition that would confound evaluation of the patient | Monitor | Monitor's list |
| [25] Evidence of active vasculitis or uveitis | Monitor | Monitor's list |
| [26] Surgical treatment of joint within 8 weeks prior to Visit 2 or will require such up to Week 24 | Monitor | Monitor's list |
| [27] Had any major surgery within 8 weeks prior to Visit 2, or will require such during the study that, in the opinion of the investigator in consultation with Lilly or its designee, would pose an unacceptable risk to the patient. | Monitor | Monitor's list |
| [28] Have active or history of malignant disease within the 5 years prior to Visit 2. Note: Patients with successfully treated basal-cell carcinoma (no more than 3), squamous-cell carcinoma of the skin (no more than 2), within the 5 years prior to Visit 2 may participate in the study. | Monitor | Monitor's list |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [29] Presence of significant uncontrolled cerebro- | Monitor | Monitor's list |
| cardiovascular (for example, MI, unstable angina, | | |
| unstable arterial hypertension, moderate-to-severe | | |
| NYHA class III/IV heart failure, or CVA), respiratory, | | |
| hepatic, renal, gastrointestinal, endocrine, | | |
| hematologic, neurologic, or neuropsychiatric | | |
| disorders, or abnormal laboratory values, or illicit drug | | |
| use (including cannabinoids, whether legalized or not) | | |
| at screening that in the opinion of the investigator pose | | |
| an unacceptable risk to the patient if participating in | | |
| the study or of interfering with the interpretation of | | |
| data. | | |
| [30] Have had uncompensated heart failure, fluid | Monitor | Monitor's list |
| overload, or MI, or evidence of new-onset ischemic | | |
| heart disease or other serious cardiac disease within 12 | | |
| weeks prior to Visit 2. | | |
| [31] Presence of significant uncontrolled | Monitor and Stats | Monitor's list, or, |
| neuropsychiatric disorder; have recent history (within | | If a patient has a yes to question 4 or 5 on the |
| 30 days prior to screening visit (Visit 1) and any time | | "Suicidal Ideation" portion of the C-SSRS or |
| between screening visit (Visit 1) and randomization | | develops suicide-related behaviors as recorded on the |
| (Visit 2) of a suicide attempt; or develops active | | C-SSRS at Visits 1 or 2. |
| suicidal ideation with some intent to act with or | | |
| without a specific plan (yes to question 4 or 5 on the | | |
| "Suicidal Ideation" portion of the C-SSRS) or | | |
| develops suicide-related behaviors as recorded on the | | |
| C-SSRS at screening or randomization (Visit 2); or are | | |
| clinically judged by the investigator to be at risk for | | |
| suicide. | | |
| [32] Have presence or personal history or family | Monitor | Monitor's list |
| history (first degree relative) of demyelinating | | |
| disorder. | | |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [33] Have serious infection, been hospitalized, | Monitor | Monitor's list |
| received IV antibiotics for an infection within 12 | | |
| weeks of Visit 2, or had a serious bone or joint | | |
| infection within 24 weeks prior to Visit 2, or have ever | | |
| had an infection of an artificial joint, or an infection | | |
| that occurs with increased incidence in an | | |
| immunocompromised host (including, but not limited | | |
| to, Pneumocystis jirovecii pneumonia, active | | |
| histoplasmosis, or coccidioidomycosis), or have a | | |
| known immunodeficiency. | | |
| [34] Have a known immunodeficiency or are | Monitor | Monitor's list |
| immunocompromised to an extent such that | | |
| participation in the study would pose an unacceptable | | |
| risk to the patient. | | |
| [35] Have or had a herpes zoster or any other clinically | Monitor | Monitor's list |
| apparent varicella-zoster virus infection within 12 | | |
| weeks prior to Visit 2. | | |
| [36] Evidence or suspicion of active or latent TB (refer | Monitor | Monitor's list |
| to RHCF Protocol Section 9.4.4.2 for details on | | |
| determining full TB exclusion criteria). | | |
| [37] Have any other active or recent infection other | Monitor | Monitor's list |
| than mentioned above within 4 weeks of | | |
| randomization (Visit 2) that, in the opinion of the | | |
| investigator, would pose an unacceptable risk to the | | |
| patient if participating in the study. | | |
| Note: These patients may be rescreened once $\geq 4$ | | |
| weeks after documented resolution of symptoms | | |
| [38] Sitting systolic blood pressure >160 mm Hg or | Monitor and Stats | Monitor's list, or, |
| diastolic blood pressure >100 mm Hg. | | If a patient's systolic blood pressure >160 mm Hg or |
| Note: Determined by 2 consecutive elevated readings. | | diastolic blood pressure >100 mm Hg at Visit 2 (pre- |
| | | dose read) |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [39] Are positive for HIV serology (positive for HIV | Monitor and Stats | Monitor's list, or, |
| antibody) | | If a patients laboratory tests at Visit 1 indicate they are positive for HIV antibody |
| [40] Have evidence of or test positive for hepatitis B | Monitor and Stats | Monitor's list; or |
| by any of the following criteria: | | If test positive for HBV at Visit 1 by testing: |
| 1) positive for hepatitis B surface antigen (HBsAg+); | | 1) positive for hepatitis B surface antigen (HBsAg+), |
| 2) positive for anti-hepatitis B core antibody | | OR |
| (HBcAb+) and positive for HBV DNA. | | 2) positive for anti-hepatitis B core antibody |
| Note: Patients who are HBsAg-, and HBcAb+ and | | (HBcAb+) AND are HBV DNA positive. |
| HBV DNA negative may be enrolled in the study. | | Note: If multiple records at Visit 1, use the last |
| Patients who meet these criteria at screening will be | | observation. Patients who are HBsAg- AND |
| identified by the central laboratory and monitored | | HBcAb+ AND HBV DNA negative can be enrolled. |
| during the study as detailed in Section 9.4.5.4 of the | | This would not be a protocol violation. |
| RHCF protocol. | | |
| [41] Have evidence of or test positive for HCV. A | Monitor and Stats | Monitor's list, or, |
| positive test for HCV is defined as: | | If a patient's laboratory tests at Visit 1 indicate they |
| 1) positive for hepatitis C antibody (anti-HCV Ab), | | are positive for HCV. |
| and | | |
| 2) positive via a confirmatory test for HCV (for | | |
| example, HCV polymerase chain reaction). | | |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [42] The most recent lab panel meet any of the | Monitor and Stats | Monitor's list, or, |
| following criteria: | | If a patients laboratory tests at Visit 1 indicate any of |
| [42a] Neutrophil count <1500 cells/μL | | the following: |
| [42b] Lymphocyte count <800 cells/μL | | Neutrophil count <1500 cells/μL |
| [42c] Platelet count <100,000 cells/μL | | Lymphocyte count <800 cells/μL |
| [42d] AST or ALT >2.5× ULN | | Platelet count <100,000 cells/μL |
| [42e] Total WBC count <3000 cells/μL | | AST or ALT >2.5× ULN |
| [42f] Hemoglobin <8.5 g/dL (85.0 g/L) for male | | Total WBC <3000 cells/μL |
| patients and <8.0 g/dL (80 g/L) for female patients | | Hemoglobin <8.5 g/dL for male patients and <8 g/dL |
| [42g] Serum creatinine >2.0 mg/dL. | | for female patients |
| [42h] Have clinical laboratory test results at screening | | Serum creatinine >2 mg/dL |
| that are outside the normal reference range for the | | |
| population and are considered clinically significant, | | |
| per investigator assessment. | | |
| Note: Laboratory tests can be repeated a maximum of | | |
| 1 time, and results must be received and reviewed | | |
| prior to randomization (Visit 2). | | |
| [43] Have any condition or contraindication as | Monitor | Monitor's list |
| addressed in the local labelling for adalimumab that | | |
| would preclude the patient from participating in this | | |
| protocol. | | |
| [44] Have any other condition that precludes the | Monitor | Monitor's list |
| patient from following and completing the protocol. | | |
| [45] Are women who are breastfeeding | Monitor | Monitor's list |
| [46] Are study site personnel directly affiliated with | Monitor | Monitor's list |
| this study and/or their immediate families. Immediate | | |
| family is defined as a spouse, parent, child, or sibling, | | |
| whether biological or legally adopted. | | |
| [47] Are Lilly employees or its designee or are | Monitor | Monitor's list |
| employees of third-party organizations involved in the | | |
| study. | | |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [48] Are currently enrolled in, or discontinued from a | Monitor | Monitor's list |
| clinical trial involving an investigational product or | | |
| nonapproved use of a drug or device within the last 4 | | |
| weeks or a period of at least 5 half-lives of the last | | |
| administration of the drug, whichever is longer, or are | | |
| concurrently enrolled in any other type of medical | | |
| research judged not to be scientifically or medically | | |
| compatible with this study. | | |
| [49] Are unwilling or unable to comply with the use of | Monitor | Monitor's list |
| a data collection device to directly record data from | | |
| the patient. | | |
| Category: Study Procedures | | |
| Sub-Category: Violation of Discontinuation Criteria | | |
| [D1] Discontinuation of the study drug after | Monitor | Monitor's list |
| consultation with medical monitor for abnormal liver | | |
| tests, defined as having 1 of the following: | | |
| ALT or AST >8× ULN | | |
| ALT or AST $>5 \times$ ULN for more than 2 weeks | | |
| ALT or AST $>3 \times$ ULN and total bilirubin level $>2 \times$ | | |
| ULN or prothrombin time $>1.5\times$ ULN | | |
| ALT or AST $>3 \times ULN$ with the appearance of fatigue, | | |
| nausea, vomiting, right upper-quadrant pain or | | |
| tenderness, fever, rash, and/or eosinophilia (>5%) | | |
| ALP >3× ULN | | |
| ALP >2.5× ULN and TBL >2× ULN | | |
| ALP $>2.5 \times$ ULN with the appearance of fatigue, | | |
| nausea, vomiting, right quadrant pain or tenderness, | | |
| fever, rash, and/or eosinophilia (>5%) | | |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [D2] Neutrophil (segmented) counts: <500 cells/μL; or ≥500 and <1000 cells/μL (from 2 test results; the second test must be performed within 1 week from knowledge of the initial result); or ≥1000 and <1500 cells/μL (from 3 test results) and an infection that is not fully resolved | Monitor and Stats | Monitor's list, or, If a patient still receives study treatment after 10 days of latest dose with confirmed segmented neutrophil counts <500 cells/µL; ≥500 and <1000 cells/µL (from a test and a re-test result; the re-test must be performed within 1 week from knowledge of the initial result); or ≥1000 and <1500 cells/µL (from a test and 2 re-test results) and an infection that is not fully resolved If there are missing re-test results, use the non-missing results |
| [D3] Total WBC count <2000 cells/μL | Monitor and Stats | Monitor's list, or, If a patient still receives study treatment after 10 days of latest dose with confirmed total WBC count <2000 cells/µL (defined as a test and a retest within 10 days); If no retest, use the test results |
| [D4] Lymphocyte count <500 cells/μL | Monitor and Stats | Monitor's list, or, If a patient still receives study treatment after 10 days of latest dose with confirmed lymphocyte count <500 cells/μL (defined as a test and a retest within 10 days) If no retest, use the test results |
| [D5] Platelet count <50,000 cells/μL | Monitor and Stats | Monitor's list, or, If a patient still receives study treatment after 10 days of latest dose with confirmed platelet count <50,000 cells/μL (defined as a test and a re-test within 10 days) If no retest, use the test results |
| [D6] Changes in BP defined as sitting systolic BP at ≥160 mm Hg plus ≥20 mm Hg increase from baseline (Week 0, Visit 2) and/or diastolic BP at ≥100 mm Hg plus ≥10 mm Hg increase from baseline that do not respond following maximal allowed intervention. | Monitor | Monitor's list |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [D7] If the investigator decides that the patient should<br>be withdrawn because of a severe AE, an SAE, or a<br>clinically significant change in a laboratory value, the<br>investigational product is to be discontinued, and | Monitor | Monitor's list |
| appropriate measures are to be taken. Lilly or its designee is to be alerted immediately. | | |
| [D8] Patient has a clinically significant systemic hypersensitivity reaction after SC administration of investigational product | Monitor | Monitor's list |
| [D9] Patient becomes pregnant | Monitor | Monitor's list |
| [D10] The patient develops a malignancy. (No more than 2 nonmelanoma skin cancers over any 12-month period during the study.) | Monitor | Monitor's list |
| [D11] Patient develops symptoms suggestive of a lupus-like syndrome or is positive for antibodies against double-stranded DNA | Monitor | Monitor's list |
| [D12] If the patient for any reason requires treatment with another therapeutic agent that has been demonstrated to be effective for the treatment of PsA. | Monitor | Monitor's list |
| [D13] Enrollment in any other clinical trial involving<br>an investigational product or enrollment in any other<br>type of medical research judged not to be scientifically<br>or medically compatible with this study | Monitor | Monitor's list |
| [D14] The patient develops active suicidal ideation with some intent to act with or without a specific plan (yes to question 4 or 5 on the "Suicidal Ideation" portion of the C-SSRS) or develops suicide-related behaviors as recorded on the C-SSRS. | Monitor and Stats | Monitor's list, or, If patient still receives study treatment on the same day or after the date with a yes to question 4 or 5 on the "Suicidal Ideation" portion of the C-SSRS or develops suicide-related behaviors as recorded on the C-SSRS. |
| [D15] The patient develops any condition or contraindication as addressed in the local labelling for adalimumab that would preclude the patient from continuing in this study protocol. | Monitor | Monitor's list |

| Important Protocol Violation | Source to Identify Protocol | Statistical Programming Guidance for Clinical |
|---|---|---|
| Category/Subcategory | Violation | Study Report |
| [D16] The investigator decides that the patient should | Monitor | Monitor's list |
| be withdrawn from the study | | |
| [D17] The patient requests to be withdrawn from the | Monitor | Monitor's list |
| study | | |
| [D18] The investigator or Lilly stops the patient's | Monitor | Monitor's list |
| participation in the study or Lilly stops the study for | | |
| medical, safety, regulatory, or other reasons consistent | | |
| with applicable laws, regulations, and GCP. | | |
| [D19] The patient becomes HBV DNA positive. | Monitor | Monitor's list |
| [D20] The patient is diagnosed with an active TB | Monitor | Monitor's list |
| infection. | | |
| Category: Study Procedures | | |
| Sub-Category: Excluded Con-meds | Monitor and Stats | Either from monitor's list, or If patient takes |
| | | prohibited concomitant medication. |
| | | Note: Prohibited concomitant medication (with |
| | | details of dose restrictions) will be provided by |
| | | medical in a separate file. |
| Sub-Category: Lab/Imaging Criteria | | |
| Missing lab chemistry and hematology: missing | Monitor and Stats | Monitor's list; or |
| baseline or not having at least 1 post-baseline | | If missing lab chemistry and hematology baseline or |
| | | not having at least 1 post-baseline |
| Sub-Category: Other | | |
| Missing ACR or PASI | Monitor and Stats | Monitor's list; or |
| | | If missing any ACR or PASI data at any visit (Weeks |
| | | 0 through 52). |
| Missing C-SSRS any visit except Visit 1 | Monitor and Stats | From monitor's list; |
| | | if missing C-SSRS at any visit except Visit 1 |
| Had unqualified site personnel perform clinical safety | Monitor | Monitor's list |
| and/or efficacy assessments | | |
| Unblinding of the blinded rater at the site | Monitor | Monitor's list |

| Category: Investigational Product | | |
|---|---|---|
| Sub-Category: Treatment Assignment/Randomizati | on Error | |
| Took incorrect study medication | Monitor and Stats | Monitor's list; or If IWRS study drug dispense data not match with the treatment label identifier on the <i>Exposure as Collected</i> eCRF page |
| Sub-Category: Compliance | Monitor and Stats | Monitor's list; or If non-compliant with study medication regimen or over-dose during the treatment period. Note: Non- compliance with therapy is defined to be missing more than 20% of expected doses and missing 2 or more consecutive doses; over-dose is defined as to take more injections at the same time point than specified in the protocol. |
| Sub-Category: Patient took medication not fit for use | Monitor | Monitor's list |
| Sub-Category: Other | | |
| Randomized but did not take any study medication | Monitor | Monitor's list |
| Sub-Category: Treatment Assignment /Randomization Error | | |
| Stratification error leading to incorrect dosing regimen | Monitor and Stats | Monitor's list; or<br>If IWRS stratification data does not match patients'<br>severity of plaque psoriasis (PASI, sPGA and BSA) |

Abbreviations: AE = adverse event; ACR = America College of Rheumatology; ALT = alanine aminotransferase; AST = aspartate aminotransferase; ATC = anatomical therapeutic chemical; BCG = Bacille de Calmette et Guérin; bDMARD = biologic disease-modifying antirheumatic drug; bHCG = beta-human chorionic gonadotropin; BP = blood pressure; BSA = body surface area; CASPAR = classification for psoriatic arthritis; CRF = case report form; C-SSRS = Columbia Suicide Severity Rating Scale; csDMARD = conventional synthetic disease-modifying antirheumatic drug; CVA = cerebrovascular accident; DNA = deoxyribonucleic acid; ECG = electrocardiogram; eCRF = electronic case report form; FSH = follicle-stimulating hormone; GCP = good clinical practice; HCV = hepatitis C virus; HIV= human immunodeficiency virus; IL = interleukin; IV = intravenous; IWRS = interactive web-response system; JAK = Janus kinase; MI = myocardial infarction; MTX = methotrexate; NSAID = nonsteroidal anti-inflammatory drug; NYHA = New York Heart Association; PASI = Psoriasis Area and Severity Index; Ps = psoriasis; PsA = psoriatic arthritis; PUVA = psoralen ultraviolet A; SAE = serious adverse event; SC = subcutaneous; SJC = swollen joint count; TB = tuberculosis; TJC = tender joint count; TNF = tumor necrosis factor; ULN = upper limit of normal; UVB = ultraviolet B; WBC = white blood cell; WHO = World Health Organization.

The term "Monitor" indicates the protocol deviation will be identified by site monitors and entered into monitor's list using a spreadsheet. The spreadsheet will be exported as Study Data Tabulation Model (SDTM) DV domain.

The term "Stats" indicates the protocol violation will be programmed based on data in clinical database by statistical programmers with the statistical programming guidance provided as the last column. The detailed programming specification will be documented in Analysis Data Model (ADaM) specification.

The terms "Monitor and Stats" indicates the protocol deviation will be a combination of monitor's list (SDTM.DV domain) and statistical programming from clinical database, the deviation will show if either source identifies.

#### 6.18. Interim Analyses and Data Monitoring

An interim database lock will occur, and the analysis will be performed at the time (that is, a cutoff date) when the last patient completes Visit 8 (Week 24), completes ETV, or discontinues from Period 2. This database lock will include all data collected by the cutoff date including data after Week 24 from the Open-Label Treatment Period and follow-up data from patients who have begun Post-Treatment Follow-Up Period (Period 3).

This interim database lock at Week 24 will be considered the primary database lock for this study because all primary and major secondary study objectives will be assessed at this time.

A final database lock will occur after all enrolled patients have completed or discontinued the Post-Treatment Follow-Up Period.

There will be no data monitoring committee.

## 6.19. Clinical Trial Registry Analyses

Additional analyses will be performed for the purpose of fulfilling the Clinical Trial Registry (CTR) requirements.

Analyses provided for the CTR requirements include the following:

Summary of adverse events, provided as a dataset which will be converted to an XML file. Both Serious Adverse Events and "Other" Adverse Events are summarized: by treatment group, by MedDRA PT.

- An adverse event is considered "Serious" whether or not it is a TEAE.
- An adverse event is considered in the "Other" category if it is both a TEAE and is not serious. For each Serious AE and "Other" AE, for each term and treatment group, the following are provided:
  - o the number of participants at risk of an event
  - o the number of participants who experienced each event term
  - o the number of events experienced
- Consistent with www.ClinicalTrials.gov requirements, "Other" AEs that occur in fewer than 5% of patients/subjects in every treatment group may not be included if a 5% threshold is chosen (5% is the minimum threshold).
- AE reporting is consistent with other document disclosures for example, the CSR, manuscripts, and so forth.

#### 7. References

- Basra MK, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. *Br J Dermatol*. 2008;159(5):997-1035.
- Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. *BMJ*. 1992;305(6846):160-164.
- Clegg DO, Reda DJ, Mejias E, Cannon GW, Weisman MH, Taylor T, Budiman-Mak E, Blackburn WD, Vasey FB, Mahowald ML, Cush JJ, Schumacher HR Jr, Silverman SL, Alepa FP, Luggen ME, Cohen MR, Makkena R, Haakenson CM, Ward RH, Manaster BJ, Anderson RJ, Ward JR, Henderson WG. Comparison of sulfasalazine and placebo in the treatment of psoriatic arthritis. A Department of Veterans Affairs Cooperative Study. *Arthritis Rheum*. 1996;39(12):2013-2020.
- Coates LC, Fransen J, Helliwell PS. Defining minimal disease activity in psoriatic arthritis: a proposed objective target for treatment. *Ann Rheum Dis.* 2010a;69(1):48-53.
- Coates LC, Helliwell PS. Validation of minimal disease activity criteria for psoriatic arthritis using interventional trial data. *Arthritis Care Res (Hoboken)*. 2010b;62(7):965-969.
- [CHMP] Committee for Medicinal Products for Human Use. Guideline on the Choice of the Noninferiority Margin. European Medicines Agency web site. EMEA/CPMP/EWP/2158/99. Available at:
  - http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2009/09/WC50 0003636.pdf. 27 July 2005. Accessed February 27, 2017.
- The EuroQol Group. EQ-5D-5L user guide, version 2.0. October 2013. Available at: http://www.euroqol.org/fileadmin/user\_upload/Documenten/PDF/Folders\_Flyers/UserGuide\_EQ-5D-5L\_v2.0\_October\_2013.pdf. Accessed April 02, 2015.
- Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI) a simple practical measure for routine clinical use. *Clin Exp Dermatol*. 1994;19(3):210-216.
- [FDA] Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER). Guidance for industry, non-inferiority clinical trials to establish effectiveness. November 2016. Available at: https://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/u cm202140.pdf. Accessed March 02, 2017.
- Fredriksson T, Pettersson U. Severe psoriasis—oral therapy with a new retinoid. *Dermatologica*. 1978;157(4):238-244.
- Fries JF, Spitz P, Kraines RG, Holman HR. Measurement of patient outcome in arthritis. *Arthritis Rheum.* 1980;23(2):137-145.
- Fries JF, Spitz PW, Young DY. The dimensions of health outcomes: the health assessment questionnaire, disability and pain scales. *J Rheumatol.* 1982;9(5):789-793.
- Healy PJ, Helliwell PS. Measuring dactylitis in clinical trials: which is the best instrument to use? *J Rheumatol.* 2007;34(6):1302-1306.

- Healy PJ, Helliwell PS. Measuring clinical enthesitis in psoriatic arthritis: assessment of existing measures and development of an instrument specific to psoriatic arthritis. *Arthritis Rheum*. 2008;59(5):686-691.
- Helliwell PS, Firth J, Ibrahim GH, Melsom RD, Shah I, Turner DE. Development of an assessment tool for dactylitis in patients with psoriatic arthritis. *J Rheumatol*. 2005;32(9):1745-1750.
- Hongbo Y, Thomas CL, Harrison MA, Salek MS, Finlay AY. Translating the science of quality of life into practice: what do Dermatology Life Quality Index scores mean? *J Invest Dermatol*. 2005;125(4):659-664.
- Khilji FA, Gonzalez M, Finlay AY. Clinical meaning of change in Dermatology Life Quality Index scores [abstract]. *Br J Dermatol.* 2002;147(Suppl 62):50.
- Mease PJ, Gladman DD, Ritchlin CT, Ruderman EM, Steinfeld SD, Choy EH, Sharp JT, Ory PA, Perdok RJ, Weinberg MA; Adalimumab Effectiveness in Psoriatic Arthritis Trial Study Group. Adalimumab for the treatment of patients with moderately to severely active psoriatic arthritis: results of a double-blind, randomized, placebo-controlled trial. *Arthritis Rheum*. 2005;52(10):3279-3289.
- Mease P, Genovese MC, Gladstein G, Kivitz AJ, Ritchlin C, Tak PP, Wollenhaupt J, Bahary O, Becker JC, Kelly S, Sigal L, Teng J, Gladman D. Abatacept in the treatment of patients with psoriatic arthritis: results of a six-month, multicenter, randomized, double-blind, placebo-controlled, phase II trial. *Arthritis Rheum*. 2011;63(4):939-948.
- Mease PJ, Okada M, Kishimoto M, Shuler CL, Carlier H, Lin CY, Mou J, Moriarty SR, Lee CH, Gladman DD. Efficacy and safety of ixekizumab in patients with active psoriatic arthritis: 52 week results from a phase 3 study (Spirit-P1). *Ann Rheum Dis.* 2016;75(suppl 2):96. Abstract OP0109.
- Mumtaz A, Gallagher P, Kirby B, Waxman R, Coates LC, Veale DJ, Helliwell P, FitzGerald O. Development of a preliminary composite disease activity index in psoriatic arthritis. *Ann Rheum Dis.* 2011;70(2):272-277.
- [NPF] National Psoriasis Foundation. The psoriasis and psoriatic arthritis pocket guide. 2009. Available at: www.psoriasis.org/document.doc?id=354. Accessed April 07, 2015.
- Ramey DR, Fries JF, Singh G. The Health Assessment Questionnaire 1995 status and review. In: Spilker B, editor. Quality of life and pharmacoleconomics in clinical trials. 2nd ed. Philadelphia: Lippincott-Raven Pub; 1996:p227-237.
- Salaffi F, Ciapetti A, Carotti M, Gasparini S, Gutierrez M. Disease activity in psoriatic arthritis: comparison of the discriminative capacity and construct validity of six composite indices in a real world. *Biomed Res Int.* 2014;(2014):528105.
- Sampson HA, Munoz-Furlong A, Campbell RL, Adkinson NF Jr, Bock SA, Branum A, Brown SG, Camargo CA Jr, Cydulka R, Galli SJ, Gidudu J, Gruchalla RS, Harlor AD Jr, Hepner DL, Lewis LM, Lieberman PL, Metcalfe DD, O'Connor R, Muraro A, Rudman A, Schmitt C, Scherrer D, Simons FE, Thomas S, Wood JP, Decker WW. Second symposium on the definition and management of anaphylaxis: Summary report—Second National Institute of

- Allergy and Infectious Disease/Food Allergy and Anaphylaxis Network symposium. *J Allergy Clin Immunol*. 2006;117(2):391-397.
- Saris-Baglama RN, Dewey CJ, Chisholm GB, Bjorner JB, Ware JE. SF health outcomes scoring software: user's guide. Lincoln (NE): QualityMetric, Incorporated; 2004.
- Smolen JS, Breedveld FC, Eberl G, Jones I, Leeming M, Wylie GL, Kirkpatrick J. Validity and reliability of the twenty-eight-joint count for the assessment of rheumatoid arthritis activity. *Arthritis Rheum.* 1995;38(1):38-43.
- Szende A, Oppe M, Devlin N, eds. EQ-5D Value sets: inventory, comparative review and user guide. Dordrecht, Netherlands: Springer; 2007.
- Vander Cruyssen B, Van Looy S, Wyns B, Westhovens R, Durez P, Van den Bosch F, Veys EM, Mielants H, De Clerck L, Peretz A, Malaise M, Verbruggen L, Vastesaeger N, Geldhof A, Boullart L, De Keyser F. DAS28 best reflects the physician's clinical judgment of response to infliximab therapy in rheumatoid arthritis patients: validation of the DAS28 score in patients under infliximab treatment. *Arthritis Res Ther.* 2005;7(5):R1063-R1071.
- Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36): I. conceptual framework and item selection. *Med Care*. 1992;30(6):473-483.
- Weinblatt ME, Schiff M, Valente R, van der Heijde D, Citera G, Zhao C, Maldonado M, Fleischmann R. Head-to-head comparison of subcutaneous abatacept versus adalimumab for rheumatoid arthritis: findings of a phase IIIb, multinational, prospective, randomized study. *Arthritis Rheum.* 2013;65(1):28-38.

# 8. Appendices

# **Appendix 1. Definition of Numbers Needed to Treat (NNT)**

Numbers needed to treat (NNT) is defined as reciprocal of the difference in response rate between active treatment and comparator (Absolute Risk Reductions [ARR]). For instance, if ADA and IXE had response rates of 30% and 60%, respectively, then NNT=1/(0.6-0.3)=3.3. As for the CI, we take the CI for NNT as the reciprocal of the CI for ARR. The NNT and its CI will not be reported if 0 is included in the CI for ARR, i.e. the superiority test for two treatment arms is not significant.

Reference Table: List of Topical Treatments that are Prescribed/Administered for Psoriasis or Psoriatic Arthritis Patients with Appropriate ATC Code

| Topical Treatments | ATC Code |
|---|---|
| Topical corticosteroids: These powerful anti-inflammatory drugs are the most frequently prescribed | D07 |
| medications for treating mild-to-moderate psoriasis. They slow cell turnover by suppressing the | (Level 2) |
| immune system, which reduces inflammation and relieves associated itching. Topical corticosteroids | (Level 2) |
| range in strength from mild to very strong. Low-potency corticosteroid ointments are usually | |
| recommended for sensitive areas, such as your face or skinfolds, and for treating widespread patches | |
| of damaged skin. Your doctor may prescribe stronger corticosteroid ointment for small areas of your | |
| skin, for persistent plaques on your hands or feet, or when other treatments have failed. Medicated | |
| foams and scalp solutions are available to treat psoriasis patches on the scalp. Long-term use or | |
| overuse of strong corticosteroids can cause thinning of the skin and resistance to the treatment's | |
| benefits. To minimize side effects and to increase effectiveness, topical corticosteroids are generally | |
| used on active outbreaks until they are under control. | |
| • | A11CC |
| Vitamin D analogs: These synthetic forms of vitamin D slow down the growth of skin cells. | ATICC |
| Calcipotriene (Dovonex) is a prescription cream or solution containing a vitamin D analog that may | |
| be used alone to treat mild-to-moderate psoriasis or in combination with other topical medications or | |
| phototherapy. This treatment can irritate the skin. Calcitriol (Rocaltrol) is expensive, but may be | |
| equally effective and possibly less irritating than calcipotriene. | D0516 |
| <b>Anthralin:</b> This medication is believed to normalize DNA activity in skin cells. Anthralin (Dritho- | D05AC |
| Scalp) can also remove scale, making the skin smoother. However, anthralin can irritate skin, and it | |
| stains virtually anything it touches, including skin, clothing, countertops, and bedding. For that | |
| reason, doctors often recommend short-contact treatment – allowing the cream to stay on your skin for | |
| a brief time before washing it off. Anthralin is sometimes used in combination with ultraviolet light. | |
| <b>Topical retinoids:</b> These are commonly used to treat acne and sun-damaged skin, but tazarotene | D05BB |
| (Tazorac, Avage) was developed specifically for the treatment of psoriasis. Like other vitamin A | |
| derivatives, it normalizes DNA activity in skin cells and may decrease inflammation. The most | |
| common side effect is skin irritation. It may also increase sensitivity to sunlight, so sunscreen should | |
| be applied while using the medication. Although the risk of birth defects is far lower for topical | |
| retinoids than for oral retinoids, your doctor needs to know if you are pregnant or intend to become | |
| pregnant if you are using tazarotene. | |
| Calcineurin inhibitors: Currently, calcineurin inhibitors – tacrolimus (Prograf) and pimecrolimus | L04AD |
| (Elidel) – are approved only for the treatment of atopic dermatitis, but studies have shown them to be | |
| effective, at times, in the treatment of psoriasis. Calcineurin inhibitors are thought to disrupt the | |
| activation of T cells, which in turn reduces inflammation and plaque buildup. The most common side | |
| effect is skin irritation. Calcineurin inhibitors are not recommended for long-term or continuous use | |
| because of a potential increased risk of skin cancer and lymphoma. Calcineurin inhibitors are used | |
| only with your doctor's input and approval. They may be especially helpful in areas of thin skin, such | |
| as around the eyes, where steroid creams or retinoids are too irritating or may cause harmful effects. | |
| Salicylic acid: Available over-the-counter (nonprescription) and by prescription, salicylic acid | D02AF |
| promotes sloughing of dead skin cells, and reduces scaling. Sometimes it is combined with other | |
| medications, such as topical corticosteroids or coal tar, to increase its effectiveness. Salicylic acid is | |
| available in medicated shampoos and scalp solutions to treat scalp psoriasis. | |
| Coal tar: A thick, black byproduct of the manufacture of petroleum products and coal, coal tar is | D05AA |
| probably the oldest treatment for psoriasis. It reduces scaling, itching, and inflammation. Exactly | |
| probably the oldest treatment for psoriasis. It reduces scaling, itching, and inflammation. Exactly how it works is not known. Coal tar has few known side effects, but it is messy, stains clothing and | |
| how it works is not known. Coal tar has few known side effects, but it is messy, stains clothing and bedding, and has a strong odor. Coal tar is available in over-the-counter shampoos, creams, and oils. | |

| Topical Treatments | |
|---|---|
| Moisturizers: By themselves, moisturizing creams will not heal psoriasis, but they can reduce | D02A- |
| itching and scaling and can help combat the dryness that results from other therapies. Moisturizers in | |
| an ointment base are usually more effective than are lighter creams and lotions. | |
| Calcipotriene | D05AX |
| Tazarotene | D05AX |
| Herbal and traditional preparations | V90 |

Note: ATC = WHOCC Anatomical Therapeutic Chemical classification system; WHOCC = World Health Organization Collaborating Centre for Drug Statistics Methodology.

## **Appendix 2.** Algorithm for Determining ACR Responses

Details presented in this appendix will use "x" as a generic symbol, and the appropriate number (either 20, 50, or 70) is to be filled in when implementing in dataset programming code.

ACRx response is defined as  $\ge x\%$  improvement from baseline in tender joint count (68 counts) and  $\ge x\%$  improvement in swollen joint count(66 counts), and  $\ge x\%$  improvement in at least three of the following five items:

- Patient's global assessment of arthritis pain;
- Patient's global assessment of disease activity;
- Physician's global assessment of disease activity;
- HAQ-DI;
- CRP

The following abbreviations will be used throughout this appendix to refer to the items needed in the algorithm definitions:

| Parameter | Abbreviation for the Parameter |
|---|---|
| % improvement in tender joint count | TJC68 |
| % improvement in swollen joint count | SJC66 |
| % improvement in patient's assessment pain | PATPAIN |
| % improvement in patient's global assessment of disease activity | PATGA |
| % improvement in physician's global assessment of disease activity | PHYGA |
| % improvement in HAQ-DI | HAQ |
| % improvement in CRP | CRP |

For all seven parameters mentioned above, % improvement at a visit is calculated as:

(baseline value – value at visit) \* 100 / baseline value.

To calculate the *observed* ACRx response at a visit:

- **Step1:** If the patient discontinued from the study prior to reaching the visit, then STOP assign ACRx response as blank (ie, missing). Otherwise, calculate the % improvement at the visit for all seven parameters as described above.
- Step2:
  - o If TJC68 AND SJC66 are BOTH  $\ge x\%$ , then proceed to step3.
  - o If both are nonmissing but one or both is <x%, then STOP assign the patient as a non-responder for ACRx.
  - o If either or both are missing, proceed as follows:
    - a. If both are missing, then STOP assign ACRx response as blank (ie, missing).
    - b. If one of TJC68 or SJC66 is missing and the nonmissing value is < x%, then STOP assign the patient as a non-responder for ACRx.

- c. If one of TJC68 or SJC66 is missing and the nonmissing value is  $\ge x\%$ , then STOP assign ACRx response as blank (ie, missing).
- **Step3:** Consider the following five variables: PTPAIN, PTDISACT, PHYSDISACT, HAQ, and CRP.
  - o If three or more items are missing, then STOP assign ACRx response as blank (ie, missing).
  - o If three or more items are nonmissing, then proceed with the following order:
    - a. If at least three items are  $\ge x\%$ , then STOP assign the patient as a responder for ACRx.
    - b. If at least three items are < x%, then STOP assign the patient as a non-responder for ACRx.
    - c. If less than three items are  $\ge x\%$ , then STOP assign ACRx response as blank.
### **Appendix 3. Algorithm for Calculating Joint Counts**

Joints are evaluated and recorded as either non-evaluable, or if evaluable, then if tenderness is present or absent, and if swelling is present or absent. In total, 68 joints are assessed for tenderness and 66 are assessed for swelling. Hips are not assessed for swelling.

The number of tender/swollen joints will be calculated by summing all joints checked to have tenderness/swelling present. If at least half but not all of the joints are evaluable, then the observed prorated joint count will be calculated instead. The prorated scores for TJC will be adjusted based upon the number of evaluable joints: the counted score will be multiplied by 68 then divided by the number of joints evaluated (excluding non-evaluable joints and any joints with a missing response). For example: if only 60 of the 68 joints are assessed to be evaluable at a visit, and 32 of those 60 are tender, the prorated joint count is  $(32/60) \times 68 = 36.27$  (not 32). The prorated joint count will be rounded up to the next integer and be used in calculating the percent change from baseline in TJC. The same algorithm will be applied to the calculation of percent change from baseline in SJC with the exception that the counted score will be multiplied by 66 then divided by the number of joints evaluated. If less than half of the joints are evaluable, the number of tender/swollen joints is missing.

This same algorithm will be used for the calculation of TJC and SJC based on 28 joints, which is part of the 28 diarthrodial joint count, based on C-reactive protein (DAS28-CRP) score.

### Appendix 4. Algorithm for Calculating the HAQ-DI

The HAQ-DI is a patient-reported questionnaire to measure disease-associated disability (assessment of physical function). It consists of 24 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities (Fries et al. 1980, 1982; Ramey et al. 1996).

- **Dressing and grooming** (C1. Dress yourself, including tying shoelaces and doing buttons, C2. Shampooing your Hair)
  - Includes 2 component questions, 1 device checkbox (devices used for dressing), 1 help checkbox
- **Arising** (C1. Stand up from straight chair, C2. Get in and out of bed)
  - o Includes 2 component questions, 1 device checkbox (built-up or special chair), 1 help checkbox
- **Eating** (C1. Cut your meat, C2. Lift a cup or glass to your mouth, C3. Open a new carton of milk)
  - Includes 3 component questions, 1 device checkbox (build-up or special utensils),
     1 help checkbox)
- Walking (C1. Walk outdoors on flat ground, C2. Climb up five steps)
  - o Includes 2 component questions, 4 device checkboxes (cane, walker, crutches, wheelchair), 1 help checkbox
- **Hygiene** (C1. Wash and dry your body, C2. Take a tub bath, C3. Gen on and off the toilet)
  - o Includes 3 component questions, 4 device checkboxes (raised toilet seat, bathtub seat, bathtub bar, long-handled appliances in bathroom), 1 help checkbox.
- **Reach** (C1. Reach and get down a 5 pound object (such as a bag of sugar) from just above your head, C2. Bend down to pick up clothing from the floor)
  - Includes 2 component questions, 1 device checkbox (long-handled appliances for reach), 1 help checkbox
- **Grip** (C1. Open car doors, C2. Open jars which have been previously opened, C3. Turn faucets on and off)
  - o Includes 3 component questions, 1 device checkbox (jar opener), 1 help checkbox
- Activities (C1. Run errands and shop, C2. Get in and out of a car, C3. Do chores such as vacuuming or yard work)
  - o Includes 3 component questions, 1 help checkbox

In order to compute the HAQ-DI (Standard Disability Index) score, the following scores are assigned to the responses:

Without any difficulty = 0

With some difficulty = 1

With much difficulty = 2

Unable to do = 3.

The disability section of the questionnaire scores the patient's self-perception on the degree of difficulty (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do) when dressing and grooming, arising, eating, walking, hygiene, reach, grip, and performing other daily activities. The reported use of special aids or devices and/or the need for assistance of another person to perform these activities is also assessed. The scores for each of the functional domains will be averaged to calculate the functional disability index.

#### **Calculating the HAQ-DI:**

The patient must have a score for at least 6 of the 8 categories. If there are less than six categories completed, a HAQ-DI cannot be computed.

- A category score is determined from the highest score of the sub-categories, or components, in that category. (For example, in the category ARISING there are three sub-category items. If a patient responds with a 1, 2, and 0, respectively; the category score is 2.)
- Adjust for use of aids/devices and/or help from another person when indicated :
  - When there are no aids or devices or help indicated for a category, the category's score is not modified.
  - When aids or devices or help ARE indicated by the patient, adjust the score for a
    category by increasing a zero or a one to a two. If a patient's highest score for that
    sub-category is a two it remains a two, and if a three, it remains a three.
  - o Sum the eight category scores
  - O Divide the sum by the number of categories answered (range 6-8)

The scale is not truly continuous but has 25 possible values (i.e., 0, 0.125, 0.250, 0.375 ... 3). The mapping of the aids or devices to the categories is the following:

| HAQ-DI Category | Companion Aids or Devices Item |
|---|---|
| Dressing and Grooming | Devices used for dressing (button hook, zipper pull, long handled shoe horn, etc.) |
| Arising | Built up or special chair |
| Eating | Built up or special utensils |
| Walking | Cane, walker, crutches, wheelchair |
| Hygiene | Raised toilet seat, bathtub seat, bathtub bar, long-handled appliances in bathroom |
| Reach | Long handled appliances for reach |
| Grip | Jar opener (for jars previously opened) |

#### **Appendix 5.** Algorithm for Calculating CPDAI and mCPDAI

CPDAI is a validated composite instrument to assess psoriatic disease activity and response to therapy (Mumtaz et al. 2011). This instrument assesses individual domains:

- peripheral arthritis as assessed by the number of tender and swollen joints and the HAQ-DI
- skin as assessed by the PASI and the DLQI
- enthesitis as assessed by the number of sites with enthesitis and the HAO-DI
- dactylitis as assessed by the number of digits affected and the HAQ-DI
- spinal disease as assessed by the BASDAI and ASQoL.

The table below shows the instruments for each domain and the range in their total score:

| Domain | Instrument | <b>Total Score Range</b> |
|----------------------|-------------|--------------------------|
| Peripheral arthritis | TJC/SJC | 0-68/0-66 |
| | HAQ-DI | 0-3 |
| Skin disease | PASI | 0-72 |
| | DLQI | 0-30 |
| Enthesitis | LEI | 0-6 |
| | HAQ-DI | 0-3 |
| Dactylitis | Digit Score | 0-20 |
| | HAQ-DI | 0-3 |
| Spinal disease | BASDAI | 0-10 |
| | ASQoL | 0-18 |

Each domain is scored from 0–3. Individual domain scores are summed to give an overall composite CPDAI score. The composite scores range from 0 to 15 for the assessment, with a higher score indicating higher disease activity. See the table below for details:

| Domain | Not involved (0) | Mild (1) | Moderate (2) | Severe (3) |
|---|---|---|---|---|
| Peripheral | eripheral TJC and SJC = 0 TJC or SJC $\leq$ 4; and TJ | | TJC or SJC ≤4 and HAQ- | TJC or SJC >4 and |
| arthritis | | HAQ-DI ≤0.5 | DI >0.5; or TJC or SJC >4 | HAQ-DI >0.5 |
| | | | and HAQ-DI ≤0.5 | |
| Skin | Absence of plaque | PASI ≤10 and DLQI | PASI ≤10 and DLQI >10; | PASI >10 and DLQI |
| disease | psoriasis as defined by | ≤10 | or | >10 |
| | the eCRF or PASI = $0$ | | PASI >10 and DLQI ≤10 | |
| Enthesitis | Absence of enthesitis | LEI ≤3 sites; | LEI ≤3 sites and HAQ-DI | LEI >3 and HAQ-DI |
| | as defined by the | HAQ-DI ≤0.5 | >0.5; or LEI >3 sites and | >0.5 |
| | eCRF | | HAQ-DI ≤0.5 | |
| Dactylitis | Absence of dactylitis | Digit score ≤3 digits; | Digit score ≤3 and HAQ- | Digit score >3 and |
| | as defined by the | HAQ-DI ≤0.5 | DI >0.5; or Digit score >3 | HAQ-DI >0.5 |
| | eCRF | | and HAQ-DI ≤0.5 | |
| Spinal | BASDAI = 0 and | BASDAI <4; | BASDAI <4 and ASQoL | BASDAI >4 and |
| disease | ASQoL = 0 | ASQoL <6 | ≥6; or BASDAI ≥4 and | ASQol ≥6 |
| | | | ASQoL <6 | |

The modified CPDAI will sum up each domain with the exception of spinal disease score (0–3). The composite scores range from 0 to 12 for the assessment, with a higher score indicating higher disease activity.

### Appendix 6. Deviation of SF-36v2® Health Survey, Acute Version Scores

The SF-36v2® Health Survey Scoring Software (QualityMetric Health Outcomes<sup>TM</sup> Scoring Software 4.5) will be used to calculate the SF-36v2® 8-domain and 2-component summary scores (Saris-Baglama et al. 2004). The SF-36 is a 36-item, patient-completed measure designed to be a short, multipurpose assessment of health in the areas of physical functioning, role-physical, role-emotional, bodily pain, vitality, social functioning, mental health, and general health. The 2 overarching dimensions of mental well-being and physical well-being are captured by the Physical Component Summary (PCS) and Mental Component Summary (MCS) scores, respectively. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. Items are answered on Likert scales of varying lengths. In this study, the SF-36 acute version will be used, which has a 1-week recall period (The SF Community – SF-36 Health Survey Update [WWW]).

The Scoring Software performs a 4-step process to calculate raw domain scores and t-scores consisting of

- 1. Data Cleaning and Item recording: First, data are checked for out of range values, converting invalid items to missing values. Next, items (BP01, BP02, GH01, GH03, GH05, VT01, VT02, SF01, MH03, MH05) are reverse scored, so that higher scores denote better health for all SF-36 items.
- 2. Although current research indicates a linear relationship between the SF-36 items and the underlying health concept, empirical research suggests that items GH01 and BP01 require recalibration to satisfy important scaling assumptions. Item GH01 will be rescored according to the following table:

| Response to GH01 | Recommended Value / Recalibrated Value |
|------------------|----------------------------------------|
| Excellent | 5.0 |
| Very Good | 4.4 |
| Good | 3.4 |
| Fair | 2.0 |
| Poor | 1.0 |

#### The BP01 will be rescored with

| Response Choices | Final Item Value |
|------------------|------------------|
| None | 6.0 |
| Very mild | 5.4 |
| Mild | 4.2 |
| Moderate | 3.1 |
| Severe | 2.2 |
| Very severe | 1.0 |

Item 08 (BP02) will be rescored if BP01 and BP02 were answered

| <b>Response Choices</b> | If BP02 Pre-coded<br>Item Value | and BP01 Pre-coded<br>Item Value | Then Final Item 08<br>(BP02) Value |
|---|---|---|---|
| Not at all | 1 | 1 | 6 |
| Not at all | 1 | 2-6 | 5 |
| A little bit | 2 | 1-6 | 4 |
| Moderately | 3 | 1-6 | 3 |
| Quite a bit | 4 | 1-6 | 2 |
| Extremely | 5 | 1-6 | 1 |

#### Scoring of BP02 if BP01 is not answered:

| Response Choices | Final Item Value |
|------------------|------------------|
| Not at all | 6.0 |
| A little bit | 4.75 |
| Moderately | 3.5 |
| Quite a bit | 2.25 |
| Extremely | 1.0 |

- 3. After this rescoring, the raw domain scores will be calculated for the scale. Domain scores are the simple algebraic sum of the final values for all items in that scale.
- 4. All raw domain scores will be transformed to a 0-100 scale, with 0 being the lowest and 100 the highest possible score.
- 5. Finally, the 0-100 scores will be transformed to t-score based scores. First, a z-score transformation using the mean for the respective recall period, here 1 week recall, of the 2009 general U.S. population will be used. Then the distribution of z-score is linearly transformed to have a mean of 50 and a SD of 10 by multiplying each z-score with 10 and adding 50.

The calculation of component scores is a 3-step process using the domain scores, calculated as described above:

- 1. The standardized scores from Step 5, depending on the chosen recall period, are calculated.
- These standardized Physical and Mental component scores are calculated as the weighted sums by the factor score coefficients, derived from the 1990 general U.S. population, with the domain scores. If any domain score is missing then the aggregate Physical or Mental score will not be calculated.
- 3. The PCS and MCS are linearly transformed by multiplying by 10 and adding 50 to obtain the aggregate t-score based scoring.

To run the scoring algorithm, the SF-36 items recorded in the study database will be exported into a comma- or tab-separated values file (\*.csv, \*.tab). This file will then be loaded into the

Scoring Software to perform the calculations described above. The resulting raw domain scores and t-scores (domain scores) will then be exported into a comma- or tab-separated values file and imported into SAS for storage in the SDTM/ADaM datasets.

The comma- or tab-separated values file, each row will be one patient record and the first row will comprise the header columns, will have the following column specification: (to comply with the Scoring Software requirements)

| eCRF | Column label | Annotated SF-36 eCRF | Item Number, | eCRF question / Specification |
|---|---|---|---|---|
| Row | for export to | Variable | Score range | |
| # | comma- or | [Format: | | |
| | tab-separated | SF36V2RXX_SF36V2F1] | | |
| | values file | | | |
| | [*.csv, *.tab] | | | |
| 1 | GH01 | [SF36V2R01_SF36V2F1] | Item # 1, | In general, would you say your |
| | | | Range 1-5 | health is: |
| 2 | HT | [SF36V2R02_SF36V2F1] | Item # 2, | Compared to one week ago, how |
| | | | Range 1-5 | would you rate your health in general |
| | | | | now? |
| 3 | PF01 | [SF36V2R03_SF36V2F1] | Item # 3a, | Vigorous activities, such as running, |
| | | | Range 1-3 | lifting heavy objects, participating in |
| | | | - " | strenuous sports |
| 4 | PF02 | [SF36V2R04_SF36V2F1] | Item # 3b, | Moderate activities, such as moving a |
| | | | Range 1-3 | table, pushing a vacuum cleaner, |
| _ | 2500 | FORD CLIAR OF GRACILARIA | 7. // 2 | bowling, or playing golf |
| 5 | PF03 | [SF36V2R05_SF36V2F1] | Item # 3c, | Lifting or carrying groceries |
| | DE0.4 | FORM (LIADA C. ORA (LIADA) | Range 1-3 | |
| 6 | PF04 | [SF36V2R06_SF36V2F1] | Item # 3d, | Climbing several flights of stairs |
| 7 | DE05 | [GE2(V2D07, GE2(V2E1) | Range 1-3 | Climbing and Climb of the control |
| / | PF05 | [SF36V2R07_SF36V2F1] | Item # 3e,<br>Range 1-3 | Climbing one flight of stairs |
| 8 | PF06 | [SF36V2R08_SF36V2F1] | Item # 3f, | Bending, kneeling, or stooping |
| 0 | 1100 | [5F30V2R06_5F30V2F1] | Range 1-3 | Bending, kneering, or stooping |
| 9 | PF07 | [SF36V2R09 SF36V2F1] | Item # 3g, | Walking more than a mile |
| | 1107 | [51 50 v 2R07_51 50 v 21 1] | Range 1-3 | waiking more than a finic |
| 10 | PF08 | [SF36V2R10 SF36V2F1] | Item # 3h, | Walking several hundred yards |
| | 1100 | [5156 / 2116_5156 / 211] | Range 1-3 | , wantang so veras manarea yaras |
| 11 | PF09 | [SF36V2R11_SF36V2F1] | Item # 3i, | Walking one hundred yards |
| | | | Range 1-3 | <i>S</i> |
| 12 | PF10 | [SF36V2R12_SF36V2F1] | Item # 3j, | Bathing or dressing yourself |
| | | , | Range 1-3 | |
| 13 | RP01 | [SF36V2R13_SF36V2F1] | Item # 4a, | Cut down the amount of time you |
| | | | Range 1-5 | spent on work or other activities |
| 14 | RP02 | [SF36V2R14_SF36V2F1] | Item # 4b, | Accomplished less than you would |
| | | | Range 1-5 | like |
| 15 | RP03 | [SF36V2R15_SF36V2F1] | Item # 4c, | Were limited in the kind of work or |
| | | | Range 1-5 | other activities |
| 16 | RP04 | [SF36V2R16_SF36V2F1] | Item # 4d, | Had difficulty performing the work |
| | | | Range 1-5 | or other activities (for example, it |

| eCRF<br>Row<br># | Column label<br>for export to<br>comma- or<br>tab-separated<br>values file<br>[*.csv, *.tab] | Annotated SF-36 eCRF<br>Variable<br>[Format:<br>SF36V2RXX_SF36V2F1] | Item Number,<br>Score range | eCRF question / Specification |
|---|---|---|---|---|
| | | | | took extra effort) |
| 17 | RE01 | [SF36V2R17_SF36V2F1] | Item # 5a, | Cut down the amount of time you |
| | | | Range 1-5 | spent on work or other activities |
| 18 | RE02 | [SF36V2R18_SF36V2F1] | Item # 5b, | Accomplished less than you would |
| 10 | DE02 | FORM (LIAD 10 OF A CLIAD 11 | Range 1-5 | like |
| 19 | RE03 | [SF36V2R19_SF36V2F1] | Item # 5c, | Did work or other activities less |
| 20 | CEO1 | [CE2(V2D20 CE2(V2E1] | Range 1-5 | carefully than usual |
| 20 | SF01 | [SF36V2R20_SF36V2F1] | Item # 6,<br>Range 1-5 | During the past week, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups? |
| 21 | BP01 | [SF36V2R21_SF36V2F1] | Item # 7,<br>Range 1-6 | How much bodily pain have you had during the past week? |
| 22 | BP02 | [SF36V2R22_SF36V2F1] | Item# 8,<br>Range 1-5 | During the past week, how much did pain interfere with your normal work (including both work outside the home and housework)? |
| 23 | VT01 | [SF36V2R23_SF36V2F1] | Item # 9a,<br>Range 1-5 | Did you feel full of life? |
| 24 | MH01 | [SF36V2R24_SF36V2F1] | Item # 9b,<br>Range 1-5 | Have you been very nervous? |
| 25 | MH02 | [SF36V2R25_SF36V2F1] | Item # 9c,<br>Range 1-5 | Have you felt so down in the dumps that nothing could cheer you up? |
| 26 | MH03 | [SF36V2R26_SF36V2F1] | Item # 9d,<br>Range 1-5 | Have you felt calm and peaceful? |
| 27 | VT02 | [SF36V2R27_SF36V2F1] | Item # 9e,<br>Range 1-5 | Did you have a lot of energy? |
| 28 | MH04 | [SF36V2R28_SF36V2F1] | Item # 9f,<br>Range 1-5 | Have you felt downhearted and depressed? |
| 29 | VT03 | [SF36V2R29_SF36V2F1] | Item # 9g,<br>Range 1-5 | Did you feel worn out? |
| 30 | MH05 | [SF36V2R30_SF36V2F1] | Item # 9h,<br>Range 1-5 | Have you been happy? |
| 31 | VT04 | [SF36V2R31_SF36V2F1] | Item # 9i,<br>Range 1-5 | Did you feel tired? |
| 32 | SF02 | [SF36V2R32_SF36V2F1] | Item # 10,<br>Range 1-5 | During the past week, how much of<br>the time has your physical health or<br>emotional problems interfered with<br>your social activities (like visiting<br>with friends, relatives, etc.)? |
| 33 | GH02 | [SF36V2R33_SF36V2F1] | Item # 11a,<br>Range 1-5 | I seem to get sick a little easier than other people |

| eCRF | Column label | Annotated SF-36 eCRF | Item Number, | eCRF question / Specification |
|---|---|---|---|---|
| Row | for export to | Variable | Score range | |
| # | comma- or | [Format: | | |
| | tab-separated | SF36V2RXX_SF36V2F1] | | |
| | values file | | | |
| | [*.csv, *.tab] | | | |
| 34 | GH03 | [SF36V2R34_SF36V2F1] | Item # 11b, | I am as healthy as anybody I know |
| | | | Range 1-5 | |
| 35 | GH04 | [SF36V2R35_SF36V2F1] | Item # 11c, | I expect my health to get worse |
| | | | Range 1-5 | |
| 36 | GH05 | [SF36V2R36_SF36V2F1] | Item # 11d, | My health is excellent |
| | | | Range 1-5 | |
| | SUBJID | | | Subjects ID |
| | VISID | | | Visid ID |
| | Sex | | | Sex coded as: f/m |
| | DateOfBirth | | | Date of birth formatted as: |
| | | | | mm/dd/yyyy (when scoring software |
| | | | | is run in US), or dd/mm/yyyy (when |
| | | | | scoring software is run in non-US) |
| | RecordID | | | Running number for the exported |
| | | | | records |

The SF-36 Scoring Software will derive raw domain scores and t-scores that can be exported into a comma- or tab-separated values file (\*.csv, \*.tab) with the following columns added:

| Column label added to comma- or tab-<br>separated values file from export | Scoring Software specification |
|---|---|
| [*.csv, *.tab] | |
| PF | Physical Functioning domain score |
| RP | Role Limitations Due To Physical Health domain score |
| BP | Bodily Pain domain score |
| GH | General Health Perceptions domain score |
| VT | Vitality domain score |
| SF | Social Functioning domain score |
| RE | Role Limitations Due To Emotional Problems domain score |
| MH | Mental Health domain score |
| PCS | Physical Component score |
| MCS | Mental health Component score |

For scoring the trial data, the Missing Data Estimator option will not be selected. If an item is missing, there will be no imputation conducted by the Scoring Software. <u>Only</u> complete questionnaire data will be scored.

The Scoring Software also allows for calculating domain and component scores from weights derived from a oblique factor solution for comparative purposes. This option will <u>not</u> be used.

The SF-36 scoring using the Scoring Software will be conducted by a 2 person team overseeing each other in a single scoring session. In case of relevant observations during the scoring, those will be documented in pertinent meeting minutes and filed as part of the study documentation.

## Appendix 7. Anti-infective Treatments and Anatomical Therapeutic Chemical (ATC) Code List

| ATC | ATC | |
|---|---|---|
| Code | Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
| A01AB | 4 | ANTIINFECTIVES AND ANTISEPTICS FOR LOCAL ORAL TREA |
| A02BD | 4 | COMBINATIONS FOR ERADICATION OF HELICOBACTER PYLOR |
| A07A | 3 | INTESTINAL ANTIINFECTIVES |
| A07AA | 4 | ANTIBIOTICS |
| A07AB | 4 | SULFONAMIDES |
| A07AC | 4 | IMIDAZOLE DERIVATIVES |
| A07AX | 4 | OTHER INTESTINAL ANTIINFECTIVES |
| B05CA | 4 | ANTIINFECTIVES |
| C05AB | 4 | ANTIBIOTICS |
| D01 | 2 | ANTIFUNGALS FOR DERMATOLOGICAL USE |
| D01A | 3 | ANTIFUNGALS FOR TOPICAL USE |
| D01AA | 4 | ANTIBIOTICS |
| D01AC | 4 | IMIDAZOLE AND TRIAZOLE DERIVATIVES |
| D01AE | 4 | OTHER ANTIFUNGALS FOR TOPICAL USE |
| D01B | 3 | ANTIFUNGALS FOR SYSTEMIC USE |
| D01BA | 4 | ANTIFUNGALS FOR SYSTEMIC USE |
| D06 | 2 | ANTIBIOTICS AND CHEMOTHERAPEUTICS FOR DERMATOLOGIC |
| D06A | 3 | ANTIBIOTICS FOR TOPICAL USE |
| D06AA | 4 | TETRACYCLINE AND DERIVATIVES |
| D06AX | 4 | OTHER ANTIBIOTICS FOR TOPICAL USE |
| D06B | 3 | CHEMOTHERAPEUTICS FOR TOPICAL USE |
| D06BA | 4 | SULFONAMIDES |
| D06BB | 4 | ANTIVIRALS |
| D06BX | 4 | OTHER CHEMOTHERAPEUTICS |
| D06C | 3 | ANTIBIOTICS AND CHEMOTHERAPEUTICS, COMBINATIONS |
| D07C | 3 | CORTICOSTEROIDS, COMBINATIONS WITH ANTIBIOTICS |
| D07CA | 4 | CORTICOSTEROIDS, WEAK, COMBINATIONS WITH ANTIBIOTICS |
| | | CORTICOSTEROIDS, MODERATELY POTENT, COMBINATIONS WITH |
| D07CB | 4 | ANTIBIOTICS |
| D07CC | 4 | CORTICOSTEROIDS, POTENT, COMBINATIONS WITH ANTIBIOTICS |
| D07CD | 4 | CORTICOSTEROIDS, VERY POTENT, COMBINATIONS WITH ANTIBIOTICS |
| D09AA | 4 | MEDICATED DRESSINGS WITH ANTIINFECTIVES |
| D10AF | 4 | ANTIINFECTIVES FOR TREATMENT OF ACNE |
| G01AA | 4 | ANTIBIOTICS |
| G01AC | 4 | QUINOLINE DERIVATIVES |
| G01AE | 4 | SULFONAMIDES |
| G01AF | 4 | IMIDAZOLE DERIVATIVES |
| G01AG | 4 | TRIAZOLE DERIVATIVES |
| G01AX | 4 | OTHER ANTIINFECTIVES AND ANTISEPTICS |
| G01BA | 4 | ANTIBIOTICS AND CORTICOSTEROIDS |

| ATC<br>Code | ATC<br>Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
|---|---|---|
| G01BC | 4 | QUINOLINE DERIVATIVES AND CORTICOSTEROIDS |
| G01BE | 4 | SULFONAMIDES AND CORTICOSTEROIDS |
| G01BF | 4 | IMIDAZOLE DERIVATIVES AND CORTICOSTEROIDS |
| G04AB | 4 | QUINOLONE DERIVATIVES (EXCL. J01M) |
| G04AC | 4 | NITROFURAN DERIVATIVES |
| G04AG | 4 | OTHER URINARY ANTISEPTICS AND ANTIINFECT |
| G04AH | 4 | SULFONAMIDES IN COMBINATION WITH OTHER DRUGS |
| G04AK | 4 | URINARY ANTISEPT&ANTIINF, COMB EXCL SULFONAMIDES |
| J01 | 2 | ANTIBACTERIALS FOR SYSTEMIC USE |
| J01A | 3 | TETRACYCLINES |
| J01AA | 4 | TETRACYCLINES |
| J01B | 3 | AMPHENICOLS |
| J01BA | 4 | AMPHENICOLS |
| J01C | 3 | BETA-LACTAM ANTIBACTERIALS, PENICILLINS |
| J01CA | 4 | PENICILLINS WITH EXTENDED SPECTRUM |
| J01CE | 4 | BETA-LACTAMASE SENSITIVE PENICILLINS |
| J01CF | 4 | BETA-LACTAMASE RESISTANT PENICILLINS |
| J01CG | 4 | BETA-LACTAMASE INHIBITORS |
| J01CR | 4 | COMBINATIONS OF PENICILLINS, INCL. BETA-LACTAMASE |
| J01D | 3 | OTHER BETA-LACTAM ANTIBACTERIALS |
| J01DA | 4 | CEPHALOSPORINS AND RELATED SUBSTANCES |
| J01DB | 4 | FIRST-GENERATION CEPHALOSPORINS |
| J01DC | 4 | SECOND-GENERATION CEPHALOSPORINS |
| J01DD | 4 | THIRD-GENERATION CEPHALOSPORINS |
| J01DE | 4 | FOURTH-GENERATION CEPHALOSPORINS |
| J01DF | 4 | MONOBACTAMS |
| J01DH | 4 | CARBAPENEMS |
| J01DI | 4 | OTHER CEPHALOSPORINS |
| J01E | 3 | SULFONAMIDES AND TRIMETHOPRIM |
| J01EA | 4 | TRIMETHOPRIM AND DERIVATIVES |
| J01EB | 4 | SHORT-ACTING SULFONAMIDES |
| J01EC | 4 | INTERMEDIATE-ACTING SULFONAMIDES |
| J01ED | 4 | LONG-ACTING SULFONAMIDES |
| J01EE | 4 | COMBINATIONS OF SULFONAMIDES AND TRIMETHOPRIM, INC |
| J01F | 3 | MACROLIDES, LINCOSAMIDES AND STREPTOGRAMINS |
| J01FA | 4 | MACROLIDES |
| J01FF | 4 | LINCOSAMIDES |
| J01FG | 4 | STREPTOGRAMINS |
| J01G | 3 | AMINOGLYCOSIDE ANTIBACTERIALS |
| J01GA | 4 | STREPTOMYCINS |
| J01GB | 4 | OTHER AMINOGLYCOSIDES |
| J01M | 3 | QUINOLONE ANTIBACTERIALS |
| J01MA | 4 | FLUOROQUINOLONES |
| J01MB | 4 | OTHER QUINOLONES |
| J01R | 3 | COMBINATIONS OF ANTIBACTERIALS |
| J01RA | 4 | COMBINATIONS OF ANTIBACTERIALS |

| ATC<br>Code | ATC<br>Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
|---|---|---|
| J01WA | 4 | HERBAL ANTIBACTERIALS FOR SYSTEMIC USE |
| J01WB | 4 | HERBAL URINARY ANTISEPTICS AND ANTIINFECTIVES |
| J01X | 3 | OTHER ANTIBACTERIALS |
| J01XA | 4 | GLYCOPEPTIDE ANTIBACTERIALS |
| J01XB | 4 | POLYMYXINS |
| J01XC | 4 | STEROID ANTIBACTERIALS |
| J01XD | 4 | IMIDAZOLE DERIVATIVES |
| J01XE | 4 | NITROFURAN DERIVATIVES |
| J01XX | 4 | OTHER ANTIBACTERIALS |
| J02 | 2 | ANTIMYCOTICS FOR SYSTEMIC USE |
| J02A | 3 | ANTIMYCOTICS FOR SYSTEMIC USE |
| J02AA | 4 | ANTIBIOTICS |
| J02AB | 4 | IMIDAZOLE DERIVATIVES |
| J02AC | 4 | TRIAZOLE DERIVATIVES |
| J02AX | 4 | OTHER ANTIMYCOTICS FOR SYSTEMIC USE |
| J04AA | 4 | AMINOSALICYLIC ACID AND DERIVATIVES |
| J04AB | 4 | ANTIBIOTICS |
| J04AC | 4 | HYDRAZIDES |
| J04AK | 4 | OTHER DRUGS FOR TREATMENT OF TUBERCULOSIS |
| J04AM | 4 | COMBINATIONS OF DRUGS FOR TREATMENT OF TUBERCULOSI |
| J04B | 3 | DRUGS FOR TREATMENT OF LEPRA |
| J04BA | 4 | DRUGS FOR TREATMENT OF LEPRA |
| J05 | 2 | ANTIVIRALS FOR SYSTEMIC USE |
| J05A | 3 | DIRECT ACTING ANTIVIRALS |
| J05AA | 4 | THIOSEMICARBAZONES |
| J05AB | 4 | NUCLEOSIDES AND NUCLEOTIDES EXCL. REVERSE TRANSCRI |
| J05AC | 4 | CYCLIC AMINES |
| J05AD | 4 | PHOSPHONIC ACID DERIVATIVES |
| J05AE | 4 | PROTEASE INHIBITORS |
| J05AF | 4 | NUCLEOSIDE AND NUCLEOTIDE REVERSE TRANSCRIPTASE IN |
| J05AG | 4 | NON-NUCLEOSIDE REVERSE TRANSCRIPTASE INHIBITORS |
| J05AH | 4 | NEURAMINIDASE INHIBITORS |
| J05AR | 4 | ANTIVIRALS FOR TREATMENT OF HIV INFECTIONS, COMBIN |
| J05AX | 4 | OTHER ANTIVIRALS |
| P01A | 3 | AGENTS AGAINST AMOEBIASIS AND OTHER PROTOZOAL DISE |
| P01AA | 4 | HYDROXYQUINOLINE DERIVATIVES |
| P01AB | 4 | NITROIMIDAZOLE DERIVATIVES |
| P01AC | 4 | DICHLOROACETAMIDE DERIVATIVES |
| P01AR | 4 | ARSENIC COMPOUNDS |
| P01AX | 4 | OTHER AGENTS AGAINST AMOEBIASIS AND OTHER PROTOZOA |
| P01BA | 4 | AMINOQUINOLINES |
| P01BC | 4 | METHANOLQUINOLINES |
| P01BD | 4 | DIAMINOPYRIMIDINES |
| P01BE | 4 | ARTEMISININ AND DERIVATIVES, PLAIN |
| P01BF | 4 | ARTEMISININ AND DERIVATIVES, COMBINATIONS |
| P01BX | 4 | OTHER ANTIMALARIALS |

| ATC<br>Code | ATC<br>Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
|---|---|---|
| P01C | 3 | AGENTS AGAINST LEISHMANIASIS AND TRYPANOSOMIASIS |
| P01CA | 4 | NITROIMIDAZOLE DERIVATIVES |
| P01CB | 4 | ANTIMONY COMPOUNDS |
| P01CC | 4 | NITROFURAN DERIVATIVES |
| P01CD | 4 | ARSENIC COMPOUNDS |
| P01CX | 4 | OTHER AGENTS AGAINST LEISHMANIASIS AND TRYPANOSOMI |
| P02 | 2 | ANTHELMINTICS |
| P02B | 3 | ANTITREMATODALS |
| P02BA | 4 | QUINOLINE DERIVATIVES AND RELATED SUBSTANCES |
| P02BB | 4 | ORGANOPHOSPHOROUS COMPOUNDS |
| P02BX | 4 | OTHER ANTITREMATODAL AGENTS |
| P02C | 3 | ANTINEMATODAL AGENTS |
| P02CA | 4 | BENZIMIDAZOLE DERIVATIVES |
| P02CB | 4 | PIPERAZINE AND DERIVATIVES |
| P02CC | 4 | TETRAHYDROPYRIMIDINE DERIVATIVES |
| P02CE | 4 | IMIDAZOTHIAZOLE DERIVATIVES |
| P02CF | 4 | AVERMECTINES |
| P02CX | 4 | OTHER ANTINEMATODALS |
| P02D | 3 | ANTICESTODALS |
| P02DA | 4 | SALICYLIC ACID DERIVATIVES |
| P02DW | 4 | HERBAL ANTICESTODALS |
| P02DX | 4 | OTHER ANTICESTODALS |
| P02WA | 4 | HERBAL ANTHELMINTICS |
| P03A | 3 | CTOPARASITICIDES, INCL. SCABICIDES |
| P03AA | 4 | SULFUR CONTAINING PRODUCTS |
| P03AB | 4 | CHLORINE CONTAINING PRODUCTS |
| P03AC | 4 | PYRETHRINES, INCL. SYNTHETIC COMPOUNDS |
| P03AX | 4 | OTHER ECTOPARASITICIDES, INCL. SCABICIDES |
| P03BA | 4 | PYRETHRINES |
| R02AB | 4 | ANTIBIOTICS |
| S01A | 3 | ANTIINFECTIVES |
| S01AA | 4 | ANTIBIOTICS |
| S01AB | 4 | SULFONAMIDES |
| S01AD | 4 | ANTIVIRALS |
| S01AE | 4 | FLUOROQUINOLONES |
| S01AX | 4 | OTHER ANTIINFECTIVES |
| S01C | 3 | ANTIINFLAMMATORY AGENTS AND ANTIINFECTIVES IN COMB |
| S01CA | 4 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S01CB | 4 | CORTICOSTEROIDS/ANTIINFECTIVES/MYDRIATICS IN COMBI |
| S01CC | 4 | ANTIINFLAMMATORY AGENTS, NON-STEROIDS AND ANTIINFECTIVES |
| S02A | 3 | ANTIINFECTIVES |
| S02AA | 4 | ANTIINFECTIVES |
| S02C | 3 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S02CA | 4 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S03A | 3 | ANTIINFECTIVES |
| S03AA | 4 | ANTIINFECTIVES |

| ATC | ATC | |
|-------|-------|-----------------------------------------------------|
| Code | Level | ATC Description (Based on ATC Dictionary 18JAN2016) |
| S03C | 3 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |
| S03CA | 4 | CORTICOSTEROIDS AND ANTIINFECTIVES IN COMBINATION |

Abbreviation: ATC = WHOCC Anatomical Therapeutic Chemical classification system; INCL. = including; WHOCC = World Health Organization Collaborating Centre for Drug Statistics Methodology.

# Appendix 8. Lilly-Defined MedDRA V21.0 Preferred Terms for Opportunistic Infections (OIs)

| Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|
| Pneumocystis jirovecii (II) | | Narrow |
| | Pneumocystis jirovecii infection | |
| | Pneumocystis jirovecii pneumonia | |
| | Blood beta-D-glucan | Broad |
| | Blood beta-D-glucan abnormal | |
| | Blood beta-D-glucan increased | |
| | Gomori methenamine silver stain | |
| | Carbon monoxide diffusing capacity | |
| | decreased | |
| | Carbon monoxide diffusing capacity | |
| | Pneumocystis test positive | |
| Human Polyomavirus Infection | BK virus infection | Narrow |
| including BK virus disease and | Human polyomavirus infection | |
| PVAN (V), and Progressive | JC virus granule cell neuronopathy | |
| Multifocal Leukoencephalopathy | JC virus infection | |
| (IV) | Polyomavirus-associated nephropathy | |
| | Progressive multifocal leukoencephalopathy | |
| | Anti-JC virus antibody index | Broad |
| | JC polyomavirus test | |
| | JC virus test | |
| | JC virus test positive | |
| | Polyomavirus test | |
| | Polyomavirus test positive | |
| Cytomegalovirus disease (V) | Cytomegalovirus chorioretinitis | Narrow |
| | Cytomegalovirus colitis | |
| | Cytomegalovirus duodenitis | |
| | Cytomegalovirus enteritis | |
| | Cytomegalovirus enterocolitis | |
| | Cytomegalovirus gastritis | |
| | Cytomegalovirus gastroenteritis | |
| | Cytomegalovirus gastrointestinal infection | |
| | Cytomegalovirus gastrointestinal ulcer | |
| | Cytomegalovirus hepatitis | |
| | Cytomegalovirus infection | |
| | Cytomegalovirus mononucleosis | |
| | Cytomegalovirus mucocutaneous ulcer | |
| | Cytomegalovirus myelomeningoradiculitis | |
| | Cytomegalovirus myocarditis | |

| | D., C., 1 T., | L'Ha Da Caral |
|---|---|---|
| Opportunistic Infection | Preferred Term (MedDRA Version 21.0) | Lilly Defined<br>Classification |
| opportunistic infection | Cytomegalovirus oesophagitis | Ciussification |
| | Cytomegalovirus pancreatitis | |
| | Cytomegalovirus pericarditis | |
| | Cytomegalovirus syndrome | |
| | Cytomegalovirus urinary tract infection | |
| | Cytomegalovirus viraemia | |
| | Disseminated cytomegaloviral infection | |
| | Encephalitis cytomegalovirus | |
| | Pneumonia cytomegaloviral | |
| | Cytomegalovirus test | Broad |
| | Cytomegalovirus test positive | |
| Post-transplant lymphoproliferative | Epstein-Barr virus associated lymphoma | Narrow |
| disorder (EBV) (V) | Epstein-Barr virus associated | 1 (422 ) |
| | lymphoproliferative disorder | |
| | Epstein Barr virus positive mucocutaneous | |
| | ulcer | |
| | Post transplant lymphoproliferative disorder | |
| | 1 cos umanopum ijinproprometum v ancorae. | Broad |
| | Epstein-Barr viraemia | Broad |
| | Epstein-Barr virus infection | |
| | Lymphoproliferative disorder | |
| | Lymphoproliferative disorder in remission | |
| | Oral hairy leukoplakia | |
| Bartonellosis (disseminated disease | Bacillary angiomatosis | Narrow |
| only) (V) | Peliosis hepatis | |
| 3, ( ) | Splenic peliosis | |
| | Systemic bartonellosis | |
| | Trench fever | |
| | Bartonella test | Broad |
| | Bartonella test positive | |
| | Bartonellosis | |
| | Cat scratch disease | |
| Blastomycosis (IV) | Blastomycosis | Narrow |
| | Epididymitis blastomyces | |
| | Osteomyelitis blastomyces | |
| | Pneumonia blastomyces | |
| | NA | Broad |
| Toxoplasmosis (myocarditis, | Cerebral toxoplasmosis | Narrow |
| pneumonitis, or characteristic | Eye infection toxoplasmal | |
| retinochoroiditis only) (IV) | Hepatitis toxoplasmal | |
| | Meningitis toxoplasmal | |
| | Myocarditis toxoplasmal | |
| | Pneumonia toxoplasmal | |
| | Toxoplasma serology | Broad |
| | Toxoplasma serology positive | |

|---|---|---|
| | Toxoplasmosis | |
| Coccidioidomycosis (II) | Coccidioides encephalitis | Narrow |
| | Coccidioidomycosis | |
| | Cutaneous coccidioidomycosis | |
| | Meningitis coccidioides | |
| | NA | Broad |
| Histoplasmosis (II) | Acute pulmonary histoplasmosis | Narrow |
| | Chronic pulmonary histoplasmosis | |
| | Endocarditis histoplasma | |
| | Histoplasmosis | |
| | Histoplasmosis cutaneous | |
| | Histoplasmosis disseminated | |
| | Meningitis histoplasma | |
| | Pericarditis histoplasma | |
| | Retinitis histoplasma | |
| | | Broad |
| | Presumed ocular histoplasmosis syndrome | |
| Aspergillosis (invasive disease only) | Aspergillosis oral | Narrow |
| (II) | Cerebral aspergillosis | |
| | Meningitis aspergillus | |
| | Oro-pharyngeal aspergillosis | |
| | Aspergillus infection | Broad |
| | Aspergillus test | |
| | Aspergillus test positive | |
| | Bronchopulmonary aspergillosis | |
| | Sinusitis aspergillus | |
| Candidiasis (invasive disease or oral | Candida endophthalmitis | Narrow |
| not limited to the tongue) (II) | Candida osteomyelitis | 1 (4110 ) |
| not innited to the tongue) (11) | Candida pneumonia | |
| | Candida retinitis | |
| | Candida sepsis | |
| | Cerebral candidiasis | |
| | Endocarditis candida | |
| | Fungal oesophagitis | |
| | Gastrointestinal candidiasis | |
| | Hepatic candidiasis | |
| | Hepatosplenic candidiasis | |
| | Meningitis candida | |
| | Oesophageal candidiasis | |
| | Oropharyngeal candidiasis | |
| | Peritoneal candidiasis | |
| | Splenic candidiasis | |
| | Systemia aandida | |
| | Systemic candida Bladder candidiasis | Broad |

| Candida test positive Mucocutaneous candidiasis Oral candidiasis Oral fungal infection Respiratory moniliasis Oral fungal infection Respiratory moniliasis Cryptococcal cutaneous infection Cryptococcal fungaemia Cryptococcal fungaemia Cryptococcal Cryptococcal Meningitis cryptococcal Neurocryptococcosis Osscous cryptococcosis Pneumonia cryptococcosis Cryptococcus test Pneumonia cryptococcal Cryptococcus test Daroad Cryptococcus test Positive Allescheriosis Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Mucormycosis Seedosporum infection Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test Legionella test positive Listeria encephalitis Listeria espsis Meningitis listeria Listeria test positive Listeriosis Narrow Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | Opportunistic Infection | Preferred Term<br>(MedDRA Version 21.0) | Lilly Defined<br>Classification |
|---|---|---|---|
| Mucocutaneous candidiasis Oral candidiasis Oral candidiasis Oral fungal infection Respiratory moniliasis Cryptococcal cutaneous infection Cryptococcal fungaemia Cryptococcal fungaemia Cryptococcal fungaemia Cryptococcal fungaemia Cryptococcal Cryptococcal Meningitis cryptococcal Cryptococcus test positive Other invasive fungi: Allescheriosis Pneumonia cryptococcus test positive Allescheriosis Fusarium infection Phacohyphomycosis Seedosporum/Pseudallescheria boydii, Fusarium (II) Allescheriosis Seedosporum infection Phaeohyphomycotic brain abseess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria etest Listeria test Lis | | Candida test | |
| Oral candidiasis Oral fungal infection Respiratory moniliasis Cryptococcosis (II) Cryptococcal cutaneous infection Cryptococcal fungaemia Cryptococcosis Disseminated cryptococcosis Gastroenteritis cryptococcal Meningitis cryptococcal Meningitis cryptococcal Meningitis cryptococcal Meningitis cryptococcosis Osseous cryptococcosis Pneumonia cryptococcal Cryptococcus test Cryptococcus test Cryptococcus test Cryptococcus test Cryptococcus test positive Other invasive fungi: Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporumi Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomyc | | Candida test positive | |
| Cryptococcosis (II) Cryptococcal cutaneous infection Cryptococcal fungaemia Cryptococcal fungaemia Cryptococcosis Disseminated cryptococcosis Gastroenteritis cryptococcal Meningitis cryptococcal Meningitis cryptococcosis Osseous cryptococcosis Osseous cryptococcosis Osseous cryptococcosis Osseous cryptococcosis Pneumonia cryptococcal Cryptococcus test Cryptococcus test positive Other invasive fungi: Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichthemia, Scedosporumi Pseudallescheria boydii, Fusarium (II) Alescheriosis Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycosis Pseudallescheria infection Phaeohyphomycosis Pseudallescheria infection Phaeohyphomycosis Pseudallescheria infection Phaeohyphomycosis Pseudallescheria infection Phaeohyphomycosis Dese "Non-specific terms" below Broad Legionella test Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test positive Listeria estest Listeria test Listeria test Listeria test positive Listeria estest Listeria estest Listeria este Listeria este positive Listeria este positive Listeria este positive Listeria este sisteriosis Listeria est positive Listeria este positive | | Mucocutaneous candidiasis | |
| Respiratory moniliasis | | Oral candidiasis | |
| Cryptococcal cutaneous infection Cryptococcal fungaemia Cryptococcal fungaemia Cryptococcal fungaemia Cryptococcal Disseminated cryptococcal Meningitis cryptococcal Meningitis cryptococcal Neurocryptococcosis Oseous cryptococcal Neurocryptococcal Neurocryptococcosis Oseous cryptococcal Cryptococcus test Cryptococcus test Cryptococcus test Cryptococcus test positive Allescheriosis Fusarium fiction Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phacohyphomycosis Phacohyphomycosic terin abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionella test Listeria encephalitis Listeria est Listeria test Listeria test Listeria test Listeria test Listeria test Listeria test Listeria issis Listeriosis Adrenal gland tuberculosis Bone tuberculosis Narrow | | Oral fungal infection | |
| Cryptococcal fungaemia Cryptococcosis Disseminated cryptococcal Meningitis cryptococcal Cryptococcus so Osseous cryptococcal Cryptococcus test Cryptococcus test Cryptococcus test Cryptococcus test positive Allescheriosis Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycotic brain abseess Pseudallescheria infection Phaeohyphomycotic brain abseess Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria espsis Meningitis listeria Listeria test Listeria test tostitive Listeraemia Listeria test positive Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | Respiratory moniliasis | |
| Cryptococcosis Disseminated cryptococcal Meningitis cryptococcal Meningitis cryptococcal Meningitis cryptococcal Neurocryptococcosis Osseous cryptococcosis Osseous cryptococcosis Osseous cryptococcosis Pneumonia cryptococcal Cryptococcus test Cryptococcus test Cryptococcus test positive Other invasive fungi: Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Mucormycosis Scedosporium infection Phaeohyphomycosis | Cryptococcosis (II) | Cryptococcal cutaneous infection | Narrow |
| Disseminated cryptococcosis Gastroenteritis cryptococcal Meningitis cryptococcal Neurocryptococcosis Osseous cryptococcosis Osseous cryptococcosis Osseous cryptococcosis Osseous cryptococcosis Pneumonia cryptococcal Cryptococcus test Cryptococcus test positive Other invasive fungi: Allescheriosis Narrow Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporium/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test positive Listeria test Listeriosis Adrenal gland tuberculosis Bone tuberculosis | | Cryptococcal fungaemia | |
| Gastroenteritis cryptococcal Meningitis cryptococcal Neurocryptococcosis Osseous cryptococcosis Osseous cryptococcal Cryptococcus test Cryptococcus test Cryptococcus test positive Allescheriosis Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Seedosporum infection Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test Listeriosis Adrenal gland tuberculosis Bone tuberculosis | | Cryptococcosis | |
| Meningitis cryptococcal Neurocryptococcosis Osseous cryptococcal Cryptococcus test Cryptococcus test Cryptococcus test Cryptococcus test positive Allescheriosis Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test Listeria test Listeria test Listeria test Listeria test Listeria test positive Listeramia Listeriosis Adrenal gland tuberculosis Bone tuberculosis Narrow Narrow Narrow Proad Narrow | | Disseminated cryptococcosis | |
| Neurocryptococcosis Osseous cryptococcosis Osseous cryptococcosis Pneumonia cryptococcal Cryptococcus test positive Other invasive fungi: Mucornycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Seedosporium infection Phaeohyphomycosis Phaeohyphomycosic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | Gastroenteritis cryptococcal | |
| Osseous cryptococcosis Pneumonia cryptococcal Cryptococcus test Cryptococcus test Cryptococcus test positive Allescheriosis Rhizopus, Mucor, and Lichtheimia, Scedosporum/Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Seedosporum/Pseudallescheria boydii, Fusarium (II) Legionellosis (II) Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test Legionella test Listeria monocytogenes (invasive disease only) (II) Listeria test Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Broad Narrow Broad Listerous Broad Listerous Broad Listeria test Listeria test Listeria test Listeriosis Narrow | | Meningitis cryptococcal | |
| Pneumonia cryptococcal Cryptococcus test Cryptococcus test Cryptococcus test Cryptococcus test positive Allescheriosis Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test positive Listeria test tost Listeria test positive Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | Neurocryptococcosis | |
| Cryptococcus test Cryptococcus test Cryptococcus test Cryptococcus test positive Allescheriosis Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporium / Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test Listeria test Listeria test Listeria test positive Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | | |
| Other invasive fungi: Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/Pseudallescheria boydii, Fusarium (II) Legionellosis (II) Legionellosis (II) Legionellosis (II) Legionella test Listeria monocytogenes (invasive disease only) (II) Listeria test Listeria test Listeria test positive Listeria test Listeria itest positive Listeria test Listeria itest positive Listeria test | | Pneumonia cryptococcal | |
| Other invasive fungi: Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/Pseudallescheria boydii, Fusarium (II) Legionellosis (II) Legionellosis (II) Legionellosis (II) Legionella test Listeria monocytogenes (invasive disease only) (II) Listeria test Listeria test Listeria test positive Listeria test Listeria itest positive Listeria test Listeria itest positive Listeria test | | *1 | Broad |
| Other invasive fungi: Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria infec | | | |
| Mucormycosis (zygomycosis), Rhizopus, Mucor, and Lichtheimia, Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | Other invasive fungi: | | Narrow |
| Mucornycosis Scedosporum/Pseudallescheria Scedosporum infection Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria infection Pseudallescheria sepsis | • | | |
| Scedosporum/ Pseudallescheria boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria infection Pseudallescheria sepsis | | | |
| boydii, Fusarium (II) Phaeohyphomycosis Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria encephalitis Listeria test Listeria test Listeria test positive Listeria test positive Listeria test positive Listeria test positive Li | • | - | |
| Phaeohyphomycotic brain abscess Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test Listeria test Listeria test Listeria test Listeria test Listeria test positive Listeria test Listeria test positive Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Rone tuberculosis | - | * | |
| Pseudallescheria infection Pseudallescheria sepsis See "Non-specific terms" below Broad Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria test positive Listeria test Listeria test Listeria test Donad Listeria test Listeria test Listeria test Donad Listeria test Listeria test Donad Narrow Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | (12) | ** | |
| Pseudallescheria sepsis | | ** | |
| Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria encephalitis Listeria espsis Meningitis listeria Listeria test Listeria test positive Listeria test Listeria test Listeria test Listeria test Deroad Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | | |
| Legionellosis (II) Legionella infection Pneumonia legionella Pontiac fever Legionella test Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria encephalitis Listeria sepsis Meningitis listeria Listeria test Listeria test Listeria test positive Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | 1 seddaneseneria sepsis | |
| Pneumonia legionella Pontiac fever Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria encephalitis Listeria sepsis Meningitis listeria Listeria test Listeria test Listeria test positive Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Broad Narrow Narrow | | See "Non-specific terms" below | Broad |
| Legionella test Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria encephalitis Listeria sepsis Meningitis listeria Listeria test Listeria test positive Listeria test positive Listeria test positive Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Broad Narrow Narrow | Legionellosis (II) | Pneumonia legionella | Narrow |
| Legionella test positive Listeria monocytogenes (invasive disease only) (II) Listeria sepsis Meningitis listeria Listeria test Listeria test positive Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | | Broad |
| Listeria monocytogenes (invasive disease only) (II) Listeria encephalitis Listeria sepsis Meningitis listeria Listeria test Listeria test positive Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | | |
| disease only) (II) Listeria sepsis Meningitis listeria Listeria test Listeria test positive Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | Listeria monocytogenes (invasive | | Narrow |
| Meningitis listeria Listeria test Listeria test positive Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | * | 11011011 |
| Listeria test Listeria test positive Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | * | |
| Listeria test positive Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis | | | Broad |
| Listeraemia Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis Narrow | | | Divad |
| Listeriosis Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis Narrow | | - | |
| Tuberculosis (I) Adrenal gland tuberculosis Bone tuberculosis Narrow | | | |
| Bone tuberculosis | Tuboraulosis (I) | | Norrow |
| | i dociculosis (1) | = | INallow |
| | | Choroid tubercles | |

|---|---|
| Conjunctivitis tuberculous | |
| Cutaneous tuberculosis | |
| Disseminated Bacillus Calmette-Guerin | |
| infection | |
| Disseminated tuberculosis | |
| Ear tuberculosis | |
| Epididymitis tuberculous | |
| Extrapulmonary tuberculosis | |
| Immune reconstitution inflammatory | |
| syndrome associated tuberculosis | |
| Intestinal tuberculosis | |
| Joint tuberculosis | |
| Lymph node tuberculosis | |
| Male genital tract tuberculosis | |
| Meningitis tuberculous | |
| Oesophageal tuberculosis | |
| Oral tuberculosis | |
| Pericarditis tuberculous | |
| Peritoneal tuberculosis | |
| Prostatitis tuberculous | |
| Pulmonary tuberculoma | |
| Pulmonary tuberculosis | |
| Renal tuberculosis | |
| Salpingitis tuberculous | |
| Silico tuberculosis | |
| Spleen tuberculosis | |
| Thyroid tuberculosis | |
| Tuberculid | |
| Tuberculoma of central nervous system | |
| Tuberculosis | |
| Tuberculosis bladder | |
| Tuberculosis gastrointestinal | |
| Tuberculosis liver | |
| Tuberculosis of central nervous system | |
| Tuberculosis of eye | |
| Tuberculosis of genitourinary system | |
| Tuberculosis of intrathoracic lymph nodes | |
| Tuberculosis of peripheral lymph nodes | |
| Tuberculosis of peripheral tymph hodes Tuberculosis ureter | |
| Tuberculous abscess central nervous system | |
| Tuberculous abscess central nervous system Tuberculous endometritis | |
| Tuberculous laryngitis | |
| Tuberculous pleurisy Tuberculous tenosynovitis | |
| - | Drond |
| Interferon gamma release assay Interferon gamma release assay positive | Broad |

|---|---|---|
| | Mycobacterium tuberculosis complex test | |
| | Mycobacterium tuberculosis complex test | |
| | positive | |
| | Tuberculin test | |
| | Tuberculin test false negative | |
| | Tuberculin test positive | |
| Nocardiosis (II) | Cutaneous nocardiosis | Narrow |
| | Nocardia sepsis | |
| | Nocardiosis | |
| | Pulmonary nocardiosis | |
| | Nocardia test positive | Broad |
| Nontuberculous Mycobacterium | Atypical mycobacterial infection | Narrow |
| disease (II) | Atypical mycobacterial lower respiratory tract | |
| | infection | |
| | Atypical mycobacterial lymphadenitis | |
| | Atypical mycobacterial pneumonia | |
| | Atypical mycobacterium pericarditis | |
| | Borderline leprosy | |
| | Bovine tuberculosis | |
| | Indeterminate leprosy | |
| | Leprosy | |
| | Lepromatous leprosy | |
| | Mycobacterial infection | |
| | Mycobacterial peritonitis | |
| | Mycobacterium abscessus infection | |
| | Mycobacterium avium complex immune | |
| | restoration disease | |
| | Mycobacterium avium complex infection | |
| | Mycobacterium chelonae infection | |
| | Mycobacterium fortuitum infection | |
| | Mycobacterium kansasii infection | |
| | Mycobacterium marinum infection | |
| | Mycobacterium ulcerans infection | |
| | Superinfection mycobacterial | |
| | Tuberculoid leprosy | |
| | Type 1 lepra reaction | |
| | Type 2 lepra reaction | |
| | Atypical mycobacterium test positive | Broad |
| | Mycobacterial disease carrier | |
| | Mycobacterium leprae test positive | |
| | Mycobacterium test | |
| | Mycobacterium test positive | |
| Salmonellosis (invasive disease | Aortitis salmonella | Narrow |
| only) (II) | Arthritis salmonella | |
| 3/ ( / | Meningitis salmonella | |
| | Osteomyelitis salmonella | |

|---|---|---|
| | Paratyphoid fever | |
| | Pneumonia salmonella | |
| | Salmonella bacteraemia | |
| | Salmonella sepsis | |
| | Typhoid fever | |
| | Salmonella test positive | Broad |
| | Salmonellosis | |
| HBV reactivation (IV) | | Narrow |
| | Hepatitis B reactivation | |
| | Asymptomatic viral hepatitis | Broad |
| | Chronic hepatitis B | |
| | HBV-DNA polymerase increased | |
| | Hepatitis B | |
| | Hepatitis B antigen | |
| | Hepatitis B antigen positive | |
| | Hepatitis B core antigen | |
| | Hepatitis B core antigen positive | |
| | Hepatitis B DNA assay | |
| | Hepatitis B DNA assay positive | |
| | Hepatitis B DNA increased | |
| | Hepatitis B e antigen | |
| | Hepatitis B e antigen positive | |
| | Hepatitis B surface antigen | |
| | Hepatitis B surface antigen positive | |
| | Hepatitis B virus test | |
| | Hepatitis B virus test positive | |
| | Hepatitis infectious | |
| | Hepatitis post transfusion | |
| | Hepatitis viral | |
| | Withdrawal hepatitis | |
| Herpes simplex (invasive disease | Colitis herpes | Narrow |
| only) (IV) | Gastritis herpes | |
| | Herpes oesophagitis | |
| | Herpes sepsis | |
| | Herpes simplex colitis | |
| | Herpes simplex encephalitis | |
| | Herpes simplex gastritis | |
| | Herpes simplex hepatitis | |
| | Herpes simplex meningitis | |
| | Herpes simplex meningoencephalitis | |
| | Herpes simplex meningomyelitis | |
| | Herpes simplex necrotising retinopathy | |
| | Herpes simplex oesophagitis | |
| | Herpes simplex pneumonia | |
| | Herpes simplex sepsis | |
| | Herpes simplex viraemia | |

|---|---|---|
| | Herpes simplex visceral | |
| | Meningitis herpes | |
| | Meningoencephalitis herpetic | |
| | Meningomyelitis herpes | |
| | Pneumonia herpes viral | |
| | Eczema herpeticum | Broad |
| | Herpes ophthalmic | Brown |
| | Herpes simplex | |
| | Herpes simplex DNA test positive | |
| | Herpes virus infection | |
| | Herpes virus test abnormal | |
| | Herpes simplex virus test positive | |
| | Ophthalmic herpes simplex Ophthalmic herpes simplex | |
| | Ophulannic nerpes simplex | |
| Herpes zoster (any form) (II) | Disseminated varicella zoster vaccine virus | Narrow |
| | infection | |
| | Encephalitis post varicella | |
| | Genital herpes zoster | |
| | Herpes zoster | |
| | Herpes zoster cutaneous disseminated | |
| | Herpes zoster disseminated | |
| | Herpes zoster infection neurological | |
| | Herpes zoster meningitis | |
| | Herpes zoster meningoencephalitis | |
| | Herpes zoster meningomyelitis | |
| | Herpes zoster necrotising retinopathy | |
| | Herpes zoster oticus | |
| | Herpes zoster pharyngitis | |
| | Necrotising herpetic retinopathy | |
| | Ophthalmic herpes zoster | |
| | opiniumi nerpes zoster | |
| | Varicella zoster virus infection | Broad |
| | Varicella virus test | |
| | Varicella virus test positive | |
| Stronglyoides (hyperinfection | Strongyloidiasis | Narrow |
| syndrome and disseminated forms | NA | Broad |
| only) (IV) | 1111 | Dioud |
| Paracoccidioides infections (V) | Paracoccidioides infection | Narrow |
| ` ' | Pulmonary paracoccidioidomycosis | |
| | NA | Broad |
| Penicillium marneffei (V) | Penicilliosis | Narrow |
| ······································ | Penicillium test positive | Broad |
| Sporothrix schenckii (V) | Cutaneous sporotrichosis | Narrow |
| | Pulmonary sporotrichosis | |
| | Sporotrichosis | |
| | NA | Broad |
| | 1 * ** * | 21000 |

|---|---|---|
| Cryptosporidium species (chronic | Biliary tract infection cryptosporidial | Narrow |
| disease only) (IV) | Cryptosporidiosis infection | Broad |
| | Gastroenteritis cryptosporidial | |
| Microsporidiosis (IV) | Microsporidia infection | Narrow |
| - · | NA | Broad |
| Leishmaniasis (Visceral only) (IV) | Visceral leishmaniasis | Narrow |
| | Leishmaniasis | Broad |
| Trypanosoma cruzi infection (Chagas' Disease) (progression of | Chagas' cardiomyopathy | Narrow |
| chronic and disseminated disease | Meningitis trypanosomal | |
| only) (V) | American trypanosomiasis Trypanosomiasis Trypanosoma serology positive | Broad |
| Campylobacteriosis (invasive | Campylobacter sepsis | Narrow |
| disease only) (V) | Campylobacter infection | Broad |
| discuse only) (v) | Campylobacter test positive | Broad |
| Shigellosis (invasive disease only) | Shigella sepsis | Narrow |
| (V) | Shigella infection | Broad |
| (*) | Shigella test positive | Broad |
| Vibriosis (invasive disease due to $V$ . | NA | Narrow |
| vulfnificus) (V) | Vibrio test positive | Broad |
| vuijitijieus) (*) | Vibrio test positive Vibrio vulnificus infection | Broad |
| HCV progression (V) | NA | Narrow |
| | Chronic hepatitis C | Broad |
| | Hepatitis C | |
| | Hepatitis C RNA | |
| | Hepatitis C RNA increased | |
| | Hepatitis C RNA fluctuation | |
| | Hepatitis C RNA positive | |
| | Hepatitis C virus test | |
| | Hepatitis C virus test positive | |
| Non-specific terms | | Narrow |
| - | NA | |
| | Abscess fungal | Broad |
| | Alternaria infection | |
| | Arthritis fungal | |
| | Biliary tract infection fungal | |
| | Central nervous system fungal infection | |
| | Cerebral fungal infection | |
| | Encephalitis fungal | |
| | Erythema induratum | |
| | Eye infection fungal | |
| | Fungaemia | |
| | Fungal abscess central nervous system<br>Fungal endocarditis | |

|---|
| Fungal labyrinthitis |
| Fungal peritonitis |
| Fungal pharyngitis |
| Fungal retinitis |
| Fungal sepsis |
| Hepatic infection fungal |
| Meningitis fungal |
| Mycotic endophthalmitis |
| Myocarditis mycotic |
| Oropharyngitis fungal |
| Osteomyelitis fungal |
| Otitis media fungal |
| Pancreatitis fungal |
| Parasitic lung infection |
| Parasitic pneumonia |
| Pericarditis fungal |
| Phaehyphomycosis |
| Pneumonia fungal |
| Pulmonary mycosis |
| Pulmonary trichosporonosis |
| Sinusitis fungal |
| Splenic infection fungal |
| Systemic mycosis |

Abbreviations: EBV = Epstein-Barr virus; HBV = hepatitis B virus; HCV = hepatitis C virus; NA = not applicable; PVAN = polyomavirus-associated nephropathy.

# Appendix 9. MedDRA Preferred Terms for each Category Associated with Criterion 2 for Anaphylactic Allergic Reactions/Hypersensitivity Events

| Preferred Terms (MedDRA Version 21.0) | |
|---|---|
| Category A: Involvement of the Skin/Mucosal Tissue | |
| Administration site hypersensitivity | Localised oedema |
| Administration site rash | Mouth swelling |
| Administration site urticarial | Nasal obstruction |
| Allergic oedema | Nodular rash |
| Allergic otitis externa | Ocular hyperaemia |
| Angioedema | Oedema |
| Circumoral oedema | Oedema mouth |
| Drug eruption | Oedema mucosal |
| Erythema | Orbital oedema |
| Eye allergy | Palatal oedema |
| Eye oedema | Palatal swelling |
| Eye pruritus | Perineal rash |
| Eye swelling | Periorbital oedema |
| Eyelid oedema | Pruritus |
| Face oedema | Pruritus allergic |
| Flushing | Pruritus generalised |
| Generalised erythema | Rash |
| Gingival oedema | Rash erythematous |
| Gingival swelling | Rash generalised |
| Idiopathic urticaria | Rash pruritic |
| Injection site dermatitis | Skin oedema |
| Injection site hypersensitivity | Skin swelling |
| Injection site rash | Swelling |
| Injection site urticaria | Swelling face |
| Injection site vasculitis | Swollen tongue |
| Lip oedema | Tongue oedema |
| Lip swelling | Urticaria |
| | Urticaria papular |
| Category B: Respiratory Compromise | |
| Acute respiratory failure | Laryngotracheal oedema |
| Allergic cough | Oropharyngeal spasm |
| Allergic pharyngitis | Oropharyngeal swelling |
| Asthma | Pharyngeal oedema |
| Asthmatic crisis | Respiratory arrest |
| Bronchial hyperreactivity | Respiratory distress |
| Bronchial oedema | Respiratory failure |
| Bronchospasm | Respiratory tract oedema |
| Cardio-respiratory distress | Reversible airways obstruction |
| Chest discomfort | Sensation of foreign body |
| Choking | Sneezing |

| Preferred Terms (MedDRA Version 21.0) | |
|---|---|
| Choking sensation | Spasmodic dysphonia |
| Cough | Status asthmaticus |
| Cyanosis | Stridor |
| Dyspnoea | Tachypnea |
| Epiglottic oedema | Throat tightness |
| Hyperventilation | Tracheal obstruction |
| Нурохіа | Tracheal oedema |
| Laryngeal dyspnoea | Upper airway obstruction |
| Laryngeal obstruction | Wheezing |
| Laryngeal oedema | |
| Laryngitis allergic | |
| Laryngospasm | |
| Category C: Reduced Blood Pressure or Associated Sy | ymptoms |
| Blood pressure decreased | Hypoperfusion |
| Blood pressure diastolic decreased | Hypotension |
| Blood pressure systolic decreased | Hypovolaemic shock |
| Cardiac arrest | Incontinence |
| Cardiopulmonary failure | Mean arterial pressure decreased |
| Cardio-respiratory arrest | Peripheral circulatory failure |
| Cardiovascular insufficiency | Presyncope |
| Circulatory collapse | Shock |
| Diastolic hypotension | Shock symptom |
| Distributive shock | Syncope |
| Dizziness | Urinary Incontinence |
| Category D: Persistent Gastrointestinal Symptoms | |
| Abdominal discomfort | Gastrointestinal pain |
| Abdominal pain | Intestinal angioedema |
| Abdominal pain lower | Nausea |
| Abdominal pain upper | Retching |
| Diarrhoea | Visceral pain |
| Epigastric discomfort | Vomiting |
| Gastrointestinal oedema | |

Abbreviations: MedDRA = Medical Dictionary for Regulatory Activities.

### Appendix 10. Allergic Reactions/Hypersensitivity MedDRA Preferred Term List

Allergic reactions/hypersensitivities will be defined using the following MedDRA Preferred Terms as defined in MedDRA:

- Broad and narrow terms in the Anaphylactic reaction SMQ (20000021)
- Broad and narrow terms in the Angioedema SMQ (20000024)
- Broad and narrow terms in the Severe cutaneous adverse reactions SMQ (20000020)
- Broad and narrow terms in the Hypersensitivity SMQ (20000214), excluding the preferred terms as noted below.

| Preferred Terms (MedDRA v.21.0) from Hypersensitivity SMQ Excluded from Analysis | |
|---|---|
| Administration site dermatitis | Injection site rash |
| Administration site eczema | Injection site recall reaction |
| Administration site rash | Injection site urticaria |
| Administration site recall reaction | Injection site vasculitis |
| Allergic otitis externa | Instillation site hypersensitivity |
| Allergic otitis media | Instillation site rash |
| Allergic sinusitis | Instillation site urticaria |
| Allergic transfusion reaction | Iodine allergy |
| Allergy alert test positive | Mast cell degranulation present |
| Allergy test positive | Medical device site dermatitis |
| Allergy to surgical sutures | Medical device site eczema |
| Allergy to vaccine | Medical device site hypersensitivity |
| Anaphylactic transfusion reaction | Medical device site rash |
| Antiallergic therapy | Medical device site recall reaction |
| Application site dermatitis | Medical device site urticaria |
| Application site eczema | Nodular rash |
| Application site hypersensitivity | Pathergy reaction |
| Application site rash | Radioallergosorbent test positive |
| Application site recall reaction | Reaction to azo-dyes |
| Application site urticaria | Reaction to colouring |
| Application site vasculitis | Shock |
| Arthritis allergic | Shock symptom |
| Aspirin-exacerbated respiratory disease | Skin test positive |
| Asthma-chronic obstructive pulmonary disease | Solvent sensitivity |
| overlap syndrome | Stoma site hypersensitivity |
| Blepharitis allergic | Stoma site rash |
| Blood immunoglobulin E abnormal | Urticaria contact |
| Blood immunoglobulin E increased | Urticarial vasculitis |
| Bromoderma | Vaccination site dermatitis |
| Catheter site dermatitis | Vaccination site exfoliation |
| Catheter site eczema | Vaccination site eczema |
| Catheter site hypersensitivity | Vaccination site hypersensitivity |
| Catheter site rash | Vaccination site rash |

#### Preferred Terms (MedDRA v.21.0) from Hypersensitivity SMQ Excluded from Analysis

Catheter site urticaria Catheter site vasculitis

Chronic eosinophilic rhinosinusitis

Chronic hyperplastic eosinophilic sinusitis

Circulatory collapse Conjunctivitis allergic Contact stomatitis

Complement factor decreased Complement factor C1 decreased Complement factor C1 increased Complement factor C2 decreased

Complement factor C2 decreased Complement factor C2 increased Complement factor C3 decreased Complement factor C3 increased Complement factor C4 decreased Complement factor C4 increased Complement fixation abnormal Complement fixation test positive

Contrast media allergy
Contrast media reaction
Dennie-Morgan fold
Dermatitis acneiform
Dermatitis contact
Dermatitis herpetiformis
Dermatitis infected
Device allergy

Dialysis membrane reaction

Distributive shock
Drug cross-reactivity
Drug provocation test
Eczema infantile
Eczema vaccinatum
First use syndrome
Fixed drug eruption

Giant papillary conjunctivitis

Heparin-induced thrombocytopenia

Hereditary angioedema Implant site dermatitis Implant site hypersensitivity

Implant site rash
Implant site urticaria

Immune-mediated adverse reaction

Incision site dermatitis Incision site rash Infusion site dermatitis Infusion site eczema

Infusion site hypersensitivity

Vaccination site recall reaction

Vaccination site urticaria

Vaccination site vasculitis

Vaccination site vesicles

Vessel puncture site rash

Vessel puncture site vesicles

Vulvovaginal rash

Acute respiratory failure

Allergy to chemicals

Allergy to fermented products Anti-insulin antibody increased Anti-insulin antibody positive

Anti-insulin receptor antibody increased
Anti-insulin receptor antibody positive
Blood immunoglobulin A abnormal
Blood immunoglobulin A increased

Blood immunoglobulin D increased Blood immunoglobulin G abnormal Blood immunoglobulin G increased Blood immunoglobulin M abnormal Blood immunoglobulin M increased Immune complex level increased Immunoglobulins abnormal

Immunoglobulins increased Immunology test abnormal Haemolytic transfusion reaction

Infantile asthma Fixed eruption Rhinitis perennial Seasonal allergy

| Preferred Terms (MedDRA v.21.0) from Hypersensitivity SMQ Excluded from Analysis |
|---|
| Infusion site rash |
| Infusion site recall reaction |
| Infusion site urticaria |
| Infusion site vasculitis |
| Injection site dermatitis |
| Injection site eczema |
| Injection site hypersensitivity |

# Appendix 11. Lilly-Defined MedDRA V21.0 Preferred Terms for Inflammatory Bowel Disease (IBD)

| | | Lilly-Defined |
|---|---|---|
| Condition | Preferred Term (MedDRA version 21.0) | Classification |
| Inflammatory bowel disease | Inflammatory bowel disease | Narrow |
| Crohn's disease | Crohn's disease | Narrow |
| Ulcerative colitis | Acute haemorrhagic ulcerative colitis | Narrow |
| | Colitis ulcerative | Narrow |
| | Proctitis ulcerative | Narrow |
| Non-specific terms | Abscess intestinal | Broad |
| | Anal abscess | Broad |
| | Anal fistula | Broad |
| | Anal fistula excision | Broad |
| | Anal fistula infection | Broad |
| | Anovulvar fistula | Broad |
| | Aorto-duodenal fistula | Broad |
| | Colitis | Broad |
| | Colon fistula repair | Broad |
| | Colonic fistula | Broad |
| | Diverticular fistula | Broad |
| | Duodenal fistula | Broad |
| | Enterocolitis haemorrhagic | Broad |
| | Enterocolonic fistula | Broad |
| | Enterocutaneous fistula | Broad |
| | Enterovesical fistula | Broad |
| | Gastrointestinal fistula | Broad |
| | Gastrointestinal fistula repair | Broad |
| | Fistula of small intestine | Broad |
| | Intestinal fistula | Broad |
| | Intestinal fistula infection | Broad |
| | Intestinal fistula repair | Broad |
| | Jejunal fistula | Broad |
| | Large intestinal ulcer perforation | Broad |
| | Rectal fistula repair | Broad |
| | Faecal calprotectin abnormal | Broad |
| | Faecal calprotectin increased | Broad |
| | Proctitis haemorrhagic | Broad |
| | Pseudopolyposis | Broad |
| | Rectoprostatic fistula | Broad |
| | Rectourethral fistula | Broad |